# CLINICAL RESEARCH IN INFECTIOUS DISEASES

# STATISTICAL ANALYSIS PLAN

## for

# **DMID Protocol**

17-0075: A Phase II Study in Healthy Adults 19 Years and Older to Assess the Safety, Reactogenicity and Immunogenicity of a Sanofi Pasteur A/H7N9 Inactivated Influenza Vaccine Administered Intramuscularly With or Without AS03 Adjuvant

17-0075: NCT03312231

Version 2.0

**DATE: 26 August 2019** 

THIS COMMUNICATION IS PRIVILEGED AND CONFIDENTIAL

### **STUDY TITLE**

| <b>Protocol Number Code:</b> | DMID Protocol: 17-0075 |
|---|---|
| <b>Development Phase:</b> | Phase II |
| Products: | Sanofi A/H7N9 Inactivated Influenza Vaccine<br>GSK AS03 Adjuvant |
| Form/Route: | IM |
| Indication Studied: | Influenza A/H7N9 |
| Sponsor: | Division of Microbiology and Infectious Diseases National Institute of Allergy and Infectious Diseases National Institutes of Health |
| Clinical Trial Initiation Date: | 14 February 2018 |
| Clinical Trial Completion Date: | Expected September 2019 |
| Date of the Analysis Plan: | 26 August 2019 |
| Version Number: | 2.0 |

This study was performed in compliance with Good Clinical Practice.

Information contained in this publication is the property of Division of Microbiology and Infectious Diseases and is confidential. This information may not be disclosed to third parties without written authorization from Division of Microbiology and Infectious Diseases. This report may not be reproduced, stored in a retrieval system or transmitted in any form or by any means - electronic, mechanical, recording or otherwise - without the prior authorization from Division of Microbiology and Infectious Diseases. This document must be returned to Division of Microbiology and Infectious Diseases upon request.

# TABLE OF CONTENTS

| Study Title. | | ii |
|---|---|---|
| TABLE OF | CONTENTS | iii |
| List of Abbr | reviations | Vi |
| 1. PREFA | ACE | 1 |
| 2. INTRO | DUCTION | 2 |
| 2.1. Pu | rpose of the Analyses | 2 |
| 3. STUD | Y OBJECTIVES AND ENDPOINTS | 3 |
| 3.1. Stu | dy Objectives | 3 |
| 3.1.1. | Primary | 3 |
| 3.1.2. | Secondary | 3 |
| 3.2. En | dpoints | 4 |
| 3.2.1. | Primary | 4 |
| 3.2.2. | Secondary | 5 |
| 3.2.3. | Exploratory | 5 |
| 3.3. Stu | ndy Definitions and Derived Variables | 6 |
| 4. INVES | TIGATIONAL PLAN | 7 |
| 4.1. Ov | erall Study Design and Plan | 7 |
| 4.2. Dis | scussion of Study Design, Including the Choice of Control Groups | 7 |
| 4.3. Sel | lection of Study Population | 8 |
| 4.4. Tre | eatments | 8 |
| 4.4.1. | Treatments Administered | 8 |
| 4.4.2. | Identity of Investigational Product | 8 |
| 4.4.3. | Method of Assigning Subjects to Treatment Groups (Randomization) | 8 |
| 4.4.4. | Selection of Doses in the Study | 8 |
| 4.4.5. | Selection and Timing of Dose for Each Subject | 8 |
| 4.4.6. | Blinding | 8 |
| 4.4.7. | Prior and Concomitant Therapy | 9 |
| 4.4.8. | Treatment Compliance | 9 |
| 4.5. Im: | munogenicity and Safety Variables | 9 |
| 4.5.1. | Safety Variables | 9 |
| 4.5.2. | Immunogenicity Variables | 10 |
| 5. SAMP | LE SIZE CONSIDERATIONS | 11 |

# TABLE OF CONTENTS (continued)

| 6. | GENER | AL STATISTICAL CONSIDERATIONS | 12 |
|-----|---------|-------------------------------------------------------|----|
| 6. | 1. Gen | eral Principles | 12 |
| 6.2 | 2. Tim | ing of Analyses | 12 |
| | 6.2.1. | Expedited Interim Immunogenicity Reports | 12 |
| | 6.2.2. | Preliminary Report and CSR | 13 |
| 6.3 | 3. Ana | lysis Populations | 13 |
| | 6.3.1. | Safety Population | 13 |
| | 6.3.2. | Modified Intention-to-Treat (mITT) Population | 13 |
| | 6.3.3. | Per Protocol Population | 14 |
| 6.4 | 4. Cov | ariates and Subgroups | 14 |
| 6.5 | 5. Miss | sing Data | 15 |
| 6.0 | 6. Inte | rim Analyses and Data Monitoring | 15 |
| | 6.6.1. | Interim Safety Review | 15 |
| | 6.6.2. | Interim Immunogenicity Review | 16 |
| 6. | 7. Mul | ticenter Studies | 16 |
| 6.8 | 8. Mul | tiple Comparisons/Multiplicity | 16 |
| 7. | STUDY | SUBJECTS | 17 |
| 7. | 1. Subj | ject Disposition | 17 |
| 7.2 | 2. Prot | ocol Deviations | 17 |
| 8. | IMMUN | OGENICITY EVALUATION | 18 |
| 8. | 1. Prin | nary Immunogenicity Analysis | 18 |
| 8.2 | 2. Seco | ondary Immunogenicity Analyses | 18 |
| 8.3 | 3. Exp | loratory Immunogenicity Analyses | 18 |
| | 8.3.1. | Covariate Analysis | 18 |
| | 8.3.2. | Regression Modeling | 19 |
| | 8.3.3. | Analysis of Heterologous Strains | 20 |
| | 8.3.4. | NA Serum Antibody Responses | 20 |
| 9. | SAFETY | Y EVALUATION | 21 |
| 9. | 1. Den | nographic and Other Baseline Characteristics | 21 |
| | 9.1.1. | Prior and Concurrent Illnesses and Medical Conditions | 21 |
| | 9.1.2. | Prior and Concurrent Medications | 21 |
| 9.2 | 2. Mea | surements of Treatment Compliance | 21 |

# TABLE OF CONTENTS (continued)

| 9.3. | . Adverse Events | | |
|---|---|---|---|
| 9 | .3.1. | Solicited Events and Symptoms | 22 |
| 9 | .3.2. | Unsolicited Adverse Events | |
| 9.4. | Deat | hs, Serious Adverse Events and other Significant Adverse Events | |
| 9.5. | | nancies | |
| 9.6. | _ | cal Laboratory Evaluations | |
| 9.7. | | Signs and Physical Evaluations | |
| 9.8. | | comitant Medications | |
| 10. RI | | TING CONVENTIONS | |
| | | CAL DETAILS | |
| | | RY OF CHANGES IN THE CONDUCT OF THE STUDY OR PLANNED | |
| Al | NALY | SES | 28 |
| 13. RI | EFERE | NCES | 29 |
| 14. Ap | pendi | ces | 30 |
| Append | lix 1. | Table Mock-Ups | 31 |
| Append | lix 2. | Figure Mock-Ups | 155 |
| Append | lix 3. | Listings Mock-Ups | 171 |

# LIST OF ABBREVIATIONS

| AE | Adverse Event |
|--------|--------------------------------------------------|
| ALT | Alanine Aminotransferase |
| BP | Blood Pressure |
| С | Celsius |
| CI | Confidence Interval |
| Cr | Creatinine |
| CRF | Case Report Form |
| CSR | Clinical Study Report |
| DMID | Division of Microbiology and Infectious Diseases |
| DSMB | Data and Safety Monitoring Board |
| eCRF | Electronic Case Report Form |
| ELISA | Enzyme-linked Immunosorbent Assay |
| ER | Emergency Room |
| F | Fahrenheit |
| FDA | U.S. Food and Drug Administration |
| GMT | Geometric Mean Titer |
| GSK | GlaxoSmithKline |
| HAI | hemagglutination inhibition antibody |
| Hgb | Hemoglobin |
| HHS | U.S. Department of Health and Human Services |
| ICH | International Conference on Harmonisation |
| IIV | Inactivated Influenza Vaccine |
| IM | Intramuscularly |
| IRB | Institutional Review Board |
| L | Liter |
| MAAE | Medically Attended Adverse Event |
| mcg | Microgram |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mg | Milligram |
| mITT | Modified Intention to Treat |
| N, n | Number |

# LIST OF ABBREVIATIONS (continued)

| NA | neuraminidase |
|---------|-----------------------------------------------|
| Neut | Neutralizing Antibody |
| NIH | National Institutes of Health |
| NOCMC | New Onset Chronic Medical Condition |
| PIMMC | Potentially Immune Mediated Medical Condition |
| PP | Per Protocol |
| PLT | Platelets |
| PT | Preferred Term |
| RCD | Reverse Cumulative Distribution |
| SAE | Serious Adverse Event |
| SD | Standard Deviation |
| SDCC | Statistical and Data Coordinating Center |
| SMC | Safety Monitoring Committee |
| SOC | System Organ Class |
| T. Bili | Total Bilirubin |
| WBC | White Blood Cell |
| WHO | World Health Organization |

### 1. PREFACE

This Statistical Analysis Plan (SAP) describes and expands upon the statistical information presented in the protocol.

This document describes all planned analyses and provides reasons and justifications for these analyses. It also includes sample tables, figures, listings (TFLs) planned for (1) expedited interim immunogenicity analyses, (2) final analyses included in the preliminary report, and (3) analyses included in the Clinical Study Report (CSR). Regarding the final analyses and CSR, this SAP follows the International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) Guidelines, as indicated in Topic E3 (Structure and Content of Clinical Study Reports), and more generally is consistent with Topic E8 (General Considerations for Clinical Trials) and Topic E9 (Statistical Principles for Clinical Trials). The structure and content of the SAP provides sufficient detail to meet the requirements identified by the FDA and ICH, while all work planned and reported for this SAP will follow internationally accepted guidelines published by the American Statistical Association and the Royal Statistical Society for statistical practice.

This document contains four sections: (1) a review of the study design, (2) general statistical considerations, (3) comprehensive statistical analysis methods for immunogenicity and safety outcomes, and (4) a list of proposed TFLs. Following any protocol amendment, this SAP will be reviewed and revised (if needed) to address any changes in the protocol impacting analysis. Any deviation from the final SAP will be described and justified in the CSR. The reader of this SAP is encouraged to also review the study protocol for details on conduct of the study and the operational aspects of clinical assessments.

### 2. INTRODUCTION

Since March of 2013 [1], avian influenza A/H7N9 viruses have continued to circulate in China causing discrete outbreaks (or waves) in humans with high mortality over the past 5 years. By late 2016, a fifth wave of outbreaks was identified in China and as of May 18, 2017, a total of 1,463 laboratory-confirmed human infections with avian influenza A/H7N9 virus have been reported by the World Health Organization [2, 3]. Since the onset of the fifth wave of H7N9 outbreaks in October 2016, more human cases of H7N9 infection have been reported in China than any prior H7N9 epidemic wave [3]. The U.S. Department of Health and Human Services (HHS) recently assessed H7N9 influenza virus as having a significant potential to cause a pandemic, and the greatest risk of causing severe disease. As a result, HHS has supported the production of fifth wave A/H7N9 inactivated influenza 9 vaccines (IIVs) for the U.S. stockpile and for an assessment of their safety and immunogenicity in clinical trials.

The goal of this clinical trial is to assess in healthy adults the safety, reactogenicity, and immunogenicity of two doses of a monovalent inactivated influenza A/H7N9 virus vaccine administered IM at different dosages given with or without AS03 adjuvant and to evaluate the potential of the dosage levels and adjuvant to enhance the immune response to the A/H7N9 vaccine. The two doses of the A/H7N9 vaccine given with or without AS03 adjuvant will be administered approximately 21 days apart.

### 2.1. Purpose of the Analyses

These analyses will assess the safety and immunogenicity of two doses of A/H7N9 IIV administered IM with or without AS03 adjuvant approximately 21 days apart and will be included in the clinical study report.

### 3. STUDY OBJECTIVES AND ENDPOINTS

### 3.1. Study Objectives

### 3.1.1. Primary

### Safety:

 To assess the safety and reactogenicity following receipt of two doses of 2017 H7N9 IIV administered IM at different dosages approximately 21 days apart given with or without AS03 adjuvant.

### Immunogenicity:

• To assess the serum hemagglutination inhibition (HAI) and neutralizing (Neut) antibody responses following receipt of two doses of 2017 H7N9 IIV administered IM at different dosages approximately 21 days apart with or without AS03 adjuvant, stratified by age of recipient.

### 3.1.2. Secondary

#### Safety:

- To assess unsolicited non-serious adverse events (AEs) following receipt of two
  doses of a 2017 H7N9 IIV administered IM at different dosages approximately 21
  days apart with or without AS03 adjuvant.
- To assess medically-attended adverse events (MAAEs) including new-onset chronic medical conditions (NOCMCs), potentially immune-mediated medical conditions (PIMMCs), and all serious adverse events (SAEs) following receipt of two doses of a 2017 H7N9 IIV administered IM at different dosages approximately 21 days apart with or without AS03 adjuvant.

### Immunogenicity:

• To assess the serum HAI and Neut antibody responses approximately 7 and 21 days following receipt of a single dose, and approximately 7 days following receipt of two doses of 2017 H7N9 IIV administered IM at different dosages approximately 21 days apart with or without AS03 adjuvant, stratified by age of recipient.

### **Exploratory**:

- To assess the effects of age, sex, body mass index, and prior receipt of seasonal influenza vaccine(s) on serum HAI and Neut antibody responses following receipt of two doses of a 2017 H7N9 IIV administered IM at different dosages approximately 21 days apart with or without AS03 adjuvant.
- To assess, in at least a subset of samples, the cross-reactivity of serum HAI and Neut antibody responses to antigenically drifted variants of influenza A/H7 viruses

following receipt of two doses of a 2017 H7N9 IIV administered IM at different dosages approximately 21 days apart with or without AS03 adjuvant, stratified by age of recipient.

- To assess the durability of serum HAI and Neut antibody responses at approximately 180 days following receipt of two doses of 2017 H7N9 IIV administered IM at different dosages approximately 21 days apart with or without AS03 adjuvant, stratified by age of recipient.
- To assess the neuraminidase (NA) content of the 2017 H7N9 IIV and determine the serum antibody responses to NA following receipt of 2017 H7N9 IIV. *Note: analysis plans for this objective will be described in an addendum to this SAP once the NA assay has been selected.*

# 3.2. Endpoints

### **3.2.1. Primary**

### Safety:

- Occurrence of study vaccine-related serious adverse events (SAEs) from the time of the first study vaccination through approximately 12 months after the last study vaccination.
- Occurrence of solicited injection site and systemic reactogenicity events from the time of each study vaccination through 7 days after each study vaccination.
- Occurrence of clinical safety laboratory adverse events from the time of each study vaccination through approximately 7 days after each study vaccination.

### Immunogenicity:

- For HAI and Neut antibodies, percentage of subjects achieving seroconversion against the influenza 2017 H7N9 study vaccine strain (defined as either a prevaccination titer <1:10 and a post-vaccination titer ≥1:40 or a pre-vaccination titer ≥1:10 and a minimum four-fold rise in post-vaccination titer) at approximately 21 days after the second study vaccination (Study Day 43).
- For HAI and Neut antibodies, percentage of subjects achieving titer ≥1:40 against the influenza 2017 H7N9 study vaccine strain at approximately 21 days after the second study vaccination (Study Day 43).
- Geometric Mean Titers (GMTs) of serum HAI and Neut antibodies against the influenza 2017 H7N9 vaccine strain at approximately 21 days after the second study vaccination (Study Day 43).

### 3.2.2. Secondary

### Safety:

- Occurrence of study vaccine-related unsolicited non-serious AEs from the time of each study vaccination through approximately 21 days after each study vaccination.
- Occurrence of all unsolicited adverse events, regardless of the assessment of seriousness or relatedness, from the time of each study vaccination through approximately 21 days after each study vaccination.
- Occurrence of MAAEs, including NOCMCs, and PIMMCs from the time of the first study vaccination through approximately 12 months after the last study vaccination.
- Occurrence of all serious adverse events (SAEs), regardless of the assessment of relatedness, from the time of the first vaccination through approximately 12 months after the last study vaccination.

### Immunogenicity:

- For HAI and Neut antibodies, percentage of subjects achieving seroconversion against the influenza 2017 H7N9 vaccine strain at approximately 7, 21, and 28 days after the first study vaccination (Study Days 8, 22, 29).
- For HAI and Neut antibodies, percentage of subjects achieving titers of 1:40 or greater against the influenza 2017 H7N9 vaccine strain at baseline and approximately 7, 21, and 28 days after the first study vaccination (Study Days 8, 22, 29).
- GMTs of serum HAI and Neut antibodies against the influenza 2017 H7N9 vaccine virus at baseline and approximately 7, 21, and 28 days after the first study vaccination (Study Days 8, 22, 29).

### 3.2.3. Exploratory

### Immunogenicity:

- For HAI and Neut antibodies, percentage of subjects achieving seroconversion and the GMTs of serum HAI antibody against the 2017 H7N9 study vaccine strain approximately 21 and 180 days after the second study vaccination (Study Days 43 and 202), stratified by age, sex, body mass index, and prior receipt of seasonal influenza vaccine(s).
- For HAI and Neut antibodies, for at least a subset of subjects, percentage achieving seroconversion, percentage with titer ≥1:40, and GMTs against antigenically drifted variants of influenza A/H7 viruses at baseline and approximately 21 and 180 days after the second study vaccination (Study Day 43 and 202).

- For HAI and Neut antibodies, percentage of subjects achieving seroconversion, percentage with titer ≥1:40, and GMTs against the 2017 H7N9 study vaccine strain at approximately 180 days after the second study vaccination (Study Day 202).
- Percentage of subjects with detectable levels of serum N9 NA specific antibody elicited by 2017 H7N9 vaccination, and the correlation of the NA content of 2017 H7N9 IIV with the elicited NA specific antibody responses at baseline and approximately 8 and 21 days after the first study vaccination (Study Day 1, 8 and 22) and 8, 21 and 180 days after the second study vaccination (Study Day, 29, 43 and 202). Note: analysis plans for this endpoint will be described in an addendum to this SAP once the NA assay has been selected.

# 3.3. Study Definitions and Derived Variables

For individual subjects, fold rise will be calculated as the ratio of:  $\frac{post-vaccination\ titer}{pre-vaccination\ titer}$ , where pre-vaccination value is always the result obtained at Day 1, prior to the priming vaccination.

HAI Seroconversion is defined as either a pre-vaccination HAI titer <10 and a post-vaccination HAI titer  $\ge 40$  or a pre-vaccination HAI titer  $\ge 10$  and a minimum four-fold rise in post-vaccination HAI titer [5].

Neut Seroconversion is defined as either a pre-vaccination Neut titer <1:10 and a post-vaccination Neut titer  $\ge 1:40$  or a pre-vaccination Neut titer  $\ge 1:10$  and a minimum four-fold rise in post-vaccination Neut antibody titer.

### 4. INVESTIGATIONAL PLAN

# 4.1. Overall Study Design and Plan

The protocol follows a Phase II randomized, double blind study design enrolling males and non-pregnant females aged 19 years and older who are in good health as determined by medical history and physical examination, and meet all eligibility criteria, including erythrocyte sedimentation rate (ESR), hematology, and biochemistry parameter within acceptable range, negative urine or serum pregnancy test (for females). This clinical trial is designed to assess the safety, reactogenicity, and immunogenicity of a monovalent inactivated influenza A/H7N9 virus vaccine at different dosages (3.75 mcg, 7.5 mcg, 15 mcg of HA per dose) with AS03 adjuvant, or at different dosages (15 mcg and 45 mcg of HA per dose) without adjuvant.

In this trial, subjects will be stratified by age (19-64 years or ≥65 years) then randomly assigned to 1 of 5 study groups with allocation 2:2:2:1:1 (see Table 1). The same dosage of vaccine with or without the same adjuvant will be given to subjects at both of their first and second study vaccinations. All study vaccinations will be administered IM approximately 21 days apart.

Reactogenicity will be measured by the occurrence of solicited injection site and systemic reactions from the time of each study vaccination through 7 days after each study vaccination. Unsolicited non-serious AEs will be collected from the time of each study vaccination through approximately 21 days after each study vaccination. SAEs, MAAEs, including NOCMCs, and PIMMCs, will be collected from the time of the first study vaccination through approximately 12 months after the last study vaccination. Clinical laboratory evaluations for safety will be performed on venous blood collected prior to each study vaccination and approximately 7 days after each study vaccination.

Immunogenicity testing will include performing HAI and Neut antibody assays against the 2017 A/H7N9 vaccine virus and drifted variants of the A/H7N9 virus on serum samples obtained immediately prior to each study vaccination (Days 1 and approximately Day 22), approximately 7 days after each study vaccination (Days 8 and 29), and approximately 21 and 180 days after the second study vaccination (Days 43 and 202).

Novel methods for identifying and assessing alternative correlates of protection against influenza infection are needed. To assess the NA specific antibody response to vaccination, it is first necessary to determine the NA content of inactivated influenza vaccine; this assay is under development. If successful, the NA content in a dosage specific manner can be correlated to the N9 NA-specific antibody responses elicited by the 2017 H7N9 IIV.

# **4.2.** Discussion of Study Design, Including the Choice of Control Groups

This study uses a dose comparison concurrent control design. All subjects receive the same study product (A/H7N9 IIV) with differing dosages with or without adjuvants.

## 4.3. Selection of Study Population

The study population for this clinical trial is 640 males and non-pregnant females (with over-enrollment up to 720 allowed), 19 years and older, who are in good health and meet all eligibility criteria. The subjects will be recruited from the general population at the participating Vaccine Trial and Evaluation Unit (VTEU) sites that have substantial experience conducting large influenza vaccine studies.

### 4.4. Treatments

#### 4.4.1. Treatments Administered

A/H7N9 Vaccine and AS03 Adjuvant will be administered.

### 4.4.2. Identity of Investigational Product

See the study protocol for details of study product formulation.

### 4.4.3. Method of Assigning Subjects to Treatment Groups (Randomization)

Enrollment/randomization will be performed through the enrollment module in the electronic data capture system maintained by the Statistical and Data Coordinating Center (SDCC).

Eligible subjects will be stratified by clinical site and age (19-64 years, ≥65 years) then randomly assigned with allocation (2:2:2:1:1) to one of 5 treatment arms indicated in Table 1. The treatment sequence was generated using permuted block randomization to provide an approximately balanced allocation to the treatment arms during the study.

### 4.4.4. Selection of Doses in the Study

Participants in this study are to receive two A/H7N9 vaccinations at HA doses of 3.75, 7.5, or 15 mcg with AS03 adjuvant, or at HA doses of 15 or 45 mcg without adjuvant. The 3.75, 7.5, or 15 mcg with AS03 doses are selected to evaluate safety and immunogenicity of antigen sparing dose strategies. Per FDA Guidance [5], the 15 mcg non-adjuvanted dose was selected to compare immune response with the 15 mcg adjuvanted vaccine. The 45 mcg non-adjuvanted dose is included to confirm the expected poor immunogenicity of non-adjuvanted vaccine at a high dose.

### 4.4.5. Selection and Timing of Dose for Each Subject

Each subject is to be randomly assigned to a study group which will define the A/H7N9 vaccine dose and receipt of adjuvant for both planned study vaccinations. The first vaccination takes place on the day of randomization, and the second vaccination takes place approximately 21 days after the first vaccination (protocol defined window of 21-28 days post first vaccination).

### 4.4.6. Blinding

This trial is double-blinded; subjects, investigators, study personnel performing any study-related assessments following study vaccine administration, and laboratory personnel performing antibody assays are blinded to dosage within study vaccination schedule.

The randomization scheme was generated by the SDCC and provided to unblinded study personnel (i.e., pharmacists performing study vaccination preparations and unblinded study vaccine administrators) at the participating VTEU sites who will not be not involved in study-related assessments or have subject contact for data collection following study vaccine administration.

The Data and Safety Monitoring Board (DSMB) may receive data in aggregate and presented by group. The DSMB may also be provided with expected and observed rates of the expected AEs in an unblinded fashion, and may request treatment assignment be unblinded for an individual subject if required for safety assessment. The DSMB will review grouped and unblinded data in the closed session only.

### 4.4.7. Prior and Concomitant Therapy

Administration of any medications, therapies, or vaccines (including prescription and over-the-counter drugs as well as herbals, vitamins, and supplements) from 60 days prior to study vaccination through 21 days post final vaccination will be solicited from the participant during screening, enrollment, and follow-up. Any reported prior therapies from up to 30 days prior to vaccination through 21 days post final vaccination will be recorded in the appropriate data collection form.

Use of concomitant medications is allowed prior to and during the trial with the exception of medications and therapies that might interfere with the evaluation of the investigational product. Medications in this category include the prohibited medication per the Subject Exclusion Criteria (protocol Section 5.1.2). In addition, the site principal investigator or appropriate sub-investigator may identify other medications that should not be used due to a risk to subject safety or assessment of reactogenicity and immunogenicity.

### 4.4.8. Treatment Compliance

All subjects were to receive two doses of study product administered in the clinic.

# 4.5. Immunogenicity and Safety Variables

See Table 2 and Table 3 for schedule of study procedures.

### 4.5.1. Safety Variables

Safety will be assessed by the frequency and severity of:

- 1. SAEs occurring from the time of the first study vaccination through approximately 12 months after the last study vaccination.
- 2. Solicited AEs reactogenicity events occurring from the time of each study vaccination through 7 days after each study vaccination:
  - a) Injection site reactions including pruritus, ecchymosis, erythema, induration/swelling, pain, and tenderness.
  - b) Systemic reactions including fever, feverishness, fatigue, malaise, myalgia, arthralgia, headache, and nausea.

- 3. Clinical safety laboratory AEs occurring from the time of each study vaccination through approximately 7 days after each study vaccination. Parameters to be evaluated include white blood cells (WBC), hemoglobin (Hgb), platelets (PLT), alanine aminotransferase (ALT), total bilirubin (T. Bili), and creatinine (Cr).
- 4. Unsolicited AEs non-serious AEs occurring from the time of each study vaccination through approximately 21 days after each study vaccination.
- 5. MAAEs, including NOCMCs, and PIMMCs occurring from the time of the first study vaccination through approximately 12 months after the last study vaccination.

Grading scales for injection site and systemic solicited reactions, vital signs, and clinical laboratory parameters are provided in Table 10, Table 11, Table 12, and Table 13.

### 4.5.2. Immunogenicity Variables

Individual HAI and Neut results will be reported by the central immunology laboratory for the homologous vaccine strain, A/Hong Kong/125/2017 (H7N9), and heterologous H7N9 strains (A/Shanghai/2/2013 and A/Guangdong/17SF003/2016). Assay results are reported as a reciprocal titer with values of  $10*2^k$ , where k=0, 1, 2, etc. The lower limit of detection for the HAI and Neut assays is 1:10; values below the limit of detection are imputed for analysis as one-half the limit of detection (10/2 = 5). For analysis, the geometric mean (calculated on natural log scale) of repeated results for each sample will be computed and used as the response for all subsequent calculations. The variation arising from multiple measurements for an individual at a single time point is not used in subsequent calculations. See Section 3.3 for definitions of derived variables for the analysis of HAI and Neut data.

The assay to determine the influenza virus N9 Neuraminidase (NA) antibody response to vaccination is under development. An addendum to the SAP will be generated to outline the planned analyses when assay development is complete.

All immunogenicity data will be uploaded into the SDCC's electronic data capture system.

### 5. SAMPLE SIZE CONSIDERATIONS

This study is planned to enroll a minimum of 160 subjects in each adjuvanted treatment arm (100 in 19-64 years age stratum, 60 in ≥65 years stratum), and 80 subjects in each unadjuvanted treatment arm (50 in 19-64 years age stratum, 30 in ≥65 years stratum). The sample size for this study was selected to obtain preliminary estimates in a time critical manner. While this study is not designed to test any specific null hypothesis, the following tables illustrate the precision and power that is available for select estimates and comparisons of interest.

Table 4 indicates the probability of observing one or more safety events, such as solicited injection site or systemic reactogenicity events or an unsolicited non-serious AE of a particular type for a single adjuvanted treatment arm/stratum (N = 60, or 100), for a single adjuvanted treatment arm combined over age strata (N=160), for all subjects receiving unadjuvanted vaccine (N = 160), and for all subjects receiving adjuvanted vaccine (N = 480).

Binomial confidence intervals (CI) are widest (have the least precision) when the response rate is 50%. Table 5 is presented to indicate the worst case scenario for precision of observed exact (Clopper-Pearson) binomial confidence intervals.

Table 6 illustrates the minimum detectable differences in the proportion of subjects responding (e.g., attaining seroconversion or a titer  $\ge 1:40$ ) between two adjuvanted treatment arms within each stratum using a two-sided Likelihood Ratio Test and alpha = 0.05.

Over enrollment is allowed, to ensure a minimum of n=100 per adjuvanted treatment arm in the 19-64 years age stratum, therefore power calculations for this stratum assume n=100 per group. Based on previous DMID A/H7N9 trials it is expected 5% of enrolled subjects in this stratum may be excluded from analysis of the primary endpoint. In the event that only 100 subjects are actually enrolled in a treatment arm, the small dropout rates anticipated would have a minimal impact on the calculations presented in Table 7.

Within the ≥65 years treatment arm a dropout rate of up to 12% is expected based on previous DMID trials in this population, so a minimum of 60 subjects are planned to enroll in each adjuvanted treatment arm to ensure at least 50 are available for analysis of the primary immunogenicity endpoint.

Per FDA guidance [5,6], for differences in HAI antibody response rates, the lower confidence limit on the appropriate point estimate excluding equality (i.e., 0 for the difference parameter) may be sufficient to demonstrate the added value of the adjuvant. Table 8 and Table 9 show the lower bound of the 95% confidence interval for the difference in the proportion of responders between the adjuvanted and unadjuvanted arms (e.g., 15 mcg + AS03 minus 45 mcg unadjuvanted) assuming the proportion of responders in the unadjuvanted arm is 0.10 and considering a range for the proportion of responders in the adjuvanted arm ranges from 0.50 to 0.90.

### 6. GENERAL STATISTICAL CONSIDERATIONS

# **6.1.** General Principles

All continuous variables will be summarized using the following descriptive statistics: n (non-missing sample size), mean, standard deviation, median, maximum and minimum. The frequency and percentages (based on the non-missing sample size) of observed levels will be reported for all categorical measures. In general, all data will be listed, sorted by site, treatment and subject, and when appropriate by visit number within subject. All summary tables will be structured with a column for each treatment arm in the following order:

- Group 1: 3.75 mcg A/H7N9 + AS03
- Group 2: 7.5 mcg A/H7N9 + AS03
- Group 3: 15 mcg A/H7N9 + AS03
- Group 4: 15 mcg A/H7N9
- Group 5: 45 mcg A/H7N9

Additional tables structured with a column for each age stratum (19-64,  $\geq$ 65) within treatment arm will be provided. All tables will be annotated with the total population size relevant to that table/treatment, including any missing observations.

# **6.2.** Timing of Analyses

#### **6.2.1.** Expedited Interim Immunogenicity Reports

A series of Expedited Interim Immunogenicity Reports of HAI and Neut serum antibody responses comparing venous blood samples collected at baseline (D1), Visit 03 (D8), Visit 06 (D29), and Visit 07 (D43) is planned. Reports will include HAI and Neut results for approximately 25 subjects per adjuvanted treatment arm and 13 subjects per unadjuvanted treatment arm within the 19-64 year-old stratum and the first 15 subjects per adjuvanted treatment arm and 8 subjects per unadjuvanted treatment arm within the ≥65 year-old stratum. Reports will be prepared following each post-vaccination visit with analyses as described in Section 6.6.2. This information will be reviewed due to the extraordinary need to inform public health decision makers in their preparations for their response to a potential A/H7N9 pandemic. These data will be archived by the SDCC, but will not be part of the final clinical database for this study, nor will they be made available to the clinical investigators for publication.

Expedited Immunogenicity Reports will be provided by the SDCC per the study Communication Plan. Reports will include data summarized by unblinded treatment arm, but the presentation will be in a format that prevents inadvertent unblinding of any individual subject.

Tables and figures to be included in the Expedited Immunogenicity Report are indicated with the symbol † in the title.

### 6.2.2. Preliminary Report and CSR

Clinical, safety, and reactogenicity data through approximately 180 days after the second study vaccination will represent the primary clinical database for this trial. Once the last subject completes the visit that occurs approximately 180 days after the last study vaccination, the primary clinical database will be cleaned, monitored, and locked, and all serum samples will be sent for HAI and Neut antibody assays. Unblinded analyses of safety, reactogenicity, and available immunogenicity data (HAI and Neut antibody assays through Day 202) are planned. A preliminary report may be prepared by the SDCC after the primary clinical database is locked and all HAI and Neut data through 180 days after the last study vaccination are received. Regardless of whether a preliminary report is prepared, a "topline" set of the immunogenicity tables will be provided to DMID on an expedited timeline following laboratory database lock. These analyses may be made available to the sponsor for planning subsequent trials and to the lead principal investigator for publication. These analyses will not be used to make any decisions concerning the conduct of this trial. As it is anticipated that subjects will remain in long term safety follow-up at the time of these analyses, blinded investigators and DMID medical monitors not involved in the analysis, publication, or clinical study report preparation will be responsible for assessing SAEs and MAAEs including PIMMCs and new onset chronic medical conditions until all subjects have completed the final follow-up visit. All analyses of data included in the preliminary report for early release will be considered the final analysis of these data, and also included in the final CSR.

Tables and figures to be included in the Preliminary Report are indicated with the symbol \* in the title. Topline tables to be generated after laboratory database lock are indicated with the symbol ‡ in the title.

Analysis of exploratory immunogenicity endpoints may be performed and released as the data are available from the research laboratory. Any such analyses would be considered the final analysis for the endpoint and included in the CSR.

The final CSR will be completed after the last subject's last visit is completed, and the final clinical database including all long-term safety follow-up data is cleaned, monitored and locked. Additional exploratory immunogenicity endpoint data not available at the time of CSR preparation may be included in an addendum to the CSR.

## 6.3. Analysis Populations

### **6.3.1.** Safety Population

The Safety Analysis population includes all subjects who received at least one study vaccination.

#### 6.3.2. Modified Intention-to-Treat (mITT) Population

The modified intent-to-treat (mITT) population includes all subjects who received at least one study vaccination and contributed both pre- and at least one post-study vaccination venous blood samples for immunogenicity testing (HAI or Neut antibody assays) for which valid results were reported. For analyses using the mITT population, subjects will be grouped based on randomized treatment arm.

### **6.3.3.** Per Protocol Population

The per protocol (PP) population includes all subjects in the mITT subset with the following exclusions:

- Data from all available visits for subjects found to be ineligible at baseline due to eligibility criteria that would impact immune response.
- Data from all visits subsequent to major protocol deviations, such as:
  - o Second study vaccination not received,
  - Second study vaccination received out of window,
  - Receipt of non-study licensed live vaccine within 30 days before or after each study vaccination,
  - Receipt of non-study licensed inactivated vaccine within 14 days before or after each study vaccination,
  - Receipt of immunosuppressive therapy (e.g., corticosteroids) within 30 days before or after each study vaccination.
- Data from any visit that occurs out of window by more than one day:
  - O Visit 3 data collected before 6 days or after 10 days post first study vaccination
  - o Visit 4 data collected before 20 days or after 29 days post first study vaccination.
  - o Visit 6 data collected before 6 days or after 10 days post second study vaccination.
    - o For subjects who did not receive the second study vaccination, visit 6 data collected before 27 days or after 31 days post first study vaccination.
  - o Visit 7 data collected before 20 days or after 29 days post second study vaccination.
    - o For subjects who did not receive the second study vaccination, visit 7 data collected before 41 days or after 50 days post first study vaccination.
  - Visit 10 data collected before 165 days or after 195 days post second study vaccination.
    - o For subjects who did not receive the second study vaccination, visit 10 data collected before 200 days or after 216 days post first study vaccination.

For analyses using the PP population, subjects will be grouped based on study vaccinations received.

# **6.4.** Covariates and Subgroups

As a protocol defined exploratory analysis, HAI antibody response following the second vaccination will be summarized stratified by the following covariates: age (categorical: 19-34, 35-49, 50-64, 65-80,  $\geq$ 80), sex (male, female), body mass index ( $\leq$ 30,  $\geq$ 30), and prior

receipt of seasonal influenza vaccine(s) (neither 2016-2017 nor 2017-2018, 2016-2017 only, 2017-2018 only, both 2016-2017 and 2017-2018, unknown), and these covariates will be considered in statistical modeling as described in Section 8.3. As these analyses are exploratory the study was not powered for any subgroup analyses.

### 6.5. Missing Data

All attempts will be made to collect all data per protocol. As missing data are expected to be minimal, no imputation will be performed for missing values. Any data point that appears to be erroneous or inexplicable based on clinical judgment will be investigated as a possible outlier. If data points are identified as outliers, sensitivity analyses will be performed to examine the impact of including or excluding the outliers. Any substantive differences in these analyses will be reported.

# 6.6. Interim Analyses and Data Monitoring

Interim analyses will only be used to terminate this trial in the event that unanticipated safety events deemed to be of sufficient concern require such action by the sponsor. These assessments will not be made on the basis of testing a formal statistical hypothesis; therefore, p-value adjustment will not be made to any analyses. A DSMB will be convened by DMID to review study progress and participant, clinical, safety, and reactogenicity and immunogenicity data.

An interim analysis of immunogenicity is planned, as described in section 6.2 which includes a series of Expedited Interim Immunogenicity Reports of serum HAI and Neut antibody responses. This information will be reviewed due to the extraordinary need to inform public health decision makers in their preparations for their response to a potential 2017 A/H7N9 pandemic. Although interim immunogenicity results will not be used to make decisions concerning the conduct of this trial, they may be used to make decisions on activities external to this trial, e.g., designing future trials of the 2017 H7N9 IIV with and without AS03 adjuvant in other age groups.

Additionally, a preliminary report of safety and immunogenicity data through Day 43 will be prepared as described in section protocol section 11.6; though this report will be released while subjects remain in the trial for long-term safety and immunogenicity follow-up, it will be considered the final analysis of these data.

Emergent public health needs may dictate additional interim safety, reactogenicity, and/or immunogenicity analyses be performed on available information at any time during the trial. If this occurs, immunogenicity data will be analyzed as results are available from the central immunogenicity laboratory.

#### **6.6.1. Interim Safety Review**

An interim safety review may include enrollment and demographic information, medical history, concomitant medications, physical assessments, clinical laboratory values, dosing compliance, and solicited and unsolicited AE/SAEs. Additional data may be requested by the DSMB, and interim statistical reports may be generated as deemed necessary and appropriate by DMID. The DSMB may receive data in aggregate and presented by treatment arm. The

DSMB may also be provided with expected and observed rates of the expected AEs in an unblinded fashion, and may request the treatment assignment be unblinded for an individual subject if required for safety assessment. The DSMB will review grouped and unblinded data in the closed session only. The DSMB will meet and review this data at scheduled time points or ad hoc as needed during this trial as defined in the DSMB charter. As an outcome of each review/meeting, the DSMB will make a recommendation as to the advisability of proceeding with study vaccinations (as applicable), and to continue, modify, or terminate this trial. Summaries prepared for the DSMB are defined separately in a report shell reviewed and approved by the DSMB.

Additionally, this trial will be monitored to determine if any of the halting rules described in Protocol Section 9.5 are met.

### 6.6.2. Interim Immunogenicity Review

There is no plan to halt this trial prior to full enrollment and completion of all follow-up visits based on interim immunogenicity results. A series of Expedited Interim Immunogenicity Reports of HAI and Neut serum antibody responses will be generated as described in Section 6.2.

Immune responses will be summarized in terms of strain-specific 2017 A/H7N9 HAI and Neut antibody titers and the relationship to study vaccine dosage and adjuvant use. It is anticipated that all analyses will be carried out in parallel for both assays, but reports may be prepared separately for HAI and Neuts if results are available on different timelines. Interim analyses will focus on rates of titers ≥1:40, seroconversion (defined as either a prevaccination titer <1:10 and a post-vaccination titer ≥1:40 or a pre-vaccination titer ≥1:10 and a minimum four-fold rise in post-vaccination titer) GMTs, along with corresponding 95% confidence intervals. No formal hypothesis testing will be included in the interim analysis. All interim analyses will use the mITT population.

Tables and figures to be included in in the Expedited Interim Immunogenicity Reports are indicated with the symbol † in the title. These include Table 29 and Table 31 presenting summaries and 95% CIs of HAI and Neut antibodies respectively by treatment arm, Table 33 and Table 35 presenting summaries and 95% CIs of HAI and Neut antibodies respectively by treatment arm and age stratum.

### 6.7. Multicenter Studies

Although randomization was stratified by site, data will be pooled across all clinical sites for all analyses. Center effects are not anticipated because the sites are using standardized procedures for vaccination and assessment of solicited and unsolicited AEs, and the study relies on a central laboratory for immunogenicity assessments.

# 6.8. Multiple Comparisons/Multiplicity

This study was designed to obtain preliminary estimates of safety and immune response to the A/H7N9 vaccination in healthy adults. The study was not designed to test any specific null hypothesis, and as such no adjustment for multiple comparisons will be performed.

### 7. STUDY SUBJECTS

# 7.1. Subject Disposition

Table 14 will present a summary of the reasons that subjects were screened but not enrolled.

The number and percentage of enrolled subjects excluded from each analysis population by treatment arm and age stratum, are presented in Table 15 and Table 16. A listing of subjects excluded from each analysis population will be presented in Listing 5.

The disposition of subjects in the study will be tabulated by treatment arm and age stratum (Table 17 and Table 18). The table will show the total number of subjects screened, randomized, receiving the first study vaccination, receiving the second study vaccination, completing the blood draw for the primary immunogenicity endpoints, and completing the last visit.

A flowchart showing the disposition of study subjects, adapted from the CONSORT Statement [4] will be included and will present the number of subjects screened, randomized, lost to follow up, and analyzed, by treatment arm (Figure 1).

A listing of subjects who were discontinued from treatment or terminated from study followup and the reason will be included in <u>Listing 2</u>.

### 7.2. Protocol Deviations

A summary of subject-specific protocol deviations will be presented by the deviation category and deviation type, treatment arm, and age stratum for all enrolled subjects (Table 9). Major deviations that will be reviewed for possible exclusion of immunogenicity results from the PP population include deviations related to eligibility/enrollment, treatment administration schedule, follow-up visit schedule, and receipt of exclusionary vaccines or medications. All subject-specific protocol deviations and non subject-specific protocol deviations will be included in Listing 3 and Listing 4.

### 8. IMMUNOGENICITY EVALUATION

Immunogenicity data summaries and analysis for primary and secondary endpoints will be presented for the mITT and PP populations. Immune responses in terms of strain-specific A/H7N9 HAI and Neut antibody titers will be summarized by treatment arm and age stratum at each time point. Descriptive summary statistics will be provided for all assays and time points including number of subjects with non-missing results, percentage of subjects with titers ≥1:40, percentage of subjects achieving seroconversion, and GMTs along with corresponding 95% CI. Exact confidence intervals will be presented for proportional endpoints. Summaries of primary and secondary immunogenicity endpoints are presented in Table 29, Table 30, Table 31, Table 32, Table 33, Table 34, Table 35, and Table 36.

RCD curves will be presented for post-vaccination HAI and Neut antibody titers. Plots for each assay will be generated with 4 panels (8 days post vaccination 1, 21 days post vaccination 1, 8 days post vaccination 2, 21 days post vaccination 2, and 180 days post vaccination 2), and separate curves within each panel for each treatment arm and age stratum, as shown in Figure 2, Figure 3, Figure 4, and Figure 5.

Figures depicting the HAI and Neut GMT over time will also be presented as shown in Figure 6, Figure 7, Figure 8, and Figure 9.

The spearman correlation between HAI, Neut, and Neuraminidase antibody titers will be calculated at each time point over all groups. The correlation will be depicted in scatter plots as Figure 10 and Figure 11.

Individual HAI and Neut assay results will be provided in Listing 8.

## 8.1. Primary Immunogenicity Analysis

The primary immunogenicity endpoints HAI and Neut seroconversion, percentage of subjects with titer ≥1:40, and GMTs against the homologous A/H7N9 vaccine strain 21 days after the second vaccination will be summarized as described above. Regression modelling of seroconversion and log titers is planned as described in Section 8.3.2.

# 8.2. Secondary Immunogenicity Analyses

The primary immunogenicity endpoints HAI and Neut seroconversion, percentage of subjects with titer ≥40, and GMTs against the homologous A/H7N9 vaccine strain 8 and 21 days after the first vaccination and 8 days after the second vaccination will be summarized as described above. No formal hypothesis testing is planned.

# 8.3. Exploratory Immunogenicity Analyses

Immunogenicity data summaries and analysis for exploratory endpoints will be presented for the PP populations.

### 8.3.1. Covariate Analysis

As an exploratory analysis, seroconversion and GMT of serum antibody for both HAI and Neut at 21 and 180 days after second vaccination will be summarized by treatment arm stratified by age (categorized as those subjects ages 19-34, 34-49, 50-64, 65-80, and ≥81

years) (Table 37, Table 38, Table 39, and Table 40), by sex (Table 41, Table 42, Table 43, and Table 44), by BMI (Table 45, Table 46, Table 47, and Table 48), and by prior receipt of seasonal influenza vaccines (Table 49, Table 50, Table 51, and Table 52). These stratified summaries will be presented for the PP population. It is anticipated that subjects will have little to no pre-existing antibody at baseline, so seroconversion and titer  $\geq$  40 endpoints will be similar.

### **8.3.2.** Regression Modeling

Logistic and multivariate linear regression will be utilized to test for the effects of the HA antigen dose and the AS03 adjuvant on seroconversion and GMT, respectively, for the PP population. Similar models will be fit for HAI and Neut Antibodies. Separate models will be fit for data from Day 21 post dose 2 and Day 180 post dose 2.

Logistic regression will be fit to examine the relationship of HAI seroconversion at 21 days after the 2<sup>nd</sup> study vaccination with treatment group and age strata (19-64 years, ≥65 years). If the available titer data meets the required assumptions of normality after log transformation, multiple linear regression will be fit to examine the relationship of log transformed titers at 21 days after the 2<sup>nd</sup> study vaccination with treatment arm and age strata (19-64 years, ≥65 years). Both models will be fit with and without adjustment for the following covariates (*Z*): sex (female, male), BMI (<30, ≥30), and prior receipt of seasonal influenza vaccine (none in past 2 seasons, at least once in past 2 seasons). Modeling assumptions will be checked using standard diagnostic methods (e.g., using the INFLUENCE option in PROC LOGISTIC or PROC GLM). Parameter estimates and odds ratio estimates for the logistic models will be presented in Table 53, Table 54, Table 55, Table 56, Table 57, Table 58, Table 59, and Table 60. Parameter estimates for the multiple linear regression models will be presented in Table 61, Table 62, Table 63, Table 64, Table 65, Table 66, Table 67, and Table 68.

Model 1A: Logistic Regression (without covariate adjustment):

$$logit[P(seroconversion)] = \beta_0 + \beta_1 \times Treatment + \beta_2 (Age \ge 65) + \varepsilon$$

Model 1B: Logistic Regression (with covariate adjustment):

$$logit[P(seroconversion)] = \beta_0 + \beta_1 \times Treatment + \beta_2 (Age \ge 65) + \beta_3 \times Z + \varepsilon$$

Model 2A: Multiple Linear Regression (without covariate adjustment):

$$log(titer) = \beta_0 + \beta_1 \times Treatment + \beta_2(Age \ge 65) + \varepsilon$$

Model 2B: Multiple Linear Regression (with covariate adjustment):

$$log(titer) = \beta_0 + \beta_1 \times Treatment + \beta_2(Age \ge 65) + \beta_3 \times Z + \varepsilon$$

Subjects missing data for one or more covariates will be excluded from Models 1B and 2B.

Models 1B and 2B, defined above, will also be fit for HAI at Day 21 replacing the binary age strata variable with age in years (continuous). The models as shown below assume a linear relationship between age in years and both probability of seroconversion and GMT. The validity of this assumption will be assessed prior to analysis and, if the relationship between age and response is found to be non-linear, adjustments will be made to model parameters to

satisfy regression assumptions. The results of these models will be presented in Table 69 and Table 70.

Model 3: Logistic Regression (with covariate adjustment):

$$logit[P(seroconversion)] = \beta_0 + \beta_1 \times Treatment + \beta_2 (Age in Years) + \beta_3 \times Z + \varepsilon$$

Model 4: Multiple Linear Regression (with covariate adjustment):

$$log(titer) = \beta_0 + \beta_1 \times Treatment + \beta_2(Age\ in\ Years) + \beta_3 \times Z + \varepsilon$$

Subjects missing data for one or more covariates will be excluded from Models 3 and 4.

### 8.3.3. Analysis of Heterologous Strains

HAI and Neut antibody responses against antigenically drifted variants of influenza A/H7 viruses (A/Shanghai/2/2013 and A/Guangdong/17SF003/2016) will be summarized for the Per Protocol population as described in Section 8 (Table 71 and Table 72; Figure 12, Figure 13, Figure 14, Figure 15, and Figure 16). A scatter plot of the correlation between response to the vaccine strain and each heterologous strain will be presented (Figure 17 and Figure 18). No formal hypothesis testing or modeling for the exploratory analysis of heterologous strains is planned.

### 8.3.4. NA Serum Antibody Responses

Descriptions of the NA assays and planned analyses will be described in an addendum to this SAP.

#### 9. SAFETY EVALUATION

All summaries and analysis of safety data will be presented for the Safety Analysis Population. Safety summaries will be presented overall and grouped by treatment arm overall and by age stratum.

Continuous variables will be summarized using the following descriptive statistics: n (non-missing sample size), mean, standard deviation, median, maximum and minimum. All categorical measures will be summarized by the frequency and percentages of observed levels. The denominator for the percentages may be based on the number of non-missing observations for an assessment or based on the number of subjects in a population. This will be described for each table.

### 9.1. Demographic and Other Baseline Characteristics

Summaries of age, sex, ethnicity, race, BMI, and prior receipt of seasonal influenza vaccine will be presented by site (Table 21 and Table 22) and by treatment arm overall and by age stratum (Table 23, Table 24, Table 25, and Table 26). Age will be summarized as a continuous variable as well as by strata categories. Ethnicity is categorized as Hispanic or Latino, or not Hispanic and not Latino. In accordance with NIH reporting policy, subjects may self-designate as belonging to more than one race or may refuse to identify a race, the latter reflected in the electronic case report form (eCRF) as "No" to each racial option. BMI will be summarized as a continuous as well as categorical variable, categorized as (<30, ≥30). Self-reported history of prior receipt of seasonal influenza vaccine will be categorized as follows: neither 2016-2017 and 2017-2018, 2016-2017 only, 2017-2018 only, both 2016-2017 and 2017-2018, or unknown. Demographic information for individual subjects will be provided in Listing 6.

### 9.1.1. Prior and Concurrent Illnesses and Medical Conditions

All current illnesses and past or pre-existing medical conditions will be coded using Medical Dictionary for Regulatory Activities (MedDRA®) version 20.0 or higher.

Summaries of subjects' prior and concurrent medical conditions will be presented by treatment arm (Table 27 and Table 28).

Individual subject listings will be presented for all reported medical history including prior and concurrent medical conditions (Listing 7).

### 9.1.2. Prior and Concurrent Medications

Concomitant medications will be coded to the Anatomical Therapeutic Classification using the WHO Drug Dictionary. The use of concomitant medications during the study will be summarized by ATC1 and ATC2 code and treatment arm for the Safety population (Table 131 and Table 132). A listing of concomitant medications will be presented (Listing 16).

# 9.2. Measurements of Treatment Compliance

All subjects are to receive 2 study vaccinations administered in the clinic. The number of study vaccinations administered to subjects will be presented by treatment arm and by site,

overall and by age stratum in Table 19 and Table 20 and as part of the subject disposition tables (Table 17 and Table 18). Listing 1 presents subjects who received investigational product with randomized treatment arm and study product received for each vaccination.

### 9.3. Adverse Events

A summary of all adverse events is provided in Table 73. A summary of those events that occurred in  $\geq$ 5% of subjects in any treatment group is provided in Table 74.

### 9.3.1. Solicited Events and Symptoms

Systemic solicited adverse events were collected pre-vaccination, and systemic and local solicited adverse events were collected at-least 20 minutes post-vaccination and then daily for 7 days after each vaccination and graded on a scale of 0 (absent), 1 (mild), 2 (moderate) and 3 (severe). Systemic events include fever, feverishness, fatigue, malaise, myalgia, arthralgia, headache, and nausea. The grading scale for systemic events, including quantitative grading for fever, is included in Table 11. Local events include pruritus, ecchymosis, erythema, induration/swelling, pain, and tenderness. Ecchymosis, erythema, and induration are measured by both functional and measurement grading scales as defined in Table 10.

When calculating the incidence of solicited events, each subject will be counted once at the highest severity following the applicable vaccination, and any repetitions will be ignored. For summaries presented separately for each vaccination, the denominator for percentages will be the number of subjects who received the respective vaccination with non-missing data for the event summarized. For summaries over all vaccinations the denominator will be the number of subjects who received at least one vaccination with non-missing data for the event summarized.

The number and percentage of subjects reporting at least one solicited adverse event of any severity will be summarized for each solicited symptom, any systemic symptom, any local symptom, and any symptoms. For each event the denominator is the number of subjects who received the applicable vaccination with non-missing data for the specific event. The 95% CI calculated using Clopper-Pearson methodology from a binomial distribution (SAS Proc Freq with a binomial option) will be presented (Table 75, Table 76, Table 77, Table 78, Table 79, and Table 80). Logistic regression models will be fit to estimate the effect of treatment and age on the probability of reporting any local event or reporting any systemic event (Table 81 and Table 82). If statistically significant effects are observed in the model for local events or systemic events, then additional models will be fit for each individual event of that type.

$$logit[P(Event)] = \beta_0 + \beta_1 \times Treatment + \beta_2 (Age \ge 65) + \varepsilon,$$

For each systemic and local event, any systemic event, any local event, and any solicited event, the maximum severity over 7 days after each vaccination will be summarized for the Safety population. The number and percentage of subjects reporting each event will be summarized by the maximum severity and treatment group overall and by age stratum, separately for each vaccination and over all vaccinations. For each event the denominator is the number of subjects who received the applicable vaccination with non-missing data for the specific event. The 95% CI calculated using Clopper-Pearson methodology from a binomial

distribution (SAS Proc Freq with a binomial option) will be presented (Table 83, Table 84, Table 85, Table 86, Table 87, and Table 88).

The number of subjects reporting a solicited adverse event will be summarized for each day post vaccination for each vaccination and for all vaccinations combined both in a summary table (Table 89, Table 90, and Table 91) and graphically in a bar chart (Figure 19 and Figure 20). A comparison of the event rate for each treatment group between vaccination 1 and vaccination 2 will be presented, including p-values from McNemar's test performed within each age stratum and over all subject (Table 92 and Table 93).

Systemic and Local solicited events reported by subject will be presented in Listing 9 and Listing 10, sorted by subject ID, vaccination number, parameter, and study day.

### 9.3.2. Unsolicited Adverse Events

When calculating the incidence of unsolicited AEs (i.e., on a per subject basis), each subject will only be counted once at the highest severity and/or relationship, and any repetitions of AEs within a subject will be ignored; the denominator will be the total number of subjects in the safety population. All AEs reported will be included in the summaries and analyses.

The number and percentage of subjects reporting at least one unsolicited AE will be summarized by MedDRA system organ class and preferred term. A 95% CI will be presented for the percentage of subjects reporting any unsolicited AE (serious or non-serious) for each MedDRA system organ class and preferred term over all study vaccinations (Table 94 and Table 95).

The following summaries for unsolicited AEs will be presented by MedDRA system organ class, preferred term, and treatment arm:

- Incidence of AEs by severity and relationship to study product (Table 96);
- Incidence of non-serious, related AEs by severity (Table 97);
- Incidence of AEs over time (Days 1-8, Days 9-22 post each study vaccination) (Table 98);
- Incidence of non-serious, related AEs over time (Days 1-8, Days 9-22 post each study vaccination) (Table 99) note this table presents results for secondary safety endpoint, "Occurrence of study vaccine-related unsolicited non-serious AEs from the time of each study vaccination through approximately 21 days after each study vaccination";
- Total frequency of AEs over time (Days 1-8, Days 9-22 post each study vaccination) (Table 100);
- Subject listing of non-serious AEs of moderate or greater severity (Table 104);
- Bar chart displaying total frequency of AEs by severity and MedDRA system organ class, Treatment Arm, and Age Stratum (Figure 21);

- Bar chart displaying incidence of AEs by severity and MedDRA system organ class, Treatment Arm, and Age Stratum (Figure 22);
- Bar chart displaying total frequency and incidence of AEs by relationship to study product and MedDRA system organ class, Treatment Arm and Age Stratum (Figure 23 and Figure 24).

# 9.4. Deaths, Serious Adverse Events and other Significant Adverse Events

The following listings will be presented including Subject ID, Age (years) AE Description, AE Onset Date/End Date, Last Vaccination Received/Days Post Vaccination, Reason Reported as an SAE, Relationship to Treatment, Alternate Etiology if not Related, Outcome, and Duration of Event (days):

- Deaths and Serious Adverse Events (Table 101);
- Adverse Events of Special Interest (Table 102);
- New Onset Chronic Medical Conditions (Table 103).

A listing of all reported AEs by subject will be presented in Listing 11, sorted by Treatment Arm, Age Stratum, Subject ID, and AE Number.

## 9.5. Pregnancies

For any subjects in the Safety population who became pregnant during the study, every attempt will be made to follow these subjects to completion of pregnancy to document the outcome, including information regarding any complications with pregnancy and/or delivery. Listing 17, Listing 18, Listing 19, Listing 20, and Listing 21 will present any study pregnancies and their outcomes.

# 9.6. Clinical Laboratory Evaluations

Clinical safety laboratory parameters (WBC, Hgb, PLT, ALT, T. Bili, Cr) will be collected from each subject prior to each study vaccination and approximately 7 days after each study vaccination. These evaluations will be performed by the central clinical laboratory. The grading scale for clinical laboratory evaluations is presented in Table 13. Clinical laboratory evaluations assessed on Day 1 prior to the first study vaccination will be considered as baseline.

The distribution of laboratory results by severity, study day, treatment arm and age stratum will be presented in Table 105, Table 106, Table 107, Table 108, Table 109, Table 110, and Table 111. Descriptive statistics including mean, standard deviation, median, minimum and maximum values by study day will be summarized for each parameter in Table 112, Table 113, Table 114, Table 115, Table 116, and Table 117, and for the change from baseline for each parameter in Table 118, Table 119, Table 120, Table 121, Table 122, and Table 123. Box plots illustrating the change from baseline for each laboratory parameter will be presented in Figure 25, Figure 26, Figure 27, Figure 28, Figure 29, and Figure 30. Subject

visits with abnormal laboratory results, Grade 1 severity or higher, will be presented in Table 124 and Table 125 for Chemistry and Hematology parameters, respectively.

A complete listing of individual clinical laboratory results will be presented in Listing 12 and Listing 13 for chemistry and hematology, respectively, sorted by subject ID, parameter, and visit number.

## 9.7. Vital Signs and Physical Evaluations

Vital signs oral temperature, systolic blood pressure, diastolic blood pressure, and pulse will be assessed prior to study vaccination on Day 1 and Day 22. The grading scale for vital sign evaluations is presented in Table 12. Summaries of vital signs by maximum severity will be tabulated by visit, treatment arm, and age stratum (Table 126, Table 127, Table 128, Table 129, and Table 130). A listing of vital signs will be presented (Listing 14).

Targeted physical examinations will be performed, if indicated, based on a subject's medical history. A listing of physical exam findings will be presented (Listing 15).

### 9.8. Concomitant Medications

Concomitant medications will be collected for the 30 days prior to the first study vaccination through 21 days after the second study vaccination. Concomitant medications will be coded to the Anatomical Therapeutic Classification using the WHO Drug Dictionary. The use of prior and concomitant medications taken during the study will be recorded on the CRFs. A by-subject listing of concomitant medication use will be presented (Listing 16). The use of concomitant medications during the study will be summarized by ATC1, ATC2 code, treatment arm and age stratum for the Safety population (Table 131 and Table 132).

### 10. REPORTING CONVENTIONS

P-values ≥0.001 and ≤0.999 will be reported to 3 decimal places; p-values less than 0.001 will be reported as "<0.001"; p-values greater than 0.999 will be reported as "> 0.999". The mean, standard deviation, and any other statistics other than quantiles, will be reported to one decimal place greater than the original data. Quantiles, such as median, or minimum and maximum will use the same number of decimal places as the original data. Proportions will be presented as two decimal places; values <0.01 will be presented as "<0.01". Percentages will be reported to the nearest whole number; non-zero values < 1% will be presented as "<1"; values greater than 99% but less than 100% will be presented as >99. Estimated parameters, not on the same scale as raw observations (e.g. regression coefficients) will be reported to 3 significant figures.

# 11. TECHNICAL DETAILS

SAS version 9.4 or above will be used to generate all tables, figures and listings.

# 12. SUMMARY OF CHANGES IN THE CONDUCT OF THE STUDY OR PLANNED ANALYSES

This SAP does not include any changes from the analyses described in the protocol.

### 13. REFERENCES

- 1. Gao, R., et al., *Human infection with a novel avian-origin influenza A (H7N9) virus*. N Engl J Med, 2013. **368**(20): p. 1888-97.
- 2. Analysis of recent scientific information on avian influenza A(H7N9) virus. WHO Influenza Update, 2017.
- 3. Human infection with avian influenza A(H7N9) virus China: 18 May 2017. WHO Emergencies preparedness, response, 2017.
- 4. Drummond R. CONSORT Revised: Improving the Reporting of Randomized Clinical Trials. JAMA. 2001; 285(15):2006-2007.
- 5. FDA Guidance for Industry: Clinical Data Needed to Support the Licensure of Seasonal Inactivated Influenza Vaccines (US DHHS, FDA, CBER, May 2007).
- 6. FDA Guidance for Industry: Clinical Data Needed to Support the Licensure of Pandemic Influenza Vaccines (US DHHS, FDA, CBER, May 2007).
### 14. APPENDICES

Table, figure, and listing shells are presented in Appendices 1, 2, and 3. Tables and figures included in the expedited interim immunogenicity reports are indicated by †. Tables and figures included in the Preliminary Report are indicated by \*. Topline tables are indicated by ‡.

# APPENDIX 1. TABLE MOCK-UPS

#### LIST OF TABLES

| Table 1: | Study Design | 38 |
|---|---|---|
| Table 2: | Schedule of Study Procedures – Vaccination Period | |
| Table 3: | Schedule of Study Procedures - Follow-Up Period (Including early termination and | |
| T-1.1. 4. | unscheduled visits) | |
| Table 4: | Power (%) to Detect Safety Events | |
| Table 5: | Precisions of Binomial Confidence Intervals | |
| Table 6: | Minimum Detectable Difference in Proportion Responders | 43 |
| Table 7: | Lower Confidence Bound for Difference in Proportion of Responders Between | |
| | Adjuvanted (N = 100) and Unadjuvanted (N = 50) Arms, 19-64 Years Stratum | 44 |
| Table 8: | Lower Confidence Bound for Difference in Proportion of Responders Between | |
| | Adjuvanted (N = 50) and Unadjuvanted (N = 25) Arms, $\geq$ 65 Years Stratum | 44 |
| Table 9: | Distribution of Protocol Deviations by Category, Type and Treatment Arm, All | |
| | Enrolled Subjects | |
| Table 10: | Solicited Adverse Event Grading Scale – Local | 47 |
| Table 11: | Solicited Adverse Event Grading Scale - Systemic | 48 |
| Table 12: | Vital Signs Adverse Event Grading Scale | 49 |
| Table 13: | Laboratory Adverse Event Grading Scale | 50 |
| Table 14: | Ineligibility Summary of Screen Failures* | |
| Table 15: | Analysis Populations by Treatment Arm, All Enrolled Subjects* | 52 |
| Table 16: | Analysis Populations by Treatment Arm and Age Stratum, All Enrolled Subjects* | |
| Table 17: | Subject Disposition by Treatment Arm, All Enrolled Subjects* | |
| Table 18: | Subject Disposition by Treatment Arm and Age Stratum, All Enrolled Subjects* | |
| Table 19: | Dates of First Study Vaccination by Site, Treatment Arm, and Age Stratum, for Safe | |
| | Analysis Population | |
| Table 20: | Dates of Second Study Vaccination by Site, Treatment Arm, and Age Stratum, for | • |
| 10.010 201 | Safety Analysis Population | 59 |
| Table 21: | Summary of Categorical Demographic and Baseline Characteristics by Site, All | |
| 10.010 211 | Enrolled Subjects | 60 |
| Table 22: | Summary of Continuous Demographic and Baseline Characteristics by Site, All | 00 |
| 14010 22. | Enrolled Subjects | 62 |
| Table 23: | Summary of Categorical Demographic and Baseline Characteristics by Treatment | 02 |
| 1 aoic 23. | Arm, All Enrolled Subjects* | 63 |
| Table 24: | Summary of Categorical Demographic and Baseline Characteristics by Treatment | 03 |
| 1 autc 24. | Arm and Age Stratum, All Enrolled Subjects* | 65 |
| Table 25: | Summary of Continuous Baseline Characteristics by Treatment Arm, All Enrolled | 03 |
| 1 aute 23. | Subjects* | 67 |
| Table 26: | Summary of Continuous Baseline Characteristics by Treatment Arm and Age Stratu | |
| Table 20: | | |
| T-1.1. 27. | All Enrolled Subjects* | 08 |
| Table 27: | Summary of Subjects with Prior or Concurrent Medical Conditions by MedDRA | <b>60</b> |
| T 11 20 | System Organ Class and Treatment Arm, Safety Analysis Population | 69 |
| Table 28: | Summary of Subjects with Prior or Concurrent Medical Conditions by MedDRA | <b>-</b> 0 |
| | System Organ Class, Treatment Arm and Age Stratum, Safety Analysis Population. | |
| Table 29: | Summaries of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by Stud | • |
| | Day and Treatment Arm, Modified Intent-to-Treat Population*†‡ | |
| Table 30: | Summaries of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by Stud | • |
| | Day and Treatment Arm, Per Protocol Population*‡ | 72 |
| Table 31: | Summaries of Neutralizing Antibody Against 2017 A/H7N9 by Study Day and | |
| | Treatment Arm, Modified Intent-to-Treat Population*†‡ | 72 |

| Table 32: | Summaries of Neutralizing Antibody Against 2017 A/H7N9 by Study Day and |
|---|---|
| T 11 22 | Treatment Arm, Per Protocol Population*‡ |
| Table 33: | Summaries of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by Study Day, Treatment Arm and Age Stratum, Modified Intent-to-Treat Population*†‡73 |
| Table 34: | Summaries of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by Study |
| 1 autc 54. | Day, Treatment Arm and Age Stratum, Per Protocol Population*: |
| Table 35: | Summaries of Neutralizing Antibody Against 2017 A/H7N9 by Study Day, Treatment |
| 1 4010 001 | Arm and Age Stratum, Modified Intent-to-Treat Population*†‡ |
| Table 36: | Summaries of Neutralizing Antibody Against 2017 A/H7N9 by Study Day, Treatment |
| | Arm and Age Stratum, Per Protocol Population*‡ |
| Table 37: | Summary of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by |
| | Treatment Arm and Age Categories at 21 Days Post Second Vaccination, Per-Protocol |
| | Population*76 |
| Table 38: | Summary of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by |
| | Treatment Arm and Age Stratum at 180 Days Post Second Vaccination, Per-Protocol |
| | Population*78 |
| Table 39: | Summary of Neutralizing Antibody Against 2017 A/H7N9 by Treatment Arm and |
| | Age Stratum at 21 Days Post Second Vaccination, Per-Protocol Population*78 |
| Table 40: | Summary of Neutralizing Antibody Against 2017 A/H7N9 by Treatment Arm and |
| | Age Stratum at 180 Days Post Second Vaccination, Per-Protocol Population*78 |
| Table 41: | Summary of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by |
| | Treatment Arm, Age Stratum and Sex at 21 Days Post Second Vaccination, Per- |
| | Protocol Population*79 |
| Table 42: | Summary of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by |
| | Treatment Arm, Age Stratum and Sex at 180 Days Post Second Vaccination, Per- |
| | Protocol Population*80 |
| Table 43: | Summary of Neutralizing Antibody Against 2017 A/H7N9 by Treatment Arm, Age |
| | Stratum and Sex at 21 Days Post Second Vaccination, Per-Protocol Population* 80 |
| Table 44: | Summary of Neutralizing Antibody Against 2017 A/H7N9 by Treatment Arm, Age |
| | Stratum and Sex at 180 Days Post Second Vaccination, Per-Protocol Population* 80 |
| Table 45: | Summary of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by |
| | Treatment Arm, Age Stratum and BMI at 21 Days Post Second Vaccination, Per- |
| | Protocol Population*81 |
| Table 46: | Summary of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by |
| | Treatment Arm, Age Stratum and BMI at 180 Days Post Second Vaccination, Per- |
| | Protocol Population*82 |
| Table 47: | Summary of Neutralizing Antibody Against 2017 A/H7N9 by Treatment Arm, Age |
| | Stratum and BMI at 21 Days Post Second Vaccination, Per-Protocol Population* 82 |
| Table 48: | Summary of Neutralizing Antibody Against 2017 A/H7N9 by Treatment Arm, Age |
| | Stratum and BMI at 180 Days Post Second Vaccination, Per-Protocol Population* 82 |
| Table 49: | Summary of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by |
| | Treatment Arm, Age Stratum and Prior Seasonal Influenza Vaccination at 21 Days |
| | Post Second Vaccination, Per-Protocol Population* |
| Table 50: | Summary of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by |
| | Treatment Arm, Age Stratum and Prior Seasonal Influenza Vaccination at 180 Days |
| | Post Second Vaccination, Per-Protocol Population* |
| Table 51: | Summary of Neutralizing Antibody Against 2017 A/H7N9 by Treatment Arm, Age |
| | Stratum and Prior Seasonal Influenza Vaccination at 21 Days Post Second |
| | Vaccination, Per-Protocol Population* |
| | , |

| Table 52: | Summary of Neutralizing Antibody Against 2017 A/H7N9 by Treatment Arm, Age |
|---|---|
| | Stratum and Prior Seasonal Influenza Vaccination at 180 Days Post Second |
| T 11 52 | Vaccination, Per-Protocol Population* |
| Table 53: | Logistic Regression Model to Evaluate the Relationship of HA Antigen Dose and |
| | AS03 Adjuvant with HAI Seroconversion Against 2017 A/H7N9 at 21 Days Post |
| T 11 54 | Second Study Vaccination, Per Protocol Population* |
| Table 54: | Logistic Regression Model to Evaluate the Relationship of HA Antigen Dose and |
| | AS03 Adjuvant with Neut Seroconversion Against 2017 A/H7N9 at 21 Days Post |
| T 11 55 | Second Study Vaccination, Per Protocol Population* |
| Table 55: | Logistic Regression Model to Evaluate the Relationship of HA Antigen Dose and |
| | AS03 Adjuvant with HAI Seroconversion Against 2017 A/H7N9 at 180 Days Post |
| T 11 56 | Second Study Vaccination, Per Protocol Population* |
| Table 56: | Logistic Regression Model to Evaluate the Relationship of HA Antigen Dose and |
| | AS03 Adjuvant with Neut Seroconversion Against 2017 A/H7N9 at 180 Days Post |
| | Second Study Vaccination, Per Protocol Population* |
| Table 57: | Logistic Regression Model to Evaluate the Relationship of HA Antigen Dose and |
| | AS03 Adjuvant with HAI Seroconversion Against 2017 A/H7N9 at 21 Days Post |
| | Second Study Vaccination, Adjusted for Baseline Covariates, Per Protocol |
| T 11 50 | Population* |
| Table 58: | Logistic Regression Model to Evaluate the Relationship of HA Antigen Dose and |
| | AS03 Adjuvant with Neut Seroconversion Against 2017 A/H7N9 at 21 Days Post |
| | Second Study Vaccination, Adjusted for Baseline Covariates, Per Protocol |
| T 11 50 | Population* |
| Table 59: | Logistic Regression Model to Evaluate the Relationship of HA Antigen Dose and |
| | AS03 Adjuvant with HAI Seroconversion Against 2017 A/H7N9 at 180 Days Post Second Study Vaccination, Adjusted for Baseline Covariates, Per Protocol |
| | Population* |
| Table 60: | Logistic Regression Model to Evaluate the Relationship of HA Antigen Dose and |
| Table 00. | AS03 Adjuvant with Neut Seroconversion Against 2017 A/H7N9 at 180 Days Post |
| | Second Study Vaccination, Adjusted for Baseline Covariates, Per Protocol |
| | Population* |
| Table 61: | Multiple Linear Regression Model to Evaluate the Relationship of HA Antigen Dose |
| 14010 01. | and AS03 Adjuvant with Log-Adjusted HAI Titer at 21 Days Post Second Study |
| | Vaccination, Per Protocol Population* |
| Table 62: | Multiple Linear Regression Model to Evaluate the Relationship of HA Antigen Dose |
| | and AS03 Adjuvant with Log-Adjusted Neut Titer at 21 Days Post Second Study |
| | Vaccination, Per Protocol Population* |
| Table 63: | Multiple Linear Regression Model to Evaluate the Relationship of HA Antigen Dose |
| | and AS03 Adjuvant with Log-Adjusted HAI Titer at 180 Days Post Second Study |
| | Vaccination, Per Protocol Population*90 |
| Table 64: | Multiple Linear Regression Model to Evaluate the Relationship of HA Antigen Dose |
| | and AS03 Adjuvant with Log-Adjusted Neut Titer at 180 Days Post Second Study |
| | Vaccination, Per Protocol Population*90 |
| Table 65: | Multiple Linear Regression Model to Evaluate the Relationship of HA Antigen Dose |
| | and AS03 Adjuvant with Log-Adjusted HAI Titer at 21 Days Post Second Study |
| | Vaccination, Adjusted for Baseline Covariates, Per Protocol Population*91 |
| Table 66: | Multiple Linear Regression Model to Evaluate the Relationship of HA Antigen Dose |
| | and AS03 Adjuvant with Log-Adjusted Neut Titer at 21 Days Post Second Study |
| | Vaccination, Adjusted for Baseline Covariates, Per Protocol Population* |

| Table 67: | Multiple Linear Regression Model to Evaluate the Relationship of HA Antigen Dose and AS03 Adjuvant with Log-Adjusted HAI Titer at 180 Days Post Second Study |
|---|---|
| | Vaccination, Adjusted for Baseline Covariates, Per Protocol Population*92 |
| Table 68: | Multiple Linear Regression Model to Evaluate the Relationship of HA Antigen Dose and AS03 Adjuvant with Log-Adjusted Neut Titer at 180 Days Post Second Study |
| | Vaccination, Adjusted for Baseline Covariates, Per Protocol Population* |
| Table 69: | Logistic Regression Model to Evaluate the Relationship of HA Antigen Dose and AS03 Adjuvant with HAI Seroconversion Against 2017 A/H7N9 at 21 Days Post |
| | Second Study Vaccination, Adjusted for Baseline Covariates and Age in Years, Per |
| | Protocol Population*93 |
| Table 70: | Multiple Linear Regression Model to Evaluate the Relationship of HA Antigen Dose |
| 14010 70. | and AS03 Adjuvant with Log-Adjusted HAI Titer at 21 Days Post Second Study |
| | Vaccination, Adjusted for Baseline Covariates and Age in Years, Per Protocol |
| | Population* |
| Table 71: | Summaries of Hemagglutination Inhibition Antibody Against Antigenically Drifted |
| 10010 / 11 | Variants by Study Day, Treatment Arm and Age Stratum, Per Protocol Population* 95 |
| Table 72: | Summaries of Neutralizing Antibody Against Antigenically Drifted Variants by Study |
| | Day, Treatment Arm and Age Stratum, Per Protocol Population*96 |
| Table 73: | Overall Summary of Adverse Events - Safety Population*‡ |
| Table 74: | Number of Adverse Events Occurring in 5% of Subjects in Any Treatment Group by |
| | MedDRA System Organ Class and Preferred Term, and Treatment Group - Safety |
| | Population 99 |
| Table 75: | Number and Percentage of Subjects Experiencing Solicited Events with 95% |
| | Confidence Intervals by Symptom and Treatment Arm Post Any Study Vaccination – |
| | Safety Population*100 |
| Table 76: | Number and Percentage of Subjects Experiencing Solicited Events with 95% |
| | Confidence Intervals by Symptom and Treatment Arm Post Study Vaccination 1 – |
| | Safety Population * |
| Table 77: | Number and Percentage of Subjects Experiencing Solicited Events with 95% |
| | Confidence Intervals by Symptom and Treatment Arm Post Study Vaccination 2 – |
| T. 11. 70 | Safety Population * |
| Table 78: | Number and Percentage of Subjects Experiencing Solicited Events with 95% |
| | Confidence Intervals by Symptom, Treatment Arm and Age Stratum Post Any Study |
| Table 79: | Vaccination – Safety Population * |
| Table /9: | Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom, Treatment Arm and Age Stratum Post Study |
| | Vaccination 1 – Safety Population * |
| Table 80: | Number and Percentage of Subjects Experiencing Solicited Events with 95% |
| Table 60. | Confidence Intervals by Symptom, Treatment Arm and Age Stratum Post Study |
| | Vaccination 2 – Safety Population * |
| Table 81: | Logistic Regression Model to Evaluate the Relationship of HA Antigen Dose, AS03 |
| 14010 011 | Adjuvant, and Age with Reporting Any Local Event Post Any Study Vaccination – |
| | Safety Population * |
| Table 82: | Logistic Regression Model to Evaluate the Relationship of HA Antigen Dose, AS03 |
| - | Adjuvant, and Age with Reporting Any Systemic Event Post Any Study Vaccination |
| | (N=X) – Safety Population * |
| Table 83: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, |
| | Maximum Severity and Treatment Arm Post Any Study Vaccination – Safety |
| | Population * |

| Table 84: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity and Treatment Arm Post Study Vaccination 1 – Safety Population * |
|---|---|
| Table 85: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity and Treatment Arm Post Study Vaccination 2 – Safety Population * |
| Table 86: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, Treatment Arm and Age Stratum Post Any Study Vaccination – Safety Population * |
| Table 87: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, Treatment Arm and Age Stratum Post Study Vaccination 1 – Safety Population * |
| Table 88: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, Treatment Arm and Age Stratum Post Study Vaccination 2 – Safety Population * |
| Table 89: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom,<br>Severity, Day Post Study Vaccination, Treatment Arm and Age Stratum Post Any<br>Study Vaccination – Safety Population |
| Table 90: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom,<br>Severity, Day Post Study Vaccination, Treatment Arm and Age Stratum Post Study<br>Vaccination 1 – Safety Population |
| Table 91: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom,<br>Severity, Day Post Study Vaccination, Treatment Arm and Age Stratum Post Study<br>Vaccination 2 – Safety Population |
| Table 92: | Number and Percentage of Subjects Experiencing Solicited Systemic Events for Dose 1 Compared with Dose 2 by Treatment Arm and Age Stratum – Safety Population 127 |
| Table 93: | Number and Percentage of Subjects Experiencing Solicited Local Events for Dose 1<br>Compared with Dose 2 by Treatment Arm and Age Stratum – Safety Population 130 |
| Table 94: | Number and Percentage of Subjects Experiencing Unsolicited Adverse Events with 95% Confidence Intervals by MedDRA System Organ Class and Preferred Term, and Treatment Arm – Safety Population * |
| Table 95: | Number and Percentage of Subjects Experiencing Unsolicited Adverse Events with 95% Confidence Intervals by MedDRA System Organ Class and Preferred Term, Treatment Arm and Age Stratum – Safety Population * |
| Table 96: | Number and Percentage of Subjects Experiencing Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Maximum Severity, Relationship, Treatment Arm and Age Stratum – Safety Population* |
| Table 97: | Number and Percentage of Subjects Experiencing Non-Serious Related Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Maximum Severity, Treatment Arm and Age Stratum – Safety Population |
| Table 98: | Number and Percentage of Subjects Experiencing Unsolicited Adverse Events Within 21 Days Post Study Vaccination by MedDRA System Organ Class and Preferred Term, Day Post Vaccination, Treatment Arm and Age Stratum – Safety Population135 |
| Table 99: | Number and Percentage of Subjects Experiencing Non-Serious, Related Unsolicited Adverse Events Within 21 Days Post Vaccination by MedDRA System Organ Class and Preferred Term, Study Vaccination, Treatment Arm and Age Stratum – Safety Population |
| Table 100: | Number of Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Day Post Vaccination, Treatment Arm and Age Stratum – Safety Population |
| Table 101: | Listing of Serious Adverse Events – Safety Population * |

| Table 102: | Listing of Adverse Events of Special Interest – Safety Population * |
|---|---|
| Table 103: | Listing of New Onset Chronic Medical Conditions – Safety Population * |
| Table 104: | Listing of Non-Serious, Unsolicited, Moderate or Severe Adverse Events – Safety |
| | Population * |
| Table 105: | Laboratory Results by Parameter, Maximum Severity, Study Day, Treatment Group |
| | and Age Stratum, All Laboratory Parameters – Safety Population * |
| Table 106: | Laboratory Results by Parameter, Maximum Severity, Study Day, Treatment Group |
| | and Age Stratum, Hemoglobin – Safety Population * |
| Table 107: | Laboratory Results by Parameter, Maximum Severity, Study Day, Treatment Group |
| | and Age Stratum, Alanine – Safety Population aminotransferase (ALT)*142 |
| Table 108: | Laboratory Results by Parameter, Maximum Severity, Study Day, Treatment Group |
| | and Age Stratum, Total Bilirubin – Safety Population * |
| Table 109: | Laboratory Results by Parameter, Maximum Severity, Study Day, Treatment Group |
| | and Age Stratum, Creatinine – Safety Population * |
| Table 110: | Laboratory Results by Parameter, Maximum Severity, Study Day, Treatment Arm and |
| | Age Stratum, White Blood Cells – Safety Population * |
| Table 111: | Laboratory Results by Parameter, Maximum Severity, Study Day, Treatment Arm and |
| | Age Stratum, Platelets – Safety Population * |
| Table 112: | Laboratory Summary Statistics by Parameter, Study Day, Treatment Arm and Age |
| | Stratum, White Blood Cells – Safety Population * |
| Table 113: | Laboratory Summary Statistics by Parameter, Study Day, Treatment Arm and Age |
| m 11 114 | Stratum, Hemoglobin – Safety Population * |
| Table 114: | Laboratory Summary Statistics by Parameter, Study Day, Treatment Arm and Age |
| T 11 115 | Stratum, Platelets – Safety Population * |
| Table 115: | Laboratory Summary Statistics by Parameter, Study Day, Treatment Arm and Age |
| T 11 116 | Stratum, Alanine Aminotransferase – Safety Population * (ALT) |
| Table 116: | Laboratory Summary Statistics by Parameter, Study Day, Treatment Arm and Age |
| Talala 117. | Stratum, Total Bilirubin – Safety Population * |
| Table 117: | Laboratory Summary Statistics by Parameter, Study Day, Treatment Arm and Age |
| Table 118: | Stratum, Creatinine – Safety Population * |
| Table 118: | Treatment Arm and Age Stratum, White Blood Cells – Safety Population * 146 |
| Table 119: | Laboratory Summary Statistics of Change from Baseline by Parameter, Study Day, |
| 1 aute 119. | Treatment Arm and Age Stratum, Hemoglobin – Safety Population * |
| Table 120: | Laboratory Summary Statistics of Change from Baseline by Parameter, Study Day, |
| 1 aute 120. | Treatment Arm and Age Stratum, Platelets – Safety Population *146 |
| Table 121: | Laboratory Summary Statistics of Change from Baseline by Parameter, Study Day, |
| 1 aut 121. | Treatment Arm and Age Stratum, Alanine aminotransferase (ALT) – Safety |
| | Population * |
| Table 122: | Laboratory Summary Statistics of Change from Baseline by Parameter, Study Day, |
| 14010 122. | Treatment Arm and Age Stratum, Total Bilirubin – Safety Population * |
| Table 123: | Laboratory Summary Statistics of Change from Baseline by Parameter, Study Day, |
| 14010 123. | Treatment Arm and Age Stratum, Creatinine – Safety Population * |
| Table 124: | Listing of Abnormal Laboratory Results - Chemistry |
| Table 125: | Listing of Abnormal Laboratory Results - Hematology |
| Table 126: | Vital Signs by Assessment, Maximum Severity, Study Day, Treatment Arm and Age |
| 14010 120. | Stratum, Any Assessment – Safety Population * |
| Table 127: | Vital Signs by Assessment, Maximum Severity, Study Day, Treatment Arm and Age |
| 12010 12/1 | Stratum, Oral Temperature – Safety Population |
| Table 128: | Vital Signs by Assessment, Maximum Severity, Study Day, Treatment Arm and Age |
| 12010 120. | Stratum, Systolic Blood Pressure – Safety Population |

| Table 129: | Vital Signs by Assessment, Maximum Severity, Study Day, Treatment Arm and Age |
|---|---|
| | Stratum, Diastolic Blood Pressure – Safety Population |
| Table 130: | Vital Signs by Assessment, Maximum Severity, Study Day, Treatment Arm and Age |
| | Stratum, Pulse – Safety Population |
| Table 131: | Number and Percentage of Subjects with Prior and Concurrent Medications by WHO |
| | Drug Classification and Treatment Arm – Safety Population |
| Table 132: | Number and Percentage of Subjects with Prior and Concurrent Medications by WHO |
| | Drug Classification, Treatment Arm and Age Stratum – Safety Population |

# 9.1 Overall Study Design and Plan Description

**Table 1: Study Design** 

| Treatment<br>Arms | Stratum | Day 1<br>Study Vaccination 1 | Day 22<br>Study Vaccination 2 |
|---|---|---|---|
| | | H7N9 vaccine 3.75 mcg plus<br>AS03 adjuvant | H7N9 vaccine 3.75 mcg plus<br>AS03 adjuvant |
| | Age $\ge 65$ , n=60 | | |
| Group 2, n=160 | Age 19-64, n=100 | H7N9 vaccine 7.5 mcg plus<br>AS03 adjuvant | H7N9 vaccine 7.5 mcg plus<br>AS03 adjuvant |
| | Age $\ge 65$ , n=60 | | |
| Group 3, n=160 | Age 19-64, n=100 | H7N9 vaccine 15 mcg plus<br>AS03 adjuvant | H7N9 vaccine 15 mcg plus AS03<br>adjuvant |
| | $Age \ge 65, n=60$ | A303 aujuvani | aujuvani |
| Group 4, n=80 | Age 19-64, =50 | r H7N9 vaccine 15 mcg<br>unadjuvanted | H7N9 vaccine 15 mcg<br>unadjuvanted |
| | Age ≥ 65, n=30 | unadjuvanicu | |
| Group 5, n=80 | Age 19-64, n=50 | H7N9 vaccine 45 mcg<br>unadjuvanted | H7N9 vaccine 45 mcg<br>unadjuvanted |
| | Age $\geq$ 65, n=30 | unadjuvanted | unacja vancea |
| Total Enrollment,<br>n = 640 | Age 19-64, n=400* | *Over enrollment up to 420 subjects may be allowed to e approximately 100 subjects in each AS03 adjuvanted treatm and 50 subjects in each of the unadjuvanted treatment arreligible for inclusion in post Dose 2 immunogenicity ana | |
| | Age ≥ 65, n=240** | **Over enrollment up to 300 subjects may be allowed to ensure 6 subjects in each of the AS03 adjuvanted treatment arms, and 30 subjects in each of the unadjuvanted treatment arms are eligible for inclusion in post Dose 2 immunogenicity analyses | |

## 9.5.1 Efficacy/Immunogenicity and Safety Measurements Assessed and Flow Chart

 Table 2:
 Schedule of Study Procedures – Vaccination Period

| Study Visit Number | V00 | V01 | V02** | V03 | V04 | V05** | V06 | V07 |
|---|---|---|---|---|---|---|---|---|
| Study Day post 1st<br>vaccination | Screening<br>(Optional)<br>D -28 to - | Enrollment<br>Dose 1<br>D1 | D4±1d | D8+2d | D22+7d | D25 | D29 | D43 |
| Study Day post 2 <sup>nd</sup> vaccination | | | | | Dose 2<br>D1 | D4±1d | D8+2d | D22+7d |
| | | Study Proced | ure/Evalu | ation | | | | |
| Obtain Informed Consent∞ | X | Χ¬ | | | | | | |
| Collect Demographic<br>Information | X | X <sup>†*</sup> | | | | | | |
| Review Eligibility Criteria | X | $X^{\dagger - 1}$ | | | $X^{\dagger 1}$ | | | |
| Medical History@ | X | X <sup>†</sup> ¬ | X | X | $X^{\dagger}$ | X | X | X |
| Concomitant Medications | $X^{\varsigma}$ | $X^{\dagger ightarrow \varsigma}$ | $X^{\varsigma}$ | $X^{\varsigma}$ | $X^{\dagger\varsigma}$ | $X^{\varsigma}$ | $X^{\varsigma}$ | $\mathbf{X}^{\varsigma}$ |
| Vital Signs\$ (Oral Temperature%, Pulse, and BP) | X | $X^{\dagger}$ | | | $X^{\dagger 2}$ | | | |
| Height and Weight | X | $X^{\dagger *}$ | | | | | | |
| Physical Examination <sup>3</sup> | X | X <sup>†*</sup> | | {X} | $\{X\}^{\dagger}$ | | {X} | {X} |
| Urine or Serum Pregnancy<br>Test | Χ^ | $X^{\dagger \wedge}$ | | | X <sup>†</sup> ^ | | | |
| Venous Blood Collection for<br>ESR | $X^{\neq}$ | $X^{\neq *}$ | | | | | | |
| Venous Blood Collection for<br>Clinical Safety Laboratory<br>Evaluations~ | | $X^{\dagger}$ | | X | Χ <sup>†</sup> | | X | |
| Venous Blood Collection for<br>Anti-viral Antibody Assays | | Χ <sup>†</sup> | | X | $X^{\dagger\Psi}$ | | X | X |
| Serum Sample Collected for<br>Future Research <sup>4</sup> | | $X^{\dagger}$ | | X | $X^{\dagger}$ | | X | X |
| Enrollment in AdvantageEDC <sup>SM</sup> and Randomization | | $X^{\dagger}$ | | | | | | |
| Pre-Administration<br>Reactogenicity Assessments | | $X^{\dagger}$ | | | $X^{\dagger}$ | | | |
| Study Vaccination | | X | | | X | | | |
| 20-minute Evaluation After<br>Study Vaccination | | X | | | X | | | |
| Examine Study Vaccination<br>Site | | X | | X | X | | X | |
| Post-Administration<br>Reactogenicity Assessments | | X | | | X | | | |

Table 2: Schedule of Study Procedures - Vaccination Period (continued)

| Study Visit Number | V00 | V01 | V02** | V03 | V04 | V05** | V06 | V07 |
|---|---|---|---|---|---|---|---|---|
| Study Day post 1st<br>vaccination | Screening<br>(Optional)<br>D -28 to - | Enrollment<br>Dose 1<br>D1 | D4±1d | D8+2d | D22+7d | D25 | D29 | D43 |
| Study Day post 2 <sup>nd</sup> vaccination | | | | | Dose 2<br>D1 | D4±1d | D8+2d | D22+7d |
| | | Study Proced | ure/Evalu | ation | | | | |
| Distribute Memory Aid and Study-Related Materials | | X | | | X | | | |
| Review Memory Aid | | | X | X | | X | X | |
| AE/SAE Assessment | | X <sup>&amp;</sup> | X& | X& | X& | X& | X& | X |

<sup>\*\*</sup> Phone call assessment

<sup>∞</sup> Prior to study procedures.

<sup>†</sup> Prior to study vaccination.

<sup>&</sup>lt;sup>1</sup> Review results of clinical screening (ESR) or safety laboratory evaluations.

<sup>-</sup> Review/confirm information or activity in subjects previously consented and screened

<sup>©</sup> Complete medical history will be obtained by interview of subjects at the first visit (either screening [optional] or on Day 1 prior to the first study vaccination) and interim medical history will be obtained by interview of subjects at subsequent visits.

<sup>&</sup>lt;sup>6</sup> Receipt of non-study influenza vaccines will be solicited through approximately 180 days after the last study vaccination, and reported in the eCRF.

<sup>\*</sup> Not required if done at the optional screening visit

Vital signs assessed on Day 1 prior to the first study vaccination will be considered as baseline.

<sup>&</sup>lt;sup>%</sup> Subjects must not eat or drink anything hot or cold, or smoke within 10 minutes prior to taking oral temperature.

Vital signs are not required for subjects who are discontinued from receipt of the second study vaccination and are being followed for safety.

At the screening (or baseline if not done at screening) visit, a physical examination will be performed on all subjects to include the following organs and organ systems: skin, head and neck, lungs, heart, liver, spleen, extremities, lymph nodes, and nervous system.

<sup>{}</sup> Targeted physical examination if indicated based on review of interim medical history.

Will be performed on all women of childbearing potential at screening (optional) and within 24 hours prior to each study vaccination and results must be negative and known prior to each study vaccination.

To be performed locally by the site. The ESR value must be confirmed as <30 mm/hr prior to randomization and first study vaccination.</p>

<sup>~</sup> Includes WBC, Hgb, PLT, ALT, T. Bili, Cr

<sup>&</sup>lt;sup>Ψ</sup> Subjects who do not receive the second study vaccination will continue with follow-up safety assessments (may be conducted by phone call) rather than in person continuing through approximately 12 months after their first study vaccination. These subjects will also be encouraged to provide a venous blood sample for anti-viral antibody assays at approximately 21 and 180 days after their first study vaccination

<sup>&</sup>lt;sup>4</sup> For subjects who have consented to collection of serum for future use

<sup>&</sup>amp; Inclusive of reactogenicity assessments performed on the day of each study vaccination through 7 days after each study vaccination.

Table 3: Schedule of Study Procedures - Follow-Up Period (Including early termination and unscheduled visits)

| Study Visit Number | **80\ | **60\ | V10 | V11** | needed) | eded) |
|---|---|---|---|---|---|---|
| Study Day post first study vaccination | D82 | D142 | D202 | D387 | nation (if | Unscheduled (if needed) |
| Study Day post second study vaccination | D61±7d | D121±14d | D181±14d | D366±14d | Early Termination (if needed) | Unsched |
| | | | Study Pr | ocedure/Evalua | ition | |
| Medical History <sup>@</sup> | | | X | | X | X (if indicated) |
| Concomitant Medications | $X^{\varsigma}$ | Χ <sup>ç</sup> | Χ <sup>ς</sup> | | X (if within 21 days after last<br>study vaccination and receipt of<br>any non-study influenza vaccine<br>will be recorded if within 180<br>days after the 2nd study<br>vaccination) | X (if prior to 21 days after last study vaccination and receipt of any non-study influenza vaccine will be recorded if within 180 days after the 2nd study) |
| Vital Signs<br>(Oral Temperature%, Pulse,<br>and BP) | | | | | X (may be obtained if indicated) | X (may be obtained if indicated) |
| Physical Examination <sup>3</sup> | | | {X} | | {X} | {X} |
| Venous Blood Collection for<br>Clinical Safety Laboratory<br>Evaluations~ | | | | | X (if within 7 days after the last study vaccination) | X (if indicated) |
| Venous Blood Collection for<br>Anti-viral Antibody Assays | | | X | | X (if within 21 days after last study vaccination) | X (if prior to 21 days after last study vaccination) |
| Serum Sample Collected for<br>Future Research <sup>4</sup> | | | X | | X(if within 21 days after last study vaccination | X(if prior to 21 days after last study vaccination |

| Study Visit Number | **80A | **60A | V10 | V11** | needed) | (papa |
|---|---|---|---|---|---|---|
| Study Day post first study vaccination | D82 | D142 | D202 | D387 | Termination (if needed) | Unscheduled (if needed) |
| Study Day post second study vaccination | D61±7d | D121±14d | D181±14d | D366±14d | Early Termi | |
| | | | Study Pr | rocedure/Evalua | ition | |
| Examine Study Vaccination Site | | | | | X (if within 7 days after last study vaccination) | X (if within 7 days after last study vaccination) |
| Post-Administration Reactogenicity Assessments | | | | | X (if within 7 days after last study vaccination) | X (if within 7 days after last study vaccination) |
| Review Memory Aid | | | | | X (if within 7 days after last study vaccination) | X (if within 7 days after last study vaccination) |
| AE/SAE Assessment | X# | X <sup>#</sup> ! | X# | X# | X <sup>#</sup> | $X^{\#}$ |

<sup>\*\*</sup> Phone call assessment

<sup>@</sup> Complete medical history will be obtained by interview of subjects at screening (optional) or on Day 1 prior to the first study vaccination and interim medical history will be obtained by interview of subjects at follow-up visits after the first study vaccination.

<sup>&</sup>lt;sup>6</sup> Receipt of non-study influenza vaccines will be solicited through approximately 180 days after the last study vaccination, and reported in the eCRF.

<sup>%</sup> Subjects must not eat or drink anything hot or cold, or smoke within 10 minutes prior to taking oral temperature.

<sup>{}</sup> Targeted physical examination if indicated based on review of interim medical history.

<sup>~</sup> Includes WBC, Hgb, PLT, ALT, T. Bili, Cr

Ψ Subjects who do not receive the second study vaccination will continue with follow-up safety assessments (may be conducted by phone call) rather than in person continuing through approximately 12 months after their first study vaccination. These subjects will also be encouraged to provide a venous blood sample for anti-viral antibody assays at approximately 21 and 180 days after their first study vaccination

<sup>&</sup>lt;sup>4</sup> For subjects who have consented to collection of serum for future use

<sup>\*</sup> AEs will be limited to SAEs and MAAEs, including NOCMCs and PIMMCs if after 21 days after last study vaccination

### 9.7.1 Sample Size

**Table 4:** Power (%) to Detect Safety Events

| Event<br>Frequency | N = 60 | N = 100 | N = 160 | N = 480 |
|---------------------|--------|---------|---------|---------|
| ≥10%<br>Very Common | >99 | >99 | >99 | >99 |
| ≥1%<br>Common | 45 | 63 | 80 | >99 |
| ≥0.1%<br>Uncommon | 6 | 10 | 15 | 38 |
| ≥0.01%<br>Rare | <1 | 1 | 2 | 5 |

**Table 5: Precisions of Binomial Confidence Intervals** 

| N | 95% CI |
|-----|--------|
| 60 | 37-63 |
| 100 | 40-60 |
| 160 | 42-58 |
| 480 | 45-55 |

**Table 6:** Minimum Detectable Difference in Proportion Responders

| Assumed Proportion of subjects with titer ≥40 in comparator arm | 19-64 years stratum<br>(N = 100) | ≥65 years stratum<br>(N = 50) |
|---|---|---|
| 0.40 | 0.19 | 0.27 |
| 0.50 | 0.19 | 0.27 |
| 0.60 | 0.18 | 0.25 |
| 0.70 | 0.16 | 0.21 |
| 0.80 | 0.13 | 0.16 |
| 0.90 | 0.08 | 0.10 |

Table 7: Lower Confidence Bound for Difference in Proportion of Responders Between Adjuvanted (N = 100) and Unadjuvanted (N = 50) Arms, 19-64 Years Stratum

| Adjuvanted Arm | Unadjuvanted<br>Arm | Difference | Lower Confidence<br>Bound* |
|---|---|---|---|
| 0.50 | 0.10 | 0.40 | 0.26 |
| 0.60 | 0.10 | 0.50 | 0.36 |
| 0.70 | 0.10 | 0.60 | 0.46 |
| 0.80 | 0.10 | 0.70 | 0.56 |
| 0.90 | 0.10 | 0.80 | 0.67 |

<sup>\*</sup> Farrington-Manning confidence limits.

Table 8: Lower Confidence Bound for Difference in Proportion of Responders Between Adjuvanted (N = 50) and Unadjuvanted (N = 25) Arms, ≥65 Years Stratum

| Adjuvanted Arm | Unadjuvanted<br>Arm | Difference | Lower Confidence<br>Bound* |
|---|---|---|---|
| 0.50 | 0.10 | 0.40 | 0.19 |
| 0.60 | 0.10 | 0.50 | 0.29 |
| 0.70 | 0.10 | 0.60 | 0.39 |
| 0.80 | 0.10 | 0.70 | 0.49 |
| 0.90 | 0.10 | 0.80 | 0.60 |

<sup>\*</sup> Farrington-Manning confidence limits.

#### **10.2** Protocol Deviations

Table 9: Distribution of Protocol Deviations by Category, Type and Treatment Arm, All Enrolled Subjects

| | | Grot<br>3.75<br>A/H<br>+ A<br>(N= | mcg<br>7N9<br>S03 | Grot<br>7.5 1<br>A/H<br>+ A<br>(N= | mcg<br>7N9<br>S03 | Grot<br>15 r<br>A/H<br>+ A<br>(N= | ncg<br>7N9<br>S03 | Groot<br>15 r<br>A/H<br>(N= | ncg<br>7N9 | Groot<br>45 r<br>A/H<br>(N= | ncg<br>7N9 | A<br>Subj<br>(N= | ects |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Category | Deviation Type | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. |
| Eligibility/enrollment | Any type | | | | | | | | | | | | |
| | Did not meet inclusion criterion | X | x | x | x | x | x | x | x | x | x | X | x |
| | Met exclusion criterion | | | | | | | | | | | | |
| | ICF not signed prior to study procedures | | | | | | | | | | | | |
| | Other | | | | | | | | | | | | |
| Treatment administration schedule | Any type | | | | | | | | | | | | |
| | Out of window visit | | | | | | | | | | | | |
| | Missed<br>visit/visit not<br>conducted | | | | | | | | | | | | |
| | Missed<br>treatment<br>administration | | | | | | | | | | | | |
| | Delayed<br>treatment<br>administration | | | | | | | | | | | | |
| | Other | | | | | | | | | | | | |
| Follow-up visit schedule | Any type | | | | | | | | | | | | |
| | Out of window visit | | | | | | | | | | | | |
| | Missed<br>visit/visit not<br>conducted | | | | | | | | | | | | |
| | Other | | | | | | | | | | | | |
| Protocol procedure/assessment | Any type | | | | | | | | | | | | |
| | Incorrect version of ICF signed | | | | | | | | | | | | |

Table 9: Distribution of Protocol Deviations by Category, Type and Treatment Arm, All Enrolled Subjects (continued)

| | | Grov<br>3.75<br>A/H<br>+ A/<br>(N= | up 1<br>mcg<br>7N9<br>S03 | Grou<br>7.5 I<br>A/H'<br>+ A!<br>(N= | ncg<br>7N9<br>S03 | Groot<br>15 r<br>A/H<br>+ A<br>(N= | ncg<br>7N9<br>S03 | Groot<br>15 r<br>A/H<br>(N= | ncg<br>7N9 | Grov<br>45 r<br>A/H<br>(N= | ncg<br>7N9 | A<br>Subj<br>(N= | ects |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Category | Deviation Type | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. | # of<br>Subj. | # of<br>Dev. |
| | Blood not collected | | | | | | | | | | | | |
| | Urine not collected | | | | | | | | | | | | |
| | Stool not collected | | | | | | | | | | | | |
| | Other specimen not collected | | | | | | | | | | | | |
| | Too few aliquots obtained | | | | | | | | | | | | |
| | Specimen result not obtained | | | | | | | | | | | | |
| | Required procedure not conducted | | | | | | | | | | | | |
| | Required procedure done incorrectly | | | | | | | | | | | | |
| | Study product<br>temperature<br>excursion | | | | | | | | | | | | |
| | Specimen<br>temperature<br>excursion | | | | | | | | | | | | |
| | Other | | | | | | | | | | | | |
| Treatment administration | Any type | | | | | | | | | | | | |
| | Required procedure done incorrectly | | | | | | | | | | | | |
| | Study product<br>temperature<br>excursion | | | | | | | | | | | | |
| | Other | | | | | | | | | | | | |
| Blinding policy/procedure | Any type | | | | | | | | | | | | |
| | Treatment unblinded | | | | | | | | | | | | |
| | Other | | | | | | | | | | | | |

## 12.2.2 Displays of Adverse Events

**Table 10:** Solicited Adverse Event Grading Scale – Local

| Local (Injection Site) Reactogenicity Grading | | | |
|---|---|---|---|
| Local (Injection<br>Site) Reaction | Mild (Grade 1) | Moderate (Grade 2) | Severe (Grade 3) |
| Pain – experienced<br>without touching the<br>injection site<br>(spontaneous<br>discomfort) | Subject is aware of pain,<br>but it does not interfere<br>with daily activity, and<br>no pain medication is<br>taken | Subject is aware of pain;<br>there is interference with<br>daily activity <b>or</b> it<br>requires repeated use of<br>a non-narcotic pain<br>reliever for >24 hours | Subject is aware of pain, and it prevents daily activity or requires any use of a narcotic pain reliever |
| Tenderness – hurts only<br>when injection site is<br>touched or the arm is<br>moved | The area immediately surrounding the injection site hurts only when touched or with arm motion, and it does not interfere with daily activity | The area immediately surrounding the injection site hurts when touched or with arm motion, and it interferes with daily activity | The area immediately surrounding the injection site hurts when touched or with arm motion, <b>and</b> it prevents daily activity |
| Pruritus (Itching) | Does not interfere with daily activity | Interferes with daily activity | Prevents daily activity |
| Ecchymosis<br>(Bruising)* | Does not interfere with daily activity | Interferes with daily activity | Prevents daily activity |
| Erythema (Redness)* | Does not interfere with daily activity | Interferes with daily activity | Prevents daily activity |
| Induration<br>(Hardness)/Swelling* | Does not interfere with daily activity | Interferes with daily activity | Prevents daily activity |
| <u> 1</u> | Local (Injection Site) Re | actogenicity Measuremo | <u>ents</u> |
| Local (Injection Site)<br>Reaction | Small (Grade 1) | Medium (Grade 2) | Large (Grade 3) |
| Ecchymosis<br>(Bruising)* | <20 mm | 20 mm – 50 mm | >50 mm |
| Erythema (Redness)* | <20 mm | 20 mm – 50 mm | >50 mm |
| Induration<br>(Hardness)/Swelling* | <20 mm | 20 mm – 50 mm | >50 mm |

**Table 11: Solicited Adverse Event Grading Scale - Systemic** 

| Subjective Systemic Reactogenicity Grading | | | |
|---|---|---|---|
| Systemic (Subjective) | Mild (Grade 1) | Moderate (Grade 2) | Severe (Grade 3) |
| Feverishness<br>(Chills/Shivering/Sweating) | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |
| Fatigue (Tiredness) | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |
| Malaise (General Unwell<br>Feeling) | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |
| Myalgia (Body<br>Aches/Muscular Pain)* | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |
| Arthralgia (Joint Pain)* | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |
| Headache | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |
| Nausea | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |
| Quantitative Systemic Reactogenicity Grading | | | |
| Systemic (Quantitative) | Mild (Grade 1) | Moderate (Grade 2) | Severe (Grade 3) |
| Fever# - oral† | 38.0°C – 38.4°C | 38.5°C – 38.9°C | >38.9°C |
| revei# - Orai | 100.4°F – 101.1°F | 101.2°F – 102.0°F | >102.0°F |

<sup>\*</sup> Not at injection site.

<sup>&</sup>lt;sup>#</sup> Oral temperature assessed on Day 1 prior to the first study vaccination will be considered as baseline. A fever can be considered not related to the study product if an alternative etiology can be documented.

 Table 12:
 Vital Signs Adverse Event Grading Scale

| For Individuals 19-64 years of age, pulse and blood pressure# will be graded as follows: | | | |
|---|---|---|---|
| Physiologic Parameter | Mild (Grade 1) | Moderate (Grade 2) | Severe (Grade 3) |
| Bradycardia - beats per minute | 45 – 46 | 40 – 44 | <40 |
| Tachycardia - beats per minute | 101 – 130 | 131 – 155 | >155 |
| Hypotension (systolic) mmHg | 80 - 84 | 75 – 79 | <75 |
| Hypotension (diastolic) mmHg | 50 – 54 | 45 – 49 | <45 |
| Hypertension (systolic) mmHg | 151 – 155 | 156 – 160 | >160 |
| Hypertension (diastolic) mmHg | 96 – 100 | 101 – 105 | >105 |

For Individuals >65 years of age, pulse and blood pressure<sup>#</sup> will be graded as follows:

| Physiologic Parameter | Mild (Grade 1) | Moderate (Grade 2) | Severe (Grade 3) |
|---|---|---|---|
| Bradycardia - beats per minute | 45 – 46 | 40 – 44 | <40 |
| Tachycardia - beats per minute | 101 – 130 | 131 – 155 | >155 |
| Hypotension (systolic) mm Hg | 80 – 84 | 75 – 79 | <75 |
| Hypotension (diastolic) mm Hg | 50 – 54 | 45 – 49 | <45 |
| Hypertension (systolic) mm Hg | 161 – 165 | 166 – 170 | >170 |
| Hypertension (diastolic) mm<br>Hg | 96 – 100 | 101 – 105 | >105 |

<sup>&</sup>lt;sup>#</sup> Pulse and blood pressure assessed on Day 1 prior to the first study vaccination will be considered as baseline.

# 12.4.1 Individual Laboratory Measurements and Abnormal Laboratory Values

**Table 13: Laboratory Adverse Event Grading Scale** 

| Hematology | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) |
|---|---|---|---|
| WBC 10 <sup>3</sup> /μL (Decrease) | 2.5 - 3.9 | 1.5 – 2.4 | <1.5 |
| WBC 10 <sup>3</sup> /μL (Increase) | 10.6 – 15.0 | 15.1 – 20.0 | >20.0 |
| Hgb g/dL (Decrease) (Female) | 10.1 - 11.4 | 8.5 – 10 | <8.5 |
| Hgb g/dL (Decrease) (Male) | 11.0 - 12.4 | 9.5 – 10.9 | <9.5 |
| Platelets 10 <sup>3</sup> /μL (Decrease) | 125 – 139 | 100 – 124 | <100 |
| Platelets 10 <sup>3</sup> /μL (Increase) | 416 - 550 | 551-750 | >750 |
| Chemistry | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) |
| ALT IU/L (Increase) (Female) | 44 – 100 | 101 – 200 | >200 |
| ALT IU/L (Increase) (Male) | 61 - 138 | 139 – 275 | >275 |
| Total Bilirubin mg/dL (Increase) – when accompanied by any increase in ALT | 1.30 – 1.59 | 1.60 – 1.80 | >1.80 |
| Total Bilirubin mg/dL (Increase) – when ALT is normal | 1.30 - 1.89 | 1.90 – 2.40 | >2.40 |
| Creatinine mg/dL (Increase)<br>(Female) | 1.1 – 1.7 | 1.8 – 2.0 | >2.0 |
| Creatinine mg/dL (Increase) (Male) | 1.4 – 1.7 | 1.8 – 2.0 | >2.0 |

## 14.1 Description of Study Subjects

#### 14.1.1 Disposition of Subjects

Table 14: Ineligibility Summary of Screen Failures\*

| Inclusion/Exclusion Category | Inclusion/Exclusion Criterion | nª | % b |
|---|---|---|---|
| Inclusion and Exclusion | Number of subjects failing any eligibility criterion | х | X |
| Inclusion | Any inclusion criterion | х | х |
| | [inclusion criterion 1] | Х | х |
| | [inclusion criterion 2] | Х | х |
| | [inclusion criterion 3] | Х | х |
| Exclusion | Any exclusion criterion | Х | х |
| | [exclusion criterion 1] | Х | х |
| | [exclusion criterion 2] | Х | х |
| | [exclusion criterion 3] | Х | х |

<sup>&</sup>lt;sup>a</sup>More than one criterion may be marked per subject.

<sup>&</sup>lt;sup>b</sup>Denominator for percentages is the total number of screen failures.

Table 15: Analysis Populations by Treatment Arm, All Enrolled Subjects\*

| | | 3.75<br>A/H<br>+ A | oup 1<br>5 mcg<br>17N9<br>AS03<br>=X) | 7.5<br>A/H<br>+ A | oup 2<br>mcg<br>17N9<br>AS03<br>=X) | 15<br>A/H<br>+ A | oup 3<br>mcg<br>17N9<br>AS03<br>=X) | 15<br>A/H | oup 4<br>mcg<br>I7N9<br>=X) | 45<br>A/H | oup 5<br>mcg<br>I7N9<br>=X) | | ubjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Analysis Populations | Reason Subjects Excluded | n | % | n | % | n | % | n | % | n | % | n | % |
| Safety Population | Any Reason | х | xx | x | XX | х | XX | X | xx | х | xx | х | xx |
| | Study Vaccination 1 Not Received | | | | | | | | | | | | |
| Modified Intent to Treat | Any Reason | | | | | | | | | | | | |
| | Study Vaccination 1 Not Received | | | | | | | | | | | | |
| | No Baseline Results Available | | | | | | | | | | | | |
| | No Post-Vaccination Results Available | | | | | | | | | | | | |
| Per-Protocol, Day 8 | Any Reason | | | | | | | | | | | | |
| | Study Vaccination 1 Not Received | | | | | | | | | | | | |
| | No Baseline Results Available | | | | | | | | | | | | |
| | No Day 9 Result Reported by Lab | | | | | | | | | | | | |
| | Lost to Follow-up Before Day 9 | | | | | | | | | | | | |
| | Receipt of Non-Study Vaccination | | | | | | | | | | | | |
| | Receipt of Immunosuppressive medication | | | | | | | | | | | | |
| | Day 9 Visit Out of Window | | | | | | | | | | | | |
| Per-Protocol, Day 22 | Any Reason | | | | | | | | | | | | |
| | Study Vaccination 1 Not Received | | | | | | | | | | | | |
| | No Baseline Results Available | | | | | | | | | | | | |
| | No Day 21 Result Reported by Lab | | | | | | | | | | | | |
| | Lost to Follow-up Before Day 21 | | | | | | | | | | | | |

Table 15: Analysis Populations by Treatment Arm, All Enrolled Subjects\* (continued)

| 1 | 1 | ı | 1 | | 1 | 1 | , | | | | , | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Receipt of Non-Study Vaccination | | | | | | | | | | | | |
| Receipt of Immunosuppressive medication | | | | | | | | | | | | |
| Day 21 Visit Out of Window | | | | | | | | | | | | |
| Any Reason | | | | | | | | | | | | |
| Study Vaccination 1 Not Received | | | | | | | | | | | | |
| Study Vaccination 2 Not Received | | | | | | | | | | | | |
| Study Vaccination 2 Out of Window | | | | | | | | | | | | |
| No Baseline Results Available | | | | | | | | | | | | |
| No Day 29 Result Reported by Lab | | | | | | | | | | | | |
| Lost to Follow-up Before Day 29 | | | | | | | | | | | | |
| Receipt of Non-Study Vaccination | | | | | | | | | | | | |
| Receipt of Immunosuppressive medication | | | | | | | | | | | | |
| Day 29 Visit Out of Window | | | | | | | | | | | | |
| Any Reason | | | | | | | | | | | | |
| Study Vaccination 1 Not Received | | | | | | | | | | | | |
| Study Vaccination 2 Not Received | | | | | | | | | | | | |
| Study Vaccination 2 Out of Window | | | | | | | | | | | | |
| No Baseline Results Available | | | | | | | | | | | | |
| No Day 43 Result Reported by Lab | | | | | | | | | | | | |
| Lost to Follow-up Before Day 43 | | | | | | | | | | | | |
| Receipt of Non-Study Vaccination | | | | | | | | | | | | |
| Receipt of Immunosuppressive medication | | | | | | | | | | | | |
| Day 43 Visit Out of Window | | | | | | | | | | | | |
| | Receipt of Immunosuppressive medication Day 21 Visit Out of Window Any Reason Study Vaccination 1 Not Received Study Vaccination 2 Not Received Study Vaccination 2 Out of Window No Baseline Results Available No Day 29 Result Reported by Lab Lost to Follow-up Before Day 29 Receipt of Non-Study Vaccination Receipt of Immunosuppressive medication Day 29 Visit Out of Window Any Reason Study Vaccination 1 Not Received Study Vaccination 2 Not Received Study Vaccination 2 Out of Window No Baseline Results Available No Day 43 Result Reported by Lab Lost to Follow-up Before Day 43 Receipt of Immunosuppressive medication Receipt of Immunosuppressive medication | Receipt of Immunosuppressive medication Day 21 Visit Out of Window Any Reason Study Vaccination 1 Not Received Study Vaccination 2 Not Received Study Vaccination 2 Out of Window No Baseline Results Available No Day 29 Result Reported by Lab Lost to Follow-up Before Day 29 Receipt of Non-Study Vaccination Receipt of Immunosuppressive medication Day 29 Visit Out of Window Any Reason Study Vaccination 1 Not Received Study Vaccination 2 Not Received Study Vaccination 2 Out of Window No Baseline Results Available No Day 43 Result Reported by Lab Lost to Follow-up Before Day 43 Receipt of Non-Study Vaccination Receipt of Immunosuppressive medication | Receipt of Immunosuppressive medication Day 21 Visit Out of Window Any Reason Study Vaccination 1 Not Received Study Vaccination 2 Out of Window No Baseline Results Available No Day 29 Result Reported by Lab Lost to Follow-up Before Day 29 Receipt of Immunosuppressive medication Day 29 Visit Out of Window Any Reason Study Vaccination 1 Not Received Study Vaccination 2 Not Received Study Vaccination 2 Out of Window No Baseline Results Available No Day 43 Result Reported by Lab Lost to Follow-up Before Day 43 Receipt of Non-Study Vaccination Receipt of Immunosuppressive medication | Receipt of Immunosuppressive medication Day 21 Visit Out of Window Any Reason Study Vaccination 1 Not Received Study Vaccination 2 Not Received Study Vaccination 2 Out of Window No Baseline Results Available No Day 29 Result Reported by Lab Lost to Follow-up Before Day 29 Receipt of Immunosuppressive medication Day 29 Visit Out of Window Any Reason Study Vaccination 1 Not Received Study Vaccination 2 Not Received Study Vaccination 2 Out of Window No Baseline Results Available No Day 43 Result Reported by Lab Lost to Follow-up Before Day 43 Receipt of Non-Study Vaccination Receipt of Immunosuppressive medication | Receipt of Immunosuppressive medication Day 21 Visit Out of Window Any Reason Study Vaccination 1 Not Received Study Vaccination 2 Out of Window No Baseline Results Available No Day 29 Result Reported by Lab Lost to Follow-up Before Day 29 Receipt of Non-Study Vaccination Receipt of Immunosuppressive medication Day 29 Visit Out of Window Any Reason Study Vaccination 1 Not Received Study Vaccination 2 Out of Window No Baseline Results Available No Day 43 Result Reported by Lab Lost to Follow-up Before Day 43 Receipt of Non-Study Vaccination | Receipt of Immunosuppressive medication Day 21 Visit Out of Window Any Reason Study Vaccination 1 Not Received Study Vaccination 2 Out of Window No Baseline Results Available No Day 29 Result Reported by Lab Lost to Follow-up Before Day 29 Receipt of Non-Study Vaccination Receipt of Immunosuppressive medication Day 29 Visit Out of Window Any Reason Study Vaccination 1 Not Received Study Vaccination 2 Not Received Study Vaccination 2 Out of Window No Baseline Results Available No Day 43 Result Reported by Lab Lost to Follow-up Before Day 43 Receipt of Non-Study Vaccination Receipt of Immunosuppressive medication | Receipt of Immunosuppressive medication Day 21 Visit Out of Window Any Reason Study Vaccination 1 Not Received Study Vaccination 2 Out of Window No Baseline Results Available No Day 29 Result Reported by Lab Lost to Follow-up Before Day 29 Receipt of Non-Study Vaccination Receipt of Immunosuppressive medication Day 29 Visit Out of Window Any Reason Study Vaccination 1 Not Received Study Vaccination 2 Out of Window Any Reason Study Vaccination 2 Not Received Study Vaccination 2 Out of Window No Baseline Results Available No Day 43 Result Reported by Lab Lost to Follow-up Before Day 43 Receipt of Immunosuppressive medication Receipt of Immunosuppressive medication | Receipt of Immunosuppressive medication Day 21 Visit Out of Window Any Reason Study Vaccination 1 Not Received Study Vaccination 2 Out of Window No Baseline Results Available No Day 29 Result Reported by Lab Lost to Follow-up Before Day 29 Receipt of Non-Study Vaccination Receipt of Immunosuppressive medication Day 29 Visit Out of Window Any Reason Study Vaccination 1 Not Received Study Vaccination 2 Out of Window Any Reason Study Vaccination 2 Not Received Study Vaccination 2 Out of Window No Baseline Results Available No Day 43 Result Reported by Lab Lost to Follow-up Before Day 43 Receipt of Immunosuppressive medication | Receipt of Immunosuppressive medication Day 21 Visit Out of Window Any Reason Study Vaccination 1 Not Received Study Vaccination 2 Out of Window No Baseline Results Available No Day 29 Result Reported by Lab Lost to Follow-up Before Day 29 Receipt of Immunosuppressive medication Day 29 Visit Out of Window Any Reason Study Vaccination 1 Not Received Study Vaccination 2 Out of Window Any Reason Study Vaccination 2 Not Received Study Vaccination 2 Out of Window No Baseline Results Available No Day 43 Result Reported by Lab Lost to Follow-up Before Day 43 Receipt of Immunosuppressive medication | Receipt of Immunosuppressive medication Day 21 Visit Out of Window Any Reason Study Vaccination 1 Not Received Study Vaccination 2 Not Received Study Vaccination 2 Out of Window No Baseline Results Available No Day 29 Result Reported by Lab Lost to Follow-up Before Day 29 Receipt of Non-Study Vaccination Receipt of Immunosuppressive medication Day 29 Visit Out of Window Any Reason Study Vaccination 1 Not Received Study Vaccination 2 Not Received Study Vaccination 2 Out of Window No Baseline Results Available No Day 43 Result Reported by Lab Lost to Follow-up Before Day 43 Receipt of Non-Study Vaccination Receipt of Immunosuppressive medication | Receipt of Immunosuppressive medication Day 21 Visit Out of Window Any Reason Study Vaccination 1 Not Received Study Vaccination 2 Not Received Study Vaccination 2 Out of Window No Baseline Results Available No Day 29 Result Reported by Lab Lost to Follow-up Before Day 29 Receipt of Non-Study Vaccination Receipt of Immunosuppressive medication Day 29 Visit Out of Window Any Reason Study Vaccination 1 Not Received Study Vaccination 1 Not Received Study Vaccination 2 Not Received Study Vaccination 2 Out of Window No Baseline Results Available No Day 43 Result Reported by Lab Lost to Follow-up Before Day 43 Receipt of Non-Study Vaccination Receipt of Immunosuppressive medication | Receipt of Immunosuppressive medication Day 21 Visit Out of Window Any Reason Study Vaccination 1 Not Received Study Vaccination 2 Not Received Study Vaccination 2 Out of Window No Baseline Results Available No Day 29 Result Reported by Lab Lost to Follow-up Before Day 29 Receipt of Non-Study Vaccination Receipt of Immunosuppressive medication Day 29 Visit Out of Window Any Reason Study Vaccination 1 Not Received Study Vaccination 2 Not Received Study Vaccination 2 Not Received Study Vaccination 2 Not Received Study Vaccination 2 Out of Window No Baseline Results Available No Day 43 Result Reported by Lab Lost to Follow-up Before Day 43 Receipt of Non-Study Vaccination Receipt of Immunosuppressive medication |

Table 16: Analysis Populations by Treatment Arm and Age Stratum, All Enrolled Subjects\*

| | | 3.75 | 5 mcg<br>+ A | up 1<br>; A/H<br>.S03<br>=X) | 7N9 | 7.5 | mcg<br>+ A | up 2<br>A/H7<br>S03<br>=X) | 7N9 | 15 | mcg .<br>+ A | up 3<br>A/H7<br>S03<br>=X) | 'N9 | 15 | Gro<br>mcg<br>(N= | | /N9 | 45 | mcg | up 5<br>A/H7<br>=X) | | A | All Su<br>(N= | | ts |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| A a la-rain | | 19 | -64 | > | 65 | 19 | -64 | ≥ | 65 | 19 | -64 | ≥ | 65 | 19 | -64 | > | 65 | 19 | -64 | ≥ | 65 | 19 | -64 | // | 65 |
| Analysis<br>Populations | Reason Subjects Excluded | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Safety Population | Any Reason | х | xx | х | xx | x | xx | х | xx | х | xx | х | xx | х | xx | х | xx | х | xx | x | xx | х | xx | X | xx |
| | Study Vaccination 1 Not<br>Received | | | | | | | | | | | | | | | | | | | | | | | | |
| Modified Intent to<br>Treat | Any Reason | | | | | | | | | | | | | | | | | | | | | | | | |
| | Study Vaccination 1 Not<br>Received | | | | | | | | | | | | | | | | | | | | | | | | |
| | No Baseline Results<br>Available | | | | | | | | | | | | | | | | | | | | | | | | |
| | No Post-Vaccination Results<br>Available | | | | | | | | | | | | | | | | | | | | | | | | |
| Per-Protocol, Day | Any Reason | | | | | | | | | | | | | | | | | | | | | | | | |
| | Study Vaccination 1 Not<br>Received | | | | | | | | | | | | | | | | | | | | | | | | |
| | No Baseline Results<br>Available | | | | | | | | | | | | | | | | | | | | | | | | |
| | No Day 9 Result Reported<br>by Lab | | | | | | | | | | | | | | | | | | | | | | | | |
| | Lost to Follow-up Before<br>Day 9 | | | | | | | | | | | | | | | | | | | | | | | | |
| | Receipt of Non-Study<br>Vaccination | | | | | | | | | | | | | | | | | | | | | | | | |
| | Receipt of<br>Immunosuppressive<br>medication | | | | | | | | | | | | | | | | | | | | | | | | |

Table 16: Analysis Populations by Treatment Arm and Age Stratum, All Enrolled Subjects\* (continued)

| | | <br> | <br> | <br> | <br> | <br> |
|---|---|---|---|---|---|---|
| | Day 9 Visit Out of Window | | | | | |
| Per-Protocol, Day<br>22 | Any Reason | | | | | |
| | Study Vaccination 1 Not<br>Received | | | | | |
| | No Baseline Results<br>Available | | | | | |
| | No Day 21 Result Reported by Lab | | | | | |
| | Lost to Follow-up Before<br>Day 21 | | | | | |
| | Receipt of Non-Study<br>Vaccination | | | | | |
| | Receipt of<br>Immunosuppressive<br>medication | | | | | |
| | Day 21 Visit Out of Window | | | | | |
| Per-Protocol, Day<br>29 | Any Reason | | | | | |
| | Study Vaccination 1 Not<br>Received | | | | | |
| | Study Vaccination 2 Not<br>Received | | | | | |
| | Study Vaccination 2 Out of Window | | | | | |
| | No Baseline Results<br>Available | | | | | |
| | No Day 29 Result Reported by Lab | | | | | |
| | Lost to Follow-up Before<br>Day 29 | | | | | |

Table 16: Analysis Populations by Treatment Arm and Age Stratum, All Enrolled Subjects\* (continued)

| | Receipt of Non-Study<br>Vaccination |
|---|---|
| | Receipt of<br>Immunosuppressive<br>medication |
| | Day 29 Visit Out of Window |
| Per-Protocol, Day<br>43 | Any Reason |
| | Study Vaccination 1 Not<br>Received |
| | Study Vaccination 2 Not<br>Received |
| | Study Vaccination 2 Out of Window |
| | No Baseline Results<br>Available |
| | No Day 43 Result Reported by Lab |
| | Lost to Follow-up Before<br>Day 43 |
| | Receipt of Non-Study<br>Vaccination |
| | Receipt of<br>Immunosuppressive<br>medication |
| | Day 43 Visit Out of Window |

Table 17: Subject Disposition by Treatment Arm, All Enrolled Subjects\*

| | 3.75 mc + 1 | oup 1<br>eg A/H7N9<br>AS03<br>N=X) | 7.5 mcg<br>+ A | up 2<br>A/H7N9<br>S03<br>=X) | 15 mcg<br>+ A | up 3<br>A/H7N9<br>S03<br>=X) | 1<br>A | roup 4<br>5 mcg<br>/H7N9<br>N=X) | 45 mc | roup 5<br>eg A/H7N9<br>N=X) | | ubjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Disposition | n | % | n | % | n | % | n | % | n | % | n | % |
| Screened | х | | х | | х | | х | | х | | Х | |
| Enrolled/Randomized | х | 100 | х | 100 | х | 100 | х | 100 | х | 100 | х | 100 |
| Received Vaccination 1 | х | xx | х | xx | х | xx | х | XX | х | XX | X | xx |
| Received Vaccination 2 | х | xx | х | xx | х | xx | х | xx | х | XX | х | xx |
| Received All Scheduled Vaccinations <sup>a</sup> | | | | | | | | | | | | |
| Completed Blood Draw for Primary<br>Immunogenicity Analysis (Day 43) | | | | | | | | | | | | |
| Included in Per Protocol Primary Immunogenicity<br>Analysis (Day 43) <sup>b</sup> | | | | | | | | | | | | |
| Completed Primary Follow-up (Day 43) <sup>a</sup> | | | | | | | | | | | | |
| Completed Final Study Visit (Day 387) | | | | | | | | | | | | |

<sup>a</sup>Refer to Listing 2 for reasons subjects discontinued from study vaccinations or terminated early. <sup>b</sup>Refer to Listing 5 for reasons subjects are excluded from the per protocol population.

Table 18: Subject Disposition by Treatment Arm and Age Stratum, All Enrolled Subjects\*

| | 3.7 | Grou<br>75 mcg<br>+ AS<br>(N= | A/H7<br>803 | N9 | 7.5 | | | | | Grou<br>15 mcg A<br>+ AS<br>(N= | A/H7N<br>803 | 9 | 15 | Gro<br>5 mcg<br>(N= | A/H | | 45 | Grou<br>mcg A<br>(N= | \/H7 | N9 | | All Su<br>(N= | bjec<br>=X) | ts |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 19 | <b>)-64</b> | ≥ | 65 | 19 | -64 | 2 | ≥ 65 | 1 | 9-64 | ≥ | 65 | 19 | <b>)-64</b> | > | 65 | 19 | -64 | 2 | 65 | 19 | 9-64 | > | <u>2</u> 65 |
| Subject<br>Disposition | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Screened | х | | х | | х | | х | | х | | х | | Х | | X | | х | | х | | Х | | Х | |
| Enrolled/Randomized | х | 100 | х | 100 | х | 100 | х | 100 | х | 100 | х | 100 | Х | 100 | X | 100 | х | 100 | х | 100 | Х | 100 | Х | 100 |
| Received Vaccination 1 | х | XX | х | xx | х | xx | х | XX | х | xx | X | XX | х | XX | x | XX | X | XX | х | XX | х | XX | х | xx |
| Received Vaccination 2 | Х | xx | х | xx | х | XX | х | XX | х | XX | X | XX | х | XX | X | XX | X | XX | х | XX | Х | XX | X | XX |
| Received All Scheduled<br>Vaccinations <sup>a</sup> | X | xx | Х | xx | х | xx | х | xx | X | xx | X | XX | х | XX | x | XX | X | XX | х | xx | х | XX | х | xx |
| Completed Blood Draw for<br>Primary Immunogenicity<br>Analysis (Day 43) | x | xx | х | xx | х | xx | х | xx | x | xx | х | xx | x | xx | X | XX | х | xx | x | xx | x | xx | х | xx |
| Included in Per Protocol<br>Primary Immunogenicity<br>Analysis (Day 43) <sup>b</sup> | х | XX | х | xx | x | xx | х | xx | х | xx | X | XX | х | xx | x | XX | X | XX | х | xx | х | xx | х | xx |
| Completed Primary Follow-up (Day 43) <sup>a</sup> | х | XX | х | xx | X | xx | х | xx | х | xx | X | xx | х | xx | x | XX | Х | xx | х | xx | х | xx | х | xx |
| Completed Final Study Visit (Day 387) | x | XX | х | xx | X | xx | х | xx | х | xx | х | XX | х | XX | х | XX | х | XX | х | xx | х | xx | х | xx |

<sup>a</sup>Refer to Listing 2 for reasons subjects discontinued from study vaccinations or terminated early. <sup>b</sup>Refer to Listing 5 for reasons subjects are excluded from the per protocol population.

Table 19: Dates of First Study Vaccination by Site, Treatment Arm, and Age Stratum, for Safety Analysis Population

| | 3.75 | Group 1<br>mcg A/I<br>+ AS03<br>(N=X) | H7N9 | 7.5 r | Group 2<br>ncg A/H<br>+ AS03<br>(N=X) | 17N9 | 15 n | Group 3<br>ncg A/H<br>+ AS03<br>(N=X) | 7N9 | | Group 4<br>ncg A/H<br>(N=X) | | | Group :<br>ncg A/H<br>(N=X) | 17N9 | Al | ll Subjec<br>(N=X) | ets |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| <b>Dates of Dosing</b> | 19-64 | ≥ 65 | All | 19-64 | ≥ 65 | All | 19-64 | ≥ 65 | All | 19-64 | ≥ 65 | All | 19-64 | ≥ 65 | All | 19-64 | ≥ 65 | All |
| | | | | | | | [Site 1] | | | | | | | | | | | |
| Total (Entire period of enrollment) | х | X | Х | X | X | X | X | X | X | X | X | X | X | X | х | X | X | X |
| DDMMMYYYY-DDMMMYYYY | х | X | Х | X | X | X | X | X | X | X | X | X | X | X | х | X | X | X |
| | | | | | | | [Site 2] | | | | | | | | | | | |
| Total (Entire period of enrollment) | х | X | х | х | X | X | х | X | х | х | х | X | х | X | х | х | х | х |
| DDMMMYYYY-DDMMMYYYY | х | х | х | х | х | х | х | х | х | х | х | х | х | х | х | х | х | х |
| | | | | • | | [Repo | eat for al | ll sites] | | • | | | • | | | • | | |
| N= Number of subjects in the Safety | populatio | on. | | | | | | | | | | | | | | | | |

Table with similar format:

Table 20: Dates of Second Study Vaccination by Site, Treatment Arm, and Age Stratum, for Safety Analysis Population

### 14.1.2 Demographic Data

Table 21: Summary of Categorical Demographic and Baseline Characteristics by Site, All Enrolled Subjects

| | | Univ | ıke<br>ersity<br>=X) | | ory<br>=X) | Perm | iser<br>anente<br>=X) | of I | ersity<br>owa<br>=X) | Mar | ersity<br>of<br>yland<br>=X) | | te 6]<br>=X) | | Subjects<br>N=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Variable | Characteristic | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Age | 19-64 years | х | xx | х | XX | х | XX | х | XX | х | xx | х | xx | х | XX |
| | ≥ 65 years | | | | | | | | | | | | | | |
| Sex | Male | x | XX | x | XX | X | XX | x | XX | x | xx | X | xx | x | XX |
| | Female | | | | | | | | | | | | | | |
| BMI | < 30 | | | | | | | | | | | | | | |
| | ≥ 30 | | | | | | | | | | | | | | |
| Ethnicity | Not Hispanic or Latino | х | xx | х | XX | х | XX | х | XX | х | xx | х | xx | х | XX |
| | Hispanic or Latino | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | |
| | Unknown | | | | | | | | | | | | | | |
| Race | American Indian or Alaska Native | X | xx | x | XX | X | XX | x | xx | x | xx | X | xx | x | XX |
| | Asian | | | | | | | | | | | | | | |
| | Native Hawaiian or Other Pacific Islander | | | | | | | | | | | | | | |
| | Black or African American | | | | | | | | | | | | | | |
| | White | | | | | | | | | | | | | | |
| | Multi-Racial | | | | | | | | | | | | | | |
| | Unknown | | | | | | | | | | | | | | |
| Prior Seasonal Influenza<br>Vaccination | 2016-2017 and 2017-2018 | | | | | | | | | | | | | | |
| | 2016-2017 only | | | | | | | | | | | | | | |
| | 2017-2018 only | | | | | | | | | | | | | | |

| | | Univ | ıke<br>ersity<br>=X) | Em<br>(N= | | Kai<br>Perma<br>(N= | anente | Unive<br>of Ic | owa | Unive<br>o<br>Mary<br>(N= | f<br>/land | [Sit | _ | | Subjects<br>N=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Variable | Characteristic | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | Neither | | | | | | | | | | | | | | |
| | Unknown | | | | | | | | | · | | · | | | |
| N= Number of subjects enrolled | | | | | | | | - | | | - | | | • | |

Table 22: Summary of Continuous Demographic and Baseline Characteristics by Site, All Enrolled Subjects

| Variable | Statistic | [Site 1]<br>(N=X) | [Site 2]<br>(N=X) | [Site 3]<br>(N=X) | [Site 4]<br>(N=X) | [Site 5]<br>(N=X) | [Site 6]<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|
| Age | Mean | x.x | x.x | X.X | X.X | X.X | X.X | X.X |
| | Standard Deviation | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | Median | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | Minimum | Х | Х | X | Х | X | х | X |
| | Maximum | Х | X | X | X | X | х | X |
| BMI | Mean | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | Standard Deviation | X.X | X.X | X.X | x.x | X.X | X.X | X.X |
| | Median | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | Minimum | Х | Х | X | Х | X | X | X |
| | Maximum | Х | X | X | X | X | x | x |
| N= Number of subjects enro | olled | | | • | • | • | • | |

Table 23: Summary of Categorical Demographic and Baseline Characteristics by Treatment Arm, All Enrolled Subjects\*

| Variable<br>Sex | | 3.75<br>A/H<br>+ A | oup 1<br>5 mcg<br>17N9<br>AS03<br>=X) | 7.5 mcg<br>+ A | oup 2<br>A/H7N9<br>SS03<br>=X) | 15 mcg<br>+ A | oup 3<br>A/H7N9<br>AS03<br>=X) | 15 i<br>A/H | up 4<br>mcg<br>(7N9<br>=X) | 45 mcg | up 5<br>A/H7N9<br>=X) | All Subjects<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Characteristic | n | % | n | % | n | % | n | % | n | % | n | % |
| | Male | | | | | | | | | | | | |
| | Female | | | | | | | | | | | | |
| ВМІ | < 30 | | | | | | | | | | | | |
| | ≥30 | | | | | | | | | | | | |
| Ethnicity | Not Hispanic or Latino | | | | | | | | | | | | |
| | Hispanic or Latino | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | |
| | Unknown | | | | | | | | | | | | |
| Race | American Indian or Alaska Native | | | | | | | | | | | | |
| | Asian | | | | | | | | | | | | |
| | Native Hawaiian or Other Pacific<br>Islander | | | | | | | | | | | | |
| | Black or African American | | | | | | | | | | | | |
| | White | | | | | | | | | | | | |
| | Multi-Racial | | | | | | | | | | | | |
| | Unknown | | | | | | | | | | | | |
| Prior Seasonal Influenza<br>Vaccination | 2016-2017 and 2017-2018 | | | | | | | | | | | | |
| | 2016-2017 only | | | | | | | | | | | | |
| | 2017-2018 only | | | | | | | | | | | | |

| | | 3.75<br>A/H<br>+ A | Group 1<br>3.75 mcg<br>A/H7N9<br>+ AS03<br>(N=X) | | up 2<br>A/H7N9<br>S03<br>=X) | Gro 15 mcg . + A (N= | A/H7N9<br>S03 | Gro<br>15 i<br>A/H<br>(N= | ncg<br>7N9 | Grov<br>45 mcg /<br>(N= | A/H7N9 | All Subjects<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Variable | Characteristic | n % | | n | % | n | % | n | % | n | % | n | % |
| | Neither | | | | | | | | | | | | |
| | Unknown | | | | | | | | | | | | |
| N=Number of subjects er | rolled | | • | • | | | • | | | | | | |

Table 24: Summary of Categorical Demographic and Baseline Characteristics by Treatment Arm and Age Stratum, All Enrolled Subjects\*

| | | Group 1<br>3.75 meg A/H7N9<br>+ AS03<br>(N=X) | | | Group 2<br>7.5 mcg A/H7N9<br>+ AS03<br>(N=X) | | | | Group 3<br>15 mcg A/H7N9<br>+ AS03<br>(N=X) | | | | Group 4<br>15 mcg A/H7N9<br>(N=X) | | | | Group 5<br>45 mcg A/H7N9<br>(N=X) | | | | All Subjects<br>(N=X) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Variable | | 19-64 | | ≥ 65 | | 19 | 19-64 | | ≥ 65 | | 19-64 | | ≥ 65 | | 19-64 | | ≥ 65 | | -64 | ≥ 65 | | 19-64 | | ≥ 65 | |
| | Characteristic | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Sex | Male | | | | | | | | | | | | | | | | | | | | | | | | |
| | Female | | | | | | | | | | | | | | | | | | | | | | | | |
| BMI | < 30 | | | | | | | | | | | | | | | | | | | | | | | | |
| | ≥ 30 | | | | | | | | | | | | | | | | | | | | | | | | |
| Ethnicity | Not Hispanic or Latino | | | | | | | | | | | | | | | | | | | | | | | | |
| | Hispanic or Latino | | | | | | | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | | | | | | | |
| | Unknown | | | | | | | | | | | | | | | | | | | | | | | | |
| Race | American Indian or<br>Alaska Native | | | | | | | | | | | | | | | | | | | | | | | | |
| | Asian | | | | | | | | | | | | | | | | | | | | | | | | |
| | Native Hawaiian or Other<br>Pacific Islander | | | | | | | | | | | | | | | | | | | | | | | | |
| | Black or African<br>American | | | | | | | | | | | | | | | | | | | | | | | | |
| | White | | | | | | | | | | | | | | | | | | | | | | | | |
| | Multi-Racial | | | | | | | | | | | | | | | | | | | | | | | | |
| | Unknown | | | | | | | | | | | | | | | | | | | | | | | | |
| Prior Seasonal<br>Influenza<br>Vaccination | 2016-2017 and 2017-2018 | | | | | | | | | | | | | | | | | | | | | | | | |
Table 24: Summary of Categorical Demographic and Baseline Characteristics by Treatment Arm and Age Stratum, All Enrolled Subjects (continued)

| | | 3.7 | 75 mcg<br>+ A | up 1<br>g A/H<br>S03<br>=X) | 7N9 | 7.5 | Gro<br>mcg<br>+ A<br>(N= | S03 | | 15 | Grown Hand | A/H7 | N9 | 15 | mcg . | up 4<br>A/H7<br>=X) | N9 | 45 | Gro<br>mcg<br>(N= | | N9 | | All Si<br>(N | ıbject<br>=X) | ts |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 19 | <b>)-64</b> | ≥ | 65 | 19 | -64 | ≥ | 65 | 19 | -64 | ≥ | 65 | 19 | -64 | ≥ | 65 | 19 | -64 | ≥ | 65 | 19 | -64 | ≥ | 65 |
| Variable | Characteristic | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | 2016-2017 only | | | | | | | | | | | | | | | | | | | | | | | | |
| | 2017-2018 only | | | | | | | | | | | | | | | | | | | | | | | | |
| | Neither | | | | | | | | | | | | | | | | | | | | | | | | |
| | Unknown | | | | | | | | | | | | | | | | | | | | | | | | |

Table 25: Summary of Continuous Baseline Characteristics by Treatment Arm, All Enrolled Subjects\*

| Variable | Statistic | Group 1<br>3.75 mcg A/H7N9<br>+ AS03<br>(N=X) | Group 2<br>7.5 mcg A/H7N9<br>+ AS03<br>(N=X) | Group 3<br>15 mcg A/H7N9<br>+ AS03<br>(N=X) | Group 4<br>15 mcg A/H7N9<br>(N=X) | Group 5<br>45 mcg A/H7N9<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|
| Age | Mean | X.X | X.X | X.X | x.x | x.x | X.X |
| | Standard Deviation | X.X | X.X | X.X | X.X | x.x | x.x |
| | Median | x | X | X | X | X | x |
| | Minimum | x | X | X | X | X | x |
| | Maximum | x | X | X | X | X | x |
| BMI | Mean | x.x | X.X | X.X | x.x | x.x | x.x |
| | Standard Deviation | X.X | X.X | X.X | X.X | X.X | X.X |
| | Median | x | X | X | X | X | х |
| | Minimum | x | X | X | X | X | х |
| | Maximum | x | X | X | X | X | х |
| N=Number of su | | X | X | X | X | X | Х |

Table 26: Summary of Continuous Baseline Characteristics by Treatment Arm and Age Stratum, All Enrolled Subjects\*

| | 3.75 mcg<br>+ A | A/H7N9<br>S03 | 7.5 mcg<br>+ A | A/H7N9<br>S03 | 15 mcg<br>+ A | A/H7N9<br>S03 | 15 mcg | A/H7N9 | 45 mcg | A/H7N9 | | ıbjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Statistic | 19-64 | ≥ 65 | 19-64 | ≥ 65 | 19-64 | ≥ 65 | 19-64 | ≥ 65 | 19-64 | ≥ 65 | 19-64 | ≥ 65 |
| Mean | x.x | x.x | x.x | x.x | x.x | x.x | x.x | x.x | x.x | x.x | x.x | X.X |
| Standard Deviation | x.x | x.x | x.x | x.x | x.x | x.x | x.x | x.x | x.x | x.x | x.x | X.X |
| Median | х | X | x | x | x | x | x | x | x | x | x | X |
| Minimum | х | X | x | x | x | x | x | x | x | x | x | X |
| Maximum | х | X | x | x | x | x | x | x | x | x | x | X |
| Mean | x.x | x.x | x.x | x.x | x.x | x.x | x.x | x.x | x.x | x.x | x.x | X.X |
| Standard Deviation | x.x | x.x | x.x | x.x | x.x | x.x | x.x | x.x | x.x | x.x | x.x | X.X |
| Median | х | X | х | х | х | х | х | х | х | х | х | X |
| Minimum | х | x | x | x | х | х | x | x | х | х | х | X |
| Maximum | х | Х | Х | Х | Х | Х | Х | X | х | Х | х | х |
| | Mean Standard Deviation Median Minimum Maximum Mean Standard Deviation Median Minimum | 3.75 mcg + A (N= Statistic 19-64 Mean x.x Standard Deviation x.x Median x Minimum x Maximum x Mean x.x Standard Deviation x.x Median x Minimum x Mean x.x Standard Deviation x.x Minimum x | Mean x.x x.x Standard Deviation x.x x.x Median x x Minimum x x Maximum x x Mean x.x x.x Standard Deviation x.x x.x Median x x Minimum x x | $ \begin{array}{c ccccccccccccccccccccccccccccccccccc$ | $ \begin{array}{c ccccccccccccccccccccccccccccccccccc$ | $ \begin{array}{c ccccccccccccccccccccccccccccccccccc$ | $ \begin{array}{c ccccccccccccccccccccccccccccccccccc$ | 3.75 mcg A/H7N9 + AS03 (N=X) 7.5 mcg A/H7N9 + AS03 (N=X) 15 mcg A/H7N9 + AS03 (N=X) 15 mcg A/H7N9 + AS03 (N=X) Statistic 19-64 ≥ 65 19-64 ≥ 65 19-64 ≥ 65 19-64 Mean x.x Standard Deviation x.x x.x x.x x.x x.x x.x x.x Median x x x x x x x Maximum x x x x x x x Mean x.x x.x x.x x x x x Mean x.x x.x x.x x.x x.x x x x Standard Deviation x.x x.x x.x x.x x x x x Median x x x x x x x x Minimum x x x x x x x | 3.75 mcg A/H7N9 + AS03 (N=X) 7.5 mcg A/H7N9 + AS03 (N=X) 15 mcg A/H7N9 + AS03 (N=X) 15 mcg A/H7N9 (N=X) Statistic 19-64 ≥ 65 19-64 ≥ 65 19-64 ≥ 65 19-64 ≥ 65 Mean x.x Standard Deviation x.x Median x x x x x x x x x Maximum x x x x x x x x x Mean x.x x.x x.x x.x x x x x x Mean x.x Standard Deviation x.x Median x x x x x x x x x Median x x x x x x x x x | 3.75 mcg A/H7N9 + AS03 (N=X) 7.5 mcg A/H7N9 + AS03 (N=X) 15 mcg A/H7N9 + AS03 (N=X) 15 mcg A/H7N9 (N=X) 45 mcg (N=X) Statistic 19-64 ≥ 65 19-64 ≥ 65 19-64 ≥ 65 19-64 ≥ 65 19-64 ≥ 65 19-64 ≥ 65 19-64 Mean x.x < | 3.75 mcg A/H7N9 | 3.75 mcg A/H7N9 |

### 14.1.3 Summary of Prior or Concurrent Medical Conditions

Table 27: Summary of Subjects with Prior or Concurrent Medical Conditions by MedDRA System Organ Class and Treatment Arm, Safety Analysis Population

| | 3.75 mcg<br>+ A | up 1<br>g A/H7N9<br>sS03<br>=X) | 7.5 mcg<br>+ A | up 2<br>A/H7N9<br>.S03<br>=X) | 15 mcg<br>+ A | up 3<br>A/H7N9<br>S03<br>=X) | Gro<br>15 mcg .<br>(N= | A/H7N9 | Grod<br>45 mcg /<br>(N= | | All Su<br>(N= | bjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| MedDRA System Organ Class | n | % | n | % | n | % | n | % | n | % | n | % |
| Any SOC | X | XX | X | XX | X | XX | X | xx | x | XX | х | xx |
| [SOC 1] | х | XX | x | xx | X | xx | X | XX | X | XX | х | xx |
| [SOC 2] | Х | XX | х | XX | Х | XX | X | XX | х | xx | х | xx |

Note: N=Number of subjects in the Safety population;

n = Number of subjects reporting medical history within the specified SOC. A subject is only counted once per SOC.

Table 28: Summary of Subjects with Prior or Concurrent Medical Conditions by MedDRA System Organ Class, Treatment Arm and Age Stratum, Safety Analysis Population

| | 3.7 | Gro<br>75 mcg<br>+ A<br>(N= | A/H7<br>S03 | N9 | 7.5 | Gro<br>5 mcg<br>+ A<br>(N= | S03 | N9 | 15 | Gro<br>5 mcg<br>+ A<br>(N= | S03 | N9 | 15 | Gro<br>5 mcg<br>(N= | A/H71 | N9 | 45 | Gro<br>mcg<br>(N= | | N9 | | | ibjects<br>=X) | i |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| MedDRA System Organ | 19 | -64 | ≥ | 65 | 19 | -64 | ≥ | 65 | 19 | -64 | ≥ | 65 | 19 | -64 | ≥ | 65 | 19 | -64 | ≥ | 65 | 19 | -64 | 2 | 65 |
| Class | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Any SOC | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | х | XX |
| [SOC 1] | X | XX | X | XX | Х | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX |
| [SOC 2] | X | xx | X | XX | X | XX | X | xx | X | XX | X | XX | X | xx | X | XX | X | XX | X | XX | X | XX | X | XX |

Note: N=Number of subjects in the Safety population;

n = Number of subjects reporting medical history within the specified SOC. A subject is only counted once per SOC.

## 14.2 Immunogenicity Tables

## 14.2.1 Immune Response Against 2017 A/H7N9

Table 29: Summaries of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by Study Day and Treatment Arm, Modified Intent-to-Treat Population\*†;

| Time Point | Group 1<br>3.75 mcg A/H7N9<br>+ AS03<br>(N=X) | Group 2<br>7.5 mcg A/H7N9<br>+ AS03<br>(N=X) | Group 3<br>15 mcg A/H7N9<br>+ AS03<br>(N=X) | Group 4<br>15 mcg A/H7N9<br>(N=X) | Group 5<br>45 mcg A/H7N9<br>(N=X) |
|---|---|---|---|---|---|
| Day 1 (Pre-Vaccination 1) | | | | | |
| n | Х | х | х | х | х |
| GMT (95% CI) <sup>a</sup> | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) |
| Titer ≥ 1:40 - %(95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| 7 Days Post Vaccination 1 | | | | | |
| n | Х | х | х | х | х |
| GMT (95% CI) <sup>a</sup> | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) |
| Titer ≥ 1:40 - %(95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| GMFR (95% CI) <sup>a</sup> | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) |
| Seroconversion - % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| 21 Days Post Vaccination 1 | | | | | |
| n | Х | х | х | х | х |
| GMT (95% CI) <sup>a</sup> | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) |
| Titer ≥ 1:40 - %(95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| GMFR (95% CI) <sup>a</sup> | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) |
| Seroconversion - % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| 7 Days Post Vaccination 2 | | | | | |
| n | х | х | x | x | х |
| GMT (95% CI) <sup>a</sup> | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) |
| Titer ≥ 1:40 - %(95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |

Table 29: Summaries of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by Study Day and Treatment Arm, Modified Intent-to-Treat Population (continued)

| Time Point | Group 1<br>3.75 mcg A/H7N9<br>+ AS03<br>(N=X) | Group 2<br>7.5 mcg A/H7N9<br>+ AS03<br>(N=X) | Group 3<br>15 mcg A/H7N9<br>+ AS03<br>(N=X) | Group 4<br>15 mcg A/H7N9<br>(N=X) | Group 5<br>45 mcg A/H7N9<br>(N=X) |
|---|---|---|---|---|---|
| GMFR (95% CI) <sup>a</sup> | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) |
| Seroconversion - % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| 21 Days Post Vaccination 2 | | | | | |
| n | X | X | X | X | Х |
| GMT (95% CI) <sup>a</sup> | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) |
| Titer ≥ 1:40 - %(95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| GMFR (95% CI) <sup>a</sup> | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) |
| Seroconversion - % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| 180 Days Post Vaccination 2 | | | | | |
| n | х | х | х | x | х |
| GMT (95% CI) <sup>a</sup> | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) |
| Titer ≥ 1:40 - %(95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| GMFR (95% CI) <sup>a</sup> | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) |
| Seroconversion - % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |

N=number of subjects in the Modified Intent to Treat population; n = number of subjects with available results; GMT = Geometric Mean Titer; GMFR = Geometric Mean Fold Rise <sup>a</sup> Confidence Interval calculated based on the student's T distribution.

Tables with similar format

Table 30: Summaries of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by Study Day and Treatment Arm, Per Protocol Population\*;

Table 31: Summaries of Neutralizing Antibody Against 2017 A/H7N9 by Study Day and Treatment Arm, Modified Intent-to-Treat Population\*†‡

Table 32: Summaries of Neutralizing Antibody Against 2017 A/H7N9 by Study Day and Treatment Arm, Per Protocol Population\*‡

<sup>&</sup>lt;sup>b</sup> Exact binomial confidence interval calculated using the Clopper-Pearson methodology.

Table 33: Summaries of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by Study Day, Treatment Arm and Age Stratum, Modified Intent-to-Treat Population\*†‡

| | Gro<br>3.75 mcg<br>+ A<br>(N= | A/H7N9<br>S03 | 7.5 mcg<br>+ A | up 2<br>A/H7N9<br>S03<br>=X) | 15 mcg<br>+ A | up 3<br>A/H7N9<br>S03<br>=X) | 15 mcg | up 4<br>A/H7N9<br>=X) | Group 5<br>45 mcg A/H7N9<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | 19-64 | ≥ 65 | 19-64 | ≥ 65 | 19-64 | ≥ 65 | 19-64 | ≥ 65 | 19-64 | ≥ 65 |
| Day 1 (Pre Vaccination 1) | | | | | | | | | | |
| n | X | X | X | X | X | X | X | X | X | X |
| GMT (95% CI) <sup>a</sup> | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) |
| Titer $\ge 1:40 - \% (95\% \text{ CI})^b$ | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| 7 Days Post Vaccination 1 | | | | | | | | | | |
| n | X | X | X | X | X | X | X | X | X | X |
| GMT (95% CI) <sup>a</sup> | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) |
| Titer $\geq 1:40 - \% (95\% \text{ CI})^b$ | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| GMFR (95% CI) <sup>a</sup> | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) |
| Seroconversion - % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| 21 Days Post Vaccination 1 | | | | | | | | | | |
| n | X | X | X | X | X | X | X | X | X | X |
| GMT (95% CI) <sup>a</sup> | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) |
| Titer $\geq 1:40 - \% (95\% \text{ CI})^b$ | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| GMFR (95% CI) <sup>a</sup> | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) |
| Seroconversion - % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| 7 Days Post Vaccination 2 | | | | | | | | | | |

Table 33: Summaries of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by Study Day, Treatment Arm and Age Stratum, Modified Intent-to-Treat Population (continued)

| | Gro<br>3.75 mcg<br>+ A<br>(N= | A/H7N9<br>S03 | Gro<br>7.5 mcg<br>+ A<br>(N= | A/H7N9<br>S03 | 15 mcg<br>+ A | up 3<br>A/H7N9<br>S03<br>=X) | | up 4<br>A/H7N9<br>=X) | Group 5<br>45 mcg A/H7N9<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | 19-64 | ≥ 65 | 19-64 | ≥ 65 | 19-64 | ≥ 65 | 19-64 | ≥ 65 | 19-64 | ≥ 65 |
| n | X | X | Х | X | x | х | X | X | X | X |
| GMT (95% CI) <sup>a</sup> | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) |
| Titer $\ge 1:40 - \% (95\% \text{ CI})^b$ | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| GMFR (95% CI) <sup>a</sup> | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) |
| Seroconversion - % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| 21 Days Post Vaccination 2 | | | | | | | | | | |
| n | X | X | X | X | X | X | X | X | X | X |
| GMT (95% CI) <sup>a</sup> | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) |
| Titer $\ge 1:40 - \% (95\% \text{ CI})^b$ | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| GMFR (95% CI) <sup>a</sup> | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) |
| Seroconversion - % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| 180 Days Post Vaccination<br>2 | | | | | | | | | | |
| n | X | X | Х | X | x | x | X | X | X | X |
| GMT (95% CI) <sup>a</sup> | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) |
| Titer $\geq 1:40 - \% (95\% \text{ CI})^b$ | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| GMFR (95% CI) <sup>a</sup> | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) |

Table 33: Summaries of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by Study Day, Treatment Arm and Age Stratum, Modified Intent-to-Treat Population (continued)

| | Gro<br>3.75 mcg<br>+ A<br>(N= | A/H7N9<br>S03 | | | 15 mcg + A | up 3<br>A/H7N9<br>S03<br>=X) | Gro<br>15 mcg<br>(N= | A/H7N9 | 45 mcg | up 5<br>A/H7N9<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | 19-64 | ≥ 65 | 19-64 | ≥ 65 | 19-64 | ≥ 65 | 19-64 | ≥65 | 19-64 | ≥65 |
| Seroconversion - % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |

- Table 34: Summaries of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by Study Day, Treatment Arm and Age Stratum, Per Protocol Population\*:
- Table 35: Summaries of Neutralizing Antibody Against 2017 A/H7N9 by Study Day, Treatment Arm and Age Stratum, Modified Intent-to-Treat Population\*†‡
- Table 36: Summaries of Neutralizing Antibody Against 2017 A/H7N9 by Study Day, Treatment Arm and Age Stratum, Per Protocol Population\*‡

<sup>&</sup>lt;sup>a</sup> Confidence Interval calculated based on the student's T distribution.

<sup>&</sup>lt;sup>b</sup> Exact binomial confidence interval calculated using the Clopper-Pearson methodology.

Table 37: Summary of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by Treatment Arm and Age Categories at 21 Days Post Second Vaccination, Per-Protocol Population\*

| | Group 1<br>3.75 mcg A/H7N9<br>+ AS03<br>(N=X) | Group 2<br>7.5 mcg A/H7N9<br>+ AS03<br>(N=X) | Group 3<br>15 mcg A/H7N9<br>+ AS03<br>(N=X) | Group 4<br>15 mcg A/H7N9<br>(N=X) | Group 5<br>45 mcg A/H7N9<br>(N=X) |
|---|---|---|---|---|---|
| Age 19-34 years | | | | | |
| n | x | X | х | X | х |
| GMT (95% CI) <sup>a</sup> | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) |
| Titer ≥ 1:40 - % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| GMFR (95% CI) <sup>a</sup> | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) |
| Seroconversion - % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| Age 35-49 years | | | | | |
| n | x | X | х | X | х |
| GMT (95% CI) <sup>a</sup> | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) |
| Titer ≥ 1:40 - % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| GMFR (95% CI) <sup>a</sup> | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) |
| Seroconversion - % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| Age 50-64 years | | | | | |
| n | x | X | х | X | х |
| GMT (95% CI) <sup>a</sup> | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) |
| Titer ≥ 1:40 - % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| GMFR (95% CI) <sup>a</sup> | | | | | |
| Seroconversion - % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| Age 65-80 years | | | | | |
| n | x | X | х | x | х |
| GMT (95% CI) <sup>a</sup> | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) |
| Titer ≥ 1:40 - % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| GMFR (95% CI) <sup>a</sup> | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x) |

Table 37: Summary of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by Treatment Arm and Age Categories at 21 Days Post Second Vaccination, Per-Protocol Population (continued)

| | Group 1<br>3.75 mcg A/H7N9<br>+ AS03<br>(N=X) | Group 2<br>7.5 mcg A/H7N9<br>+ AS03<br>(N=X) | Group 3<br>15 mcg A/H7N9<br>+ AS03<br>(N=X) | Group 4<br>15 mcg A/H7N9<br>(N=X) | Group 5<br>45 mcg A/H7N9<br>(N=X) |
|---|---|---|---|---|---|
| Seroconversion - % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| Age≥81 years | | | | | |
| n | X | X | X | X | X |
| GMT (95% CI) <sup>a</sup> | xxx.x (xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) |
| Titer ≥ 1:40 - % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| GMFR (95% CI) <sup>a</sup> | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) | xxx.x(xxx.x,xxx.x) |
| Seroconversion - % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |

<sup>&</sup>lt;sup>a</sup> Confidence Interval calculated based on the student's T distribution.

<sup>&</sup>lt;sup>b</sup> Exact binomial confidence interval calculated using the Clopper-Pearson methodology.

- Table 38: Summary of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by Treatment Arm and Age Stratum at 180 Days Post Second Vaccination, Per-Protocol Population\*
- Table 39: Summary of Neutralizing Antibody Against 2017 A/H7N9 by Treatment Arm and Age Stratum at 21 Days Post Second Vaccination, Per-Protocol Population\*
- Table 40: Summary of Neutralizing Antibody Against 2017 A/H7N9 by Treatment Arm and Age Stratum at 180 Days Post Second Vaccination, Per-Protocol Population\*

Table 41: Summary of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by Treatment Arm, Age Stratum and Sex at 21 Days Post Second Vaccination, Per-Protocol Population\*

| | Gro<br>3.75 mcg<br>+ A<br>(N= | A/H7N9 | Group 2<br>7.5 mcg A/H7N9<br>+ AS03<br>(N=X) | | Group 3<br>15 mcg A/H7N9<br>+ AS03<br>(N=X) | | 15 mcg | oup 4<br>A/H7N9<br>=X) | Group 5<br>45 mcg A/H7N9<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|
| | 19-64 | ≥65 | 19-64 | ≥ 65 | 19-64 | ≥ 65 | 19-64 | ≥ 65 | 19-64 | ≥ 65 |
| Female | | | | | | | | | | |
| n | X | Х | X | X | X | X | х | X | Х | х |
| GMT (95% CI) <sup>a</sup> | XXX.X<br>(XXX.X,XXX.X) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) |
| Titer $\ge 1:40 - \% (95\% \text{ CI})^b$ | xx(xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| GMFR (95% CI) <sup>a</sup> | XXX.X<br>(XXX.X,XXX.X) | XXX.X<br>(XXX.X,XXX.X) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) |
| Seroconversion - % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| Male | | | | | | | | | | |
| n | Х | Х | X | X | X | Х | х | Х | Х | х |
| GMT (95% CI) <sup>a</sup> | XXX.X<br>(XXX.x,XXX.X) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) |
| Titer ≥ 1:40 - % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| GMFR (95% CI) <sup>a</sup> | XXX.X<br>(XXX.x,XXX.X) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) |
| Seroconversion - % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |

<sup>&</sup>lt;sup>a</sup> Confidence Interval calculated based on the student's T distribution.

<sup>&</sup>lt;sup>b</sup> Exact binomial confidence interval calculated using the Clopper-Pearson methodology.

- Table 41: Summary of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by Treatment Arm, Age Stratum and Sex at 21 Days Post Second Vaccination, Per-Protocol Population (continued)
- Table 42: Summary of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by Treatment Arm, Age Stratum and Sex at 180 Days Post Second Vaccination, Per-Protocol Population\*
- Table 43: Summary of Neutralizing Antibody Against 2017 A/H7N9 by Treatment Arm, Age Stratum and Sex at 21 Days Post Second Vaccination, Per-Protocol Population\*
- Table 44: Summary of Neutralizing Antibody Against 2017 A/H7N9 by Treatment Arm, Age Stratum and Sex at 180 Days Post Second Vaccination, Per-Protocol Population\*

Table 45: Summary of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by Treatment Arm, Age Stratum and BMI at 21 Days Post Second Vaccination, Per-Protocol Population\*

| | + A | up 1<br>3 A/H7N9<br>3 S03<br>=X) | 7.5 mcg<br>+ A | up 2<br>A/H7N9<br>.S03<br>=X) | Gro<br>15 mcg<br>+ A<br>(N= | A/H7N9<br>S03 | 15 mcg | up 4<br>A/H7N9<br>=X) | 45 mcg | up 5<br>A/H7N9<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|
| | 19-64 | ≥ 65 | 19-64 | ≥ 65 | 19-64 | ≥ 65 | 19-64 | ≥ 65 | 19-64 | ≥ 65 |
| BMI < 30 | | | | | | | | | | |
| n | X | X | X | x | X | X | x | x | X | х |
| GMT (95%<br>CI) <sup>a</sup> | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | XXX.X<br>(XXX.X,XXX.X) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) |
| Titer ≥ 1:40 - %<br>(95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| GMFR (95% CI) <sup>a</sup> | xxx.x<br>(xxx.x,xxx.x) | | | | | | | | | |
| Seroconversion<br>- % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| BMI ≥ 30 | | | | | | | | | | |
| n | X | X | X | х | X | X | Х | X | X | X |
| GMT (95%<br>CI) <sup>a</sup> | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) |
| Titer ≥ 1:40 - %<br>(95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| GMFR (95% CI) <sup>a</sup> | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) |
| Seroconversion<br>- % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| | 1 | l | TD 1 1 | I | 1 1 1 1 1 1 | 21 1 1 1 1. | C) (T) C | · 16 m | CL (ED. C | |

<sup>&</sup>lt;sup>a</sup> Confidence Interval calculated based on the student's T distribution.

<sup>&</sup>lt;sup>b</sup> Exact binomial confidence interval calculated using the Clopper-Pearson methodology.

Table 45: Summary of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by Treatment Arm, Age Stratum and BMI at 21 Days Post Second Vaccination, Per-Protocol Population (continued)

- Table 46: Summary of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by Treatment Arm, Age Stratum and BMI at 180 Days Post Second Vaccination, Per-Protocol Population\*
- Table 47: Summary of Neutralizing Antibody Against 2017 A/H7N9 by Treatment Arm, Age Stratum and BMI at 21 Days Post Second Vaccination, Per-Protocol Population\*
- Table 48: Summary of Neutralizing Antibody Against 2017 A/H7N9 by Treatment Arm, Age Stratum and BMI at 180 Days Post Second Vaccination, Per-Protocol Population\*

Table 49: Summary of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by Treatment Arm, Age Stratum and Prior Seasonal Influenza Vaccination at 21 Days Post Second Vaccination, Per-Protocol Population\*

| | Gro<br>3.75 mcg<br>+ A<br>(N= | A/H7N9<br>S03 | Group 2<br>7.5 mcg A/H7N9<br>+ AS03<br>(N=X) | | 15 mcg<br>+ A | Group 3<br>15 mcg A/H7N9<br>+ AS03<br>(N=X) | | up 4<br>A/H7N9<br>=X) | 45 mcg | up 5<br>A/H7N9<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|
| | 19-64 | ≥ 65 | 19-64 | ≥ 65 | 19-64 | ≥ 65 | 19-64 | ≥ 65 | 19-64 | ≥ 65 |
| Did Not Receive 2016-2017<br>or 2017-2018 Seasonal<br>Influenza Vaccination | | | | | | | | | | |
| n | X | X | X | X | X | X | X | X | X | X |
| GMT (95% CI) <sup>a</sup> | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) |
| Titer ≥ 1:40 - % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| GMFR (95% CI) <sup>a</sup> | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) |
| Seroconversion - % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| Received 2016-2017 and/or<br>2017-2018 Seasonal<br>Influenza Vaccination | | | | | | | | | | |
| n | Х | X | X | X | X | X | X | X | X | X |
| GMT (95% CI) <sup>a</sup> | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) |
| Titer ≥ 1:40 - % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| GMFR (95% CI) <sup>a</sup> | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) |
| Seroconversion - % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |

<sup>&</sup>lt;sup>a</sup> Confidence Interval calculated based on the student's T distribution.

<sup>&</sup>lt;sup>b</sup> Exact binomial confidence interval calculated using the Clopper-Pearson methodology.

- Table 50: Summary of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by Treatment Arm, Age Stratum and Prior Seasonal Influenza Vaccination at 180 Days Post Second Vaccination, Per-Protocol Population\*
- Table 51: Summary of Neutralizing Antibody Against 2017 A/H7N9 by Treatment Arm, Age Stratum and Prior Seasonal Influenza Vaccination at 21 Days Post Second Vaccination, Per-Protocol Population\*
- Table 52: Summary of Neutralizing Antibody Against 2017 A/H7N9 by Treatment Arm, Age Stratum and Prior Seasonal Influenza Vaccination at 180 Days Post Second Vaccination, Per-Protocol Population\*

Table 53: Logistic Regression Model to Evaluate the Relationship of HA Antigen Dose and AS03 Adjuvant with HAI Seroconversion Against 2017 A/H7N9 at 21 Days Post Second Study Vaccination, Per Protocol Population\*

| Model Parameter | Parameter Levels | Parameter<br>Estimate | SE | p-value | Odds Ratio | 95%CI |
|---|---|---|---|---|---|---|
| Treatment | 3.75 mcg with AS03 Adjuvant (reference) | - | - | - | - | - |
| | 7.5 mcg with AS03 Adjuvant | XXX.X | xxx.x | x.xxx | xx.x | xx.x-xx.x |
| | 15 mcg with AS03 Adjuvant | xxx.x | xxx.x | x.xxx | xx.x | xx.x-xx.x |
| | 15 mcg without AS03 Adjuvant | xxx.x | xxx.x | x.xxx | xx.x | xx.x-xx.x |
| | 45 mcg without AS03 Adjuvant | xxx.x | xxx.x | x.xxx | xx.x | xx.x-xx.x |
| Age | 19-64 years (reference) | - | - | - | - | - |
| | ≥65 years | XXX.X | xxx.x | x.xxx | xx.x | xx.x-xx.x |
| Interaction: Age*Treatment | Age*3.75 mcg with AS03 Adjuvant | - | - | - | - | - |
| | Age*7.5 mcg with AS03 Adjuvant | XXX.X | xxx.x | x.xxx | xx.x | xx.x-xx.x |
| | Age*15 mcg with AS03 Adjuvant | XXX.X | xxx.x | x.xxx | xx.x | xx.x-xx.x |
| | Age*15 mcg without AS03 Adjuvant | XXX.X | xxx.x | x.xxx | xx.x | xx.x-xx.x |
| | Age*45 mcg without AS03 Adjuvant | XXX.X | xxx.x | X.XXX | xx.x | xx.x-xx.x |
| | Age*3.75 mcg with AS03 adjuvant | - | - | - | - | - |

N = XX subjects with results available at 21 days post second vaccination in the per protocol population. XX subjects missing covariate data were excluded from this analysis.

P-value for Treatment = 0.XXX; P-value for Age = 0.XXX; P-value for interaction of Treatment and Age = 0.XXX.

- Table 54: Logistic Regression Model to Evaluate the Relationship of HA Antigen Dose and AS03 Adjuvant with Neut Seroconversion Against 2017 A/H7N9 at 21 Days Post Second Study Vaccination, Per Protocol Population\*
- Table 55: Logistic Regression Model to Evaluate the Relationship of HA Antigen Dose and AS03 Adjuvant with HAI Seroconversion Against 2017 A/H7N9 at 180 Days Post Second Study Vaccination, Per Protocol Population\*
- Table 56: Logistic Regression Model to Evaluate the Relationship of HA Antigen Dose and AS03 Adjuvant with Neut Seroconversion Against 2017 A/H7N9 at 180 Days Post Second Study Vaccination, Per Protocol Population\*

Table 57: Logistic Regression Model to Evaluate the Relationship of HA Antigen Dose and AS03 Adjuvant with HAI Seroconversion Against 2017 A/H7N9 at 21 Days Post Second Study Vaccination, Adjusted for Baseline Covariates, Per Protocol Population\*

| Model Parameter | Parameter Levels | Parameter<br>Estimate | SE | p-value | Odds Ratio | 95%CI |
|---|---|---|---|---|---|---|
| Intercept | - | XXX.X | xxx.x | x.xxx | - | - |
| Treatment | 3.75 mcg with AS03 Adjuvant (reference) | - | - | - | - | - |
| | 7.5 mcg with AS03 Adjuvant | xxx.x | xxx.x | x.xxx | XX.X | xx.x-xx.x |
| | 15 mcg with AS03 Adjuvant | xxx.x | xxx.x | x.xxx | XX.X | xx.x-xx.x |
| | 15 mcg without AS03 Adjuvant | xxx.x | xxx.x | x.xxx | XX.X | xx.x-xx.x |
| | 45 mcg without AS03 Adjuvant | XXX.X | xxx.x | x.xxx | xx.x | xx.x-xx.x |
| Age | 19-64 years (reference) | - | - | - | - | - |
| | ≥65 years | XXX.X | xxx.x | x.xxx | xx.x | xx.x-xx.x |
| Interaction: Age*Treatment | Age*3.75 mcg with AS03 Adjuvant | - | - | - | - | - |
| | Age*7.5 mcg with AS03 Adjuvant | XXX.X | xxx.x | x.xxx | xx.x | xx.x-xx.x |
| | Age*15 mcg with AS03 Adjuvant | XXX.X | xxx.x | x.xxx | xx.x | xx.x-xx.x |
| | Age*15 mcg without AS03 Adjuvant | XXX.X | xxx.x | x.xxx | xx.x | xx.x-xx.x |
| | Age*45 mcg without AS03 Adjuvant | XXX.X | xxx.x | x.xxx | xx.x | xx.x-xx.x |
| Sex | Female (reference) | - | - | - | - | - |
| | Male | xxx.x | xxx.x | x.xxx | XX.X | xx.x-xx.x |
| BMI Category | <30 (reference) | - | - | - | - | - |
| | ≥30 | XXX.X | xxx.x | x.xxx | xx.x | xx.x-xx.x |
| Prior Receipt of Influenza Vaccine | Did Not Receive 2016-2017 or 2017-<br>2018 Seasonal Influenza Vaccine<br>(reference) | - | - | - | - | - |
| | Received 2016-2017 or 2017-2018<br>Seasonal Influenza Vaccine | xxx.x | xxx.x | x.xxx | XX.X | xx.x-xx.x |

N = XX subjects with results available at 21 days post second vaccination in the per protocol population. XX subjects missing covariate data were excluded from this analysis. P-value for Treatment = 0.XXX; P-value for Age = 0.XXX; P-value for interaction of Treatment and Age = 0.XXX.

- Table 58: Logistic Regression Model to Evaluate the Relationship of HA Antigen Dose and AS03 Adjuvant with Neut Seroconversion Against 2017 A/H7N9 at 21 Days Post Second Study Vaccination, Adjusted for Baseline Covariates, Per Protocol Population\*
- Table 59: Logistic Regression Model to Evaluate the Relationship of HA Antigen Dose and AS03 Adjuvant with HAI Seroconversion Against 2017 A/H7N9 at 180 Days Post Second Study Vaccination, Adjusted for Baseline Covariates, Per Protocol Population\*
- Table 60: Logistic Regression Model to Evaluate the Relationship of HA Antigen Dose and AS03 Adjuvant with Neut Seroconversion Against 2017 A/H7N9 at 180 Days Post Second Study Vaccination, Adjusted for Baseline Covariates, Per Protocol Population\*

Table 61: Multiple Linear Regression Model to Evaluate the Relationship of HA Antigen Dose and AS03 Adjuvant with Log-Adjusted HAI Titer at 21 Days Post Second Study Vaccination, Per Protocol Population\*

| Model Parameter | Parameter Levels | Parameter<br>Estimate | SE | 95%CI | p-value |
|---|---|---|---|---|---|
| Intercept | | xxx.x | xxx.x | - | x.xxx |
| Treatment | 3.75 mcg with AS03 adjuvant (reference) | - | - | - | - |
| | 7.5 mcg with AS03 adjuvant | xxx.x | xxx.x | xx.x-xx.x | x.xxx |
| | 15 mcg with AS03 adjuvant | xxx.x | xxx.x | xx.x-xx.x | x.xxx |
| | 15 mcg without AS03 adjuvant | xxx.x | xxx.x | xx.x-xx.x | x.xxx |
| | 45 mcg without AS03 adjuvant | xxx.x | xxx.x | xx.x-xx.x | x.xxx |
| Age | 19-64 years (reference) | - | - | - | - |
| | ≥65 years | xxx.x | xxx.x | xx.x-xx.x | x.xxx |
| Interaction: Age*Treatment | Age*3.75 mcg with AS03 adjuvant | - | - | - | - |
| | Age*7.5 mcg with AS03 adjuvant | xxx.x | xxx.x | xx.x-xx.x | x.xxx |
| | Age*15 mcg with AS03 adjuvant | xxx.x | xxx.x | xx.x-xx.x | x.xxx |
| | Age*15 mcg without AS03 adjuvant | xxx.x | xxx.x | xx.x-xx.x | x.xxx |
| 7777 11 | Age*45 mcg without AS03 adjuvant | xxx.x | xxx.x | xx.x-xx.x | x.xxx |

N = XX subjects with results available at 21 days post second vaccination in the per protocol population. XX subjects missing covariate data were excluded from this analysis. P-value for Treatment = 0.XXX; P-value for Age = 0.XXX; P-value for interaction of Treatment and Age = 0.XXX.

- Table 62: Multiple Linear Regression Model to Evaluate the Relationship of HA Antigen Dose and AS03 Adjuvant with Log-Adjusted Neut Titer at 21 Days Post Second Study Vaccination, Per Protocol Population\*
- Table 63: Multiple Linear Regression Model to Evaluate the Relationship of HA Antigen Dose and AS03 Adjuvant with Log-Adjusted HAI Titer at 180 Days Post Second Study Vaccination, Per Protocol Population\*
- Table 64: Multiple Linear Regression Model to Evaluate the Relationship of HA Antigen Dose and AS03 Adjuvant with Log-Adjusted Neut Titer at 180 Days Post Second Study Vaccination, Per Protocol Population\*

Table 65: Multiple Linear Regression Model to Evaluate the Relationship of HA Antigen Dose and AS03 Adjuvant with Log-Adjusted HAI Titer at 21 Days Post Second Study Vaccination, Adjusted for Baseline Covariates, Per Protocol Population\*

| Model Parameter | Parameter Levels | Parameter<br>Estimate | SE | 95%CI | p-value |
|---|---|---|---|---|---|
| Intercept | - | XXX.X | xxx.x | - | x.xxx |
| Treatment | 3.75 mcg with AS03 adjuvant (reference) | - | - | - | - |
| | 7.5 mcg with AS03 adjuvant | xxx.x | xxx.x | XX.X-XX.X | x.xxx |
| | 15 mcg with AS03 adjuvant | xxx.x | xxx.x | xx.x-xx.x | x.xxx |
| | 15 mcg without AS03 adjuvant | xxx.x | xxx.x | XX.X-XX.X | x.xxx |
| | 45 mcg without AS03 adjuvant | xxx.x | xxx.x | XX.X-XX.X | x.xxx |
| Age | 19-64 (reference) | - | - | - | - |
| | ≥65 | xxx.x | xxx.x | XX.X-XX.X | x.xxx |
| Interaction: Age*Treatment | Age*3.75 mcg with AS03 adjuvant | - | - | - | - |
| | Age*7.5 mcg with AS03 adjuvant | xxx.x | xxx.x | XX.X-XX.X | x.xxx |
| | Age*15 mcg with AS03 adjuvant | xxx.x | xxx.x | XX.X-XX.X | x.xxx |
| | Age*15 mcg without AS03 adjuvant | xxx.x | xxx.x | XX.X-XX.X | x.xxx |
| | Age*45 mcg without AS03 adjuvant | XXX.X | XXX.X | XX.X-XX.X | x.xxx |
| Sex | Female (reference) | - | - | - | - |
| | Male | xxx.x | xxx.x | XX.X-XX.X | x.xxx |
| BMI Category | <30 (reference) | - | - | - | - |
| | ≥30 | xxx.x | xxx.x | XX.X-XX.X | x.xxx |
| Prior Receipt of Influenza Vaccine | Did Not Receive 2016-2017 or 2017-2018<br>Seasonal Influenza Vaccine (reference) | - | - | - | - |
| | Received 2016-2017 or 2017-2018 Seasonal Influenza Vaccine | xxx.x | xxx.x | xx.x-xx.x | x.xxx |

N = XX subjects with results available at 21 days post second vaccination in the per protocol population.. XX subjects missing covariate data were excluded from this analysis.

P-value for Treatment = 0.XXX; P-value for Age = 0.XXX; P-value for interaction of Treatment and Age = 0.XXX.

- Table 66: Multiple Linear Regression Model to Evaluate the Relationship of HA Antigen Dose and AS03 Adjuvant with Log-Adjusted Neut Titer at 21 Days Post Second Study Vaccination, Adjusted for Baseline Covariates, Per Protocol Population\*
- Table 67: Multiple Linear Regression Model to Evaluate the Relationship of HA Antigen Dose and AS03 Adjuvant with Log-Adjusted HAI Titer at 180 Days Post Second Study Vaccination, Adjusted for Baseline Covariates, Per Protocol Population\*
- Table 68: Multiple Linear Regression Model to Evaluate the Relationship of HA Antigen Dose and AS03 Adjuvant with Log-Adjusted Neut Titer at 180 Days Post Second Study Vaccination, Adjusted for Baseline Covariates, Per Protocol Population\*

Table 69: Logistic Regression Model to Evaluate the Relationship of HA Antigen Dose and AS03 Adjuvant with HAI Seroconversion Against 2017 A/H7N9 at 21 Days Post Second Study Vaccination, Adjusted for Baseline Covariates and Age in Years, Per Protocol Population\*

| Model Parameter | Parameter Levels | Parameter | | | Odds Ratio | |
|---|---|---|---|---|---|---|
| | | Estimate | SE | p-value | | 95%CI |
| Intercept | - | xxx.x | xxx.x | x.xxx | - | - |
| Treatment | 3.75 mcg with AS03 adjuvant (reference) | - | - | - | - | - |
| | 7.5 mcg with AS03 adjuvant | xxx.x | xxx.x | x.xxx | xx.x | XX.X-XX.X |
| | 15 mcg with AS03 adjuvant | XXX.X | xxx.x | xx.x-xx.x | x.xxx | |
| | 15 mcg without AS03 adjuvant | XXX.X | xxx.x | x.xxx | xx.x | XX.X-XX.X |
| 45 mcg without AS03 adjuvant | | xxx.x | xxx.x | x.xxx | XX.X | XX.X-XX.X |
| Age (years) | - | XXX.X | xxx.x | x.xxx | xx.x | XX.X-XX.X |
| Interaction: Age*Treatment | Age*3.75 mcg with AS03 adjuvant | - | - | - | - | - |
| | Age*7.5 mcg with AS03 adjuvant | XXX.X | xxx.x | x.xxx | xx.x | XX.X-XX.X |
| | Age*15 mcg with AS03 adjuvant | xxx.x | xxx.x | x.xxx | XX.X | XX.X-XX.X |
| | Age*15 mcg without AS03 adjuvant | XXX.X | xxx.x | xx.x-xx.x | x.xxx | |
| | Age*45 mcg without AS03 adjuvant | XXX.X | xxx.x | x.xxx | xx.x | XX.X-XX.X |
| Sex | Female (reference) | - | - | - | - | - |
| | Male | XXX.X | xxx.x | x.xxx | xx.x | XX.X-XX.X |
| BMI Category | <30 (reference) | - | - | - | - | - |
| | ≥30 | XXX.X | xxx.x | x.xxx | xx.x | XX.X-XX.X |
| Prior Receipt of Influenza Vaccine | Did Not Receive 2016-2017 or 2017-<br>2018 Seasonal Influenza Vaccine<br>(reference) | - | - | - | - | - |
| ex<br>MI Category | Received 2016-2017 or 2017-2018<br>Seasonal Influenza Vaccine | xxx.x | xxx.x | x.xxx | XX.X | xx.x-xx.x |

N = XX subjects with results available at 21 days post second vaccination in the per protocol population.. XX subjects missing covariate data were excluded from this analysis. P-value for Treatment = 0.XXX; P-value for Age = 0.XXX; P-value for interaction of Treatment and Age = 0.XXX.

Table 70: Multiple Linear Regression Model to Evaluate the Relationship of HA Antigen Dose and AS03 Adjuvant with Log-Adjusted HAI Titer at 21 Days Post Second Study Vaccination, Adjusted for Baseline Covariates and Age in Years, Per Protocol Population\*

| Model Parameter | Parameter Levels | | | | |
|---|---|---|---|---|---|
| | | Parameter Estimate | SE | 95%CI | p-value |
| Intercept | - | xxx.x | xxx.x | - | x.xxx |
| Treatment | 3.75 mcg with AS03 Adjuvant (reference) | - | - | - | - |
| | 7.5 mcg with AS03 Adjuvant | xxx.x | XXX.X | xx.x-xx.x | x.xxx |
| | 15 mcg with AS03 Adjuvant | xxx.x | XXX.X | xx.x-xx.x | x.xxx |
| | 15 mcg without AS03 Adjuvant | xxx.x | XXX.X | xx.x-xx.x | x.xxx |
| | 45 mcg without AS03 Adjuvant | xxx.x | XXX.X | xx.x-xx.x | x.xxx |
| Age (years) | - | xxx.x | XXX.X | xx.x-xx.x | x.xxx |
| Interaction: Age*Treatment | Age*3.75 mcg with AS03 Adjuvant | - | - | - | - |
| | Age*7.5 mcg with AS03 Adjuvant | xxx.x | XXX.X | xx.x-xx.x | x.xxx |
| | Age*15 mcg with AS03 Adjuvant | xxx.x | XXX.X | xx.x-xx.x | x.xxx |
| | Age*15 mcg without AS03 Adjuvant | xxx.x | XXX.X | xx.x-xx.x | x.xxx |
| | Age*45 mcg without AS03 Adjuvant | xxx.x | XXX.X | XX.X-XX.X | x.xxx |
| Sex | Female (reference) | - | - | - | - |
| | Male | xxx.x | XXX.X | xx.x-xx.x | x.xxx |
| BMI Category | <30 (reference) | - | - | - | - |
| | ≥30 | xxx.x | XXX.X | XX.X-XX.X | x.xxx |
| Prior Receipt of Influenza<br>Vaccine | Did Not Receive 2016-2017 or 2017-2018<br>Seasonal Influenza Vaccine (reference) | - | - | - | - |
| | Received 2016-2017 or 2017-2018 Seasonal Influenza Vaccine | xxx.x | XXX.X | xx.x-xx.x | x.xxx |

N = XX subjects with results available at 21 days post second vaccination in the per protocol population. XX subjects missing covariate data were excluded from this analysis.

P-value for Treatment = 0.XXX; P-value for Age = 0.XXX; P-value for interaction of Treatment and Age = 0.XXX.

Table 71: Summaries of Hemagglutination Inhibition Antibody Against Antigenically Drifted Variants by Study Day, Treatment Arm and Age Stratum, Per Protocol Population\*

| | 3.75 mcg<br>+ A | up 1<br>; A/H7N9<br>S03<br>=X) | + <b>A</b> | up 2<br>A/H7N9<br>S03<br>=X) | 15 mcg + A | up 3<br>A/H7N9<br>S03<br>=X) | Group 4<br>15 mcg A/H7N9<br>(N=X) | | 45 mcg | up 5<br>A/H7N9<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | 19-64 | ≥ 65 | 19-64 | ≥ 65 | 19-64 | ≥ 65 | 19-64 | ≥ 65 | 19-64 | ≥ 65 |
| Strain = [Antigenically Drifted | d Variant] | | | | | | | | | |
| Day 1 (Pre Vaccination 1) | | | | | | | | | | |
| n | X | Х | X | X | Х | X | x | х | X | X |
| GMT (95% CI) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) |
| Titer ≥ 1:40 - %(95% CI) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| Day 21 Post Vaccination 2 | | | | | | | | | | |
| n | Х | Х | Х | Х | Х | X | х | х | X | X |
| GMT (95% CI) <sup>a</sup> | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) |
| Titer $\ge 1:40 - \% (95\% \text{ CI})^b$ | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| GMFR (95% CI) <sup>a</sup> | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) |
| Seroconversion - % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| Day 180 Post Vaccination 2 | | | | | | | | | | |
| n | X | X | X | X | X | X | X | X | X | X |
| GMT (95% CI) <sup>a</sup> | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) |
| Titer ≥ 1:40 - % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| GMFR (95% CI) <sup>a</sup> | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) | xxx.x<br>(xxx.x,xxx.x) |
| Seroconversion - % (95% CI) <sup>b</sup> | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| [repeat for each antigenica | ally drifted v | ariant of the | A/H7 virus] | | | | | | | |

Table 71: Summaries of Hemagglutination Inhibition Antibody Against Antigenically Drifted Variants by Study Day, Treatment Arm and Age Stratum, Per Protocol Population (continued)

| | 3.75 mcg<br>+ A | up 1<br>3 A/H7N9<br>S03<br>=X) | 7.5 mcg<br>+ A | oup 2<br>A/H7N9<br>.S03<br>=X) | 15 mcg<br>+ A | up 3<br>A/H7N9<br>.S03<br>=X) | 15 mcg | up 4<br>A/H7N9<br>=X) | 45 mcg | up 5<br>A/H7N9<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | 19-64 | 19-64 ≥ 65 | | ≥ 65 | 19-64 | ≥ 65 | 19-64 | ≥ 65 | 19-64 | ≥ 65 |

Table 72: Summaries of Neutralizing Antibody Against Antigenically Drifted Variants by Study Day, Treatment Arm and Age Stratum, Per Protocol Population\*

<sup>&</sup>lt;sup>a</sup> Confidence Interval calculated based on the student's T distribution.

<sup>&</sup>lt;sup>b</sup> Exact binomial confidence interval calculated using the Clopper-Pearson methodology.

## 14.3 Safety Data

# 14.3.1 Displays of Adverse Events

Table 73: Overall Summary of Adverse Events - Safety Population\*‡

| | 3.7<br>A/<br>+ | roup 1<br>75 mcg<br>H7N9<br>AS03<br>N=X) | 7.:<br>A/<br>+ | roup 2<br>5 mcg<br>H7N9<br>AS03<br>N=X) | 15<br>A/F<br>+ A | oup 3<br>mcg<br>H7N9<br>AS03<br>=X) | 15<br>A/H | oup 4<br>mcg<br>H7N9<br>(=X) | Group 5<br>45 mcg<br>A/H7N9<br>(N=X) | | All Subjects<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subjects <sup>a</sup> with | n | % | n | % | n | % | n | % | n | % | n | % |
| At least one local solicited adverse event | X | X | x | X | X | x | x | X | x | X | X | X |
| At least one systemic solicited adverse event | Х | х | х | Х | х | х | х | x | x | x | X | X |
| At least one unsolicited adverse event | X | X | Х | X | X | X | X | X | X | X | X | X |
| At least one related unsolicited adverse event | X | X | x | X | X | x | x | x | X | x | X | X |
| Mild (Grade 1) | X | X | X | X | X | Х | Х | X | X | Х | Х | X |
| Moderate (Grade 2) | X | X | Х | X | X | Х | Х | X | X | X | X | X |
| Severe (Grade 3) | X | X | Х | X | X | Х | Х | X | X | X | Х | X |
| Not yet assessed | | | | | | | | | | | | |
| At least one severe (Grade 3) unsolicited adverse event | X | X | x | X | X | x | x | X | X | X | X | X |
| Related | X | X | Х | X | X | Х | Х | X | X | X | X | X |
| Unrelated | X | x | Х | X | X | X | X | X | X | X | Х | X |
| Not yet assessed | | | | | | | | | | | | |
| At least one serious adverse event <sup>b</sup> | X | X | х | X | X | X | X | X | X | X | Х | X |
| At least one related, serious adverse event | X | X | Х | X | X | Х | Х | X | X | Х | Х | X |

Table 73: Overall Summary of Adverse Events – Safety Population \* (continued)

| | 3.7.<br>A/I<br>+ . | oup 1<br>5 mcg<br>H7N9<br>AS03<br>N=X) | 7.5<br>A/I<br>+ A | oup 2<br>5 mcg<br>H7N9<br>AS03<br>I=X) | Group 3<br>15 mcg<br>A/H7N9<br>+ AS03<br>(N=X) | | Group 4<br>15 mcg<br>A/H7N9<br>(N=X) | | Group 5<br>45 mcg<br>A/H7N9<br>(N=X) | | All Subjects<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subjects <sup>a</sup> with | n | % | n | % | n | % | n | % | n | % | n | % |
| At least one adverse event leading to early termination <sup>c</sup> | X | Х | X | X | Х | X | X | X | Х | X | X | Х |
| At least one medically attended adverse event | X | X | x | X | Х | X | X | x | Х | X | X | X |
| At least one new onset chronic medical condition | X | X | X | X | X | X | X | X | X | X | X | x |
| At least one potentially immune mediated medical condition | X | X | X | X | X | X | X | X | X | X | X | X |

N = Number of subjects who received at least one study vaccination

<sup>a</sup> Subjects are counted once for each category regardless of the number of events.

<sup>b</sup> A listing of Serious Adverse Events is included in Table 99

<sup>&</sup>lt;sup>c</sup> As reported on the Adverse Event eCRF

Table 74: Number of Adverse Events Occurring in 5% of Subjects in Any Treatment Group by MedDRA System Organ Class and Preferred Term, and Treatment Group - Safety Population

| Preferred Term | MedDRA System<br>Organ Class | Group 1<br>3.75 mcg A/H7N9<br>+ AS03<br>(N=X) | | | Group 2<br>7.5 mcg A/H7N9<br>+ AS03<br>(N=X) | | | Group 3<br>15 mcg A/H7N9<br>+ AS03<br>(N=X) | | | Group 4<br>15 mcg A/H7N9<br>(N=X) | | | Group 5<br>45 mcg A/H7N9<br>(N=X) | | | All Subjects<br>(N=X) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | Events | n | % | Events | n | % | Events | n | % | Events | n | % | Events | n | % | Events |
| erious Adverse Events | | | | | | | | | | | | | | | | | | | |
| All | All | X | X | X | X | X | X | X | х | X | Х | х | x | X | X | X | X | х | X |
| PT1 | SOC1 | X | X | X | X | X | X | X | х | X | Х | х | x | X | X | X | X | х | X |
| Etc. | Etc. | | | | | | | | | | | | | | | | | | |
| Other (Non-serious) Adverse l | Events | | | | | | | | | | | | | | | | | | |
| All | All | X | X | X | X | X | X | X | Х | X | X | х | X | X | X | X | X | X | X |
| PT1 | SOC1 | X | X | X | X | X | X | X | х | X | X | х | х | X | X | X | X | X | X |
| Etc. | Etc. | | | | | | | | | | | | | | | | | | |

N = number of subjects in the safety population (number of subjects at risk). n= number of subjects reporting event. Events = total frequency of events reported. MedDRA Version X.X.

The preferred term "Pain injection site" identifies both injection site tenderness and injection site pain. To distinguish between the two events, the preferred term "Pain injection site (tenderness)" was used to identify injection site tenderness.

### 14.3.1.1 Solicited Adverse Events

Table 75: Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom and Treatment Arm Post Any Study Vaccination – Safety Population\*

| Symptom | Group 1<br>3.75 mcg A/H7N9<br>+ AS03<br>(N=X) | | | Group 2<br>7.5 mcg A/H7N9<br>+ AS03<br>(N=X) | | | 15 n | Group 3<br>neg A/H7<br>+ AS03<br>(N=X) | 7N9 | 15 | Group 4<br>mcg A/H<br>(N=X) | | Group 5<br>45 mcg A/H7N9<br>(N=X) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI |
| Any Symptom | х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Any Systemic Symptom | х | XX | xx-xx | X | xx | xx-xx | X | xx | xx-xx | Х | XX | xx-xx | X | XX | xx-xx |
| Fever | х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Feverishness | х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Fatigue | х | XX | xx-xx | x | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | x | XX | xx-xx |
| Malaise | х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Myalgia | х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Arthralgia | х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Headache | х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Nausea | х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Any Local Symptom | х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Pain | х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Tenderness | х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Pruritus | х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Ecchymosis | х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Ecchymosis (measurement) | Х | XX | xx-xx | X | xx | xx-xx | X | xx | xx-xx | Х | XX | xx-xx | X | XX | xx-xx |
| Erythema | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Erythema (measurement) | Х | XX | xx-xx | X | xx | xx-xx | X | xx | xx-xx | Х | XX | xx-xx | X | XX | xx-xx |
| Induration/Swelling | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |

Table 75: Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom and Treatment Arm– Post Any Study Vaccination – Safety Population (continued)

| Induration/Swelling (measurement) | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| N N 1 C 1' 4' 4 C C 4 D 14' 1 ' 1 4 1 ' 4' | | | | | | | | | | | | | | | |

N = Number of subjects in the Safety Population who received any study vaccination.

95% CI estimated using Clopper-Pearson exact method

Tables with similar format:

Table 76: Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom and Treatment Arm Post Study Vaccination 1 – Safety Population \*

[Footnote update] N = Number of subjects in the Safety Population who received the first vaccination.

Table 77: Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom and Treatment Arm Post Study Vaccination 2 – Safety Population \*

[Footnote update] N = Number of subjects in the Safety Population who received the second vaccination.
Table 78: Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom, Treatment Arm and Age Stratum Post Any Study Vaccination – Safety Population \*

| | 3.75 | Group 1<br>5 mcg A/F<br>+ AS03<br>(N=X) | | 7.5 | Group 2<br>mcg A/H<br>+ AS03<br>(N=X) | | 15 | Group 3<br>mcg A/H'<br>+ AS03<br>(N=X) | | 15 | Group 4<br>mcg A/H<br>(N=X) | | 45 | Group 5<br>mcg A/H<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI |
| | l | | | | | Age 19 | <b>)</b> -64 | l | | | l | | | | <u>.I</u> |
| Any Symptom | х | XX | xx-xx | X | xx | xx-xx | X | xx | xx-xx | X | xx | xx-xx | X | xx | xx-xx |
| Any Systemic Symptom | х | XX | xx-xx | X | xx | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Fever | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Feverishness | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Fatigue | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Malaise | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Myalgia | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Arthralgia | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Headache | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Nausea | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Any Local Symptom | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Pain | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Tenderness | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Pruritus | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Ecchymosis | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Ecchymosis (measurement) | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Erythema | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Erythema (measurement) | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Induration/Swelling | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |

Table 78: Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom, Treatment Arm and Age Stratum – Post Any Study Vaccination – Safety Population (continued)

| | 3.75 | Group 1<br>5 mcg A/F<br>+ AS03<br>(N=X) | | 7.5 | Group 2<br>mcg A/H<br>+ AS03<br>(N=X) | | 15 | Group 3<br>mcg A/H'<br>+ AS03<br>(N=X) | | 15 | Group 4<br>mcg A/H<br>(N=X) | | 45 | Group 5<br>mcg A/H<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI |
| Induration/Swelling (measurement) | х | XX | xx-xx | X | xx | xx-xx | X | xx | xx-xx | X | xx | xx-xx | X | xx | xx-xx |
| | • | | • | | • | Age 6 | 5+ | • | • | | | • | | • | • |
| Any Symptom | х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Any Systemic Symptom | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Fever | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Feverishness | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Fatigue | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Malaise | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Myalgia | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Arthralgia | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Headache | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Nausea | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Any Local Symptom | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Pain | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Tenderness | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Pruritus | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Ecchymosis | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Ecchymosis (measurement) | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Erythema | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Erythema (measurement) | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Induration/Swelling | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |

Table 78: Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom, Treatment Arm and Age Stratum - Post Any Study Vaccination - Safety Population (continued)

| | 3.75 | Group 1<br>mcg A/H<br>+ AS03<br>(N=X) | 7.5 | Group 2<br>mcg A/H'<br>+ AS03<br>(N=X) | | 15 1 | Group 3<br>mcg A/H7<br>+ AS03<br>(N=X) | | 15 | Group 4<br>mcg A/H?<br>(N=X) | 7N9 | 45 1 | Group 5<br>mcg A/H′<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | n | 95% | | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI |
| Induration/Swelling (measurement) | х | v vv vv | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |

N = Number of subjects in the Safety Population who received any study vaccination. 95% CI estimated using Clopper-Pearson exact method

Table 79: Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom, Treatment Arm and Age Stratum Post Study Vaccination 1 – Safety Population \*

[Footnote update] N = Number of subjects in the Safety Population who received the first vaccination.

Table 80: Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom, Treatment Arm and Age Stratum Post Study Vaccination 2 – Safety Population \*

[Footnote update] N = Number of subjects in the Safety Population who received the second vaccination.

Table 81: Logistic Regression Model to Evaluate the Relationship of HA Antigen Dose, AS03 Adjuvant, and Age with Reporting Any Local Event Post Any Study Vaccination – Safety Population \*

| Model Parameter | Parameter Levels | Parameter<br>Estimate | SE | p-value | Odds Ratio | 95%CI |
|---|---|---|---|---|---|---|
| Intercept | - | xxx.x | xxx.x | x.xxx | - | - |
| Freatment | 3.75 mcg with AS03 adjuvant (reference) | - | - | - | - | - |
| | 7.5 mcg with AS03 adjuvant | xxx.x | xxx.x | x.xxx | xx.x | xx.x-xx.x |
| | 15 mcg with AS03 adjuvant | XXX.X | xxx.x | x.xxx | XX.X | XX.X-XX.X |
| | 15 mcg without AS03 adjuvant | XXX.X | xxx.x | x.xxx | xx.x | XX.X-XX.X |
| | 45 mcg without AS03 adjuvant | xxx.x | xxx.x | x.xxx | xx.x | xx.x-xx.x |
| Age | 19-64 years (reference) | - | - | - | - | - |
| | ≥65 years | XXX.X | xxx.x | x.xxx | xx.x | XX.X-XX.X |
| Interaction (Age * Treatment) | ≥65 years * 7.5 mcg with AS03 adjuvant | XXX.X | XXX.X | x.xxx | XX.X | xx.x-xx.x |
| | ≥65 years * 15 mcg with AS03 adjuvant | XXX.X | xxx.x | x.xxx | XX.X | XX.X-XX.X |
| | ≥65 years * 15 mcg without AS03 adjuvant | XXX.X | xxx.x | x.xxx | XX.X | XX.X-XX.X |
| | ≥65 years * 45 mcg without AS03 adjuvant | XXX.X | XXX.X | x.xxx | XX.X | xx.x-xx.x |

N = XX subjects in the safety population.

P-value for Treatment = 0.XXX; P-value for Age = 0.XXX; P-value for interaction of Treatment and Age = 0.XXX.

Table with similar format:

Table 82: Logistic Regression Model to Evaluate the Relationship of HA Antigen Dose, AS03 Adjuvant, and Age with Reporting Any Systemic Event Post Any Study Vaccination (N=X) – Safety Population \*

Table 83: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity and Treatment Arm Post Any Study Vaccination – Safety Population \*

| | | 3.75 | Group 1<br>mcg A/I<br>+ AS03<br>(N=X) | H7N9 | | Group 2<br>mcg A/H<br>+ AS03<br>(N=X) | | | Group 3<br>mcg A/H<br>+ AS03<br>(N=X) | 7N9 | | Group 4<br>mcg A/H<br>(N=X) | | | Group :<br>mcg A/H<br>(N=X) | 17N9 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | 95% CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI |
| Any Symptom | None | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | х | XX | xx-xx | X | XX | xx-xx |
| | Mild | х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Moderate | х | xx | xx-xx | X | XX | xx-xx | X | xx | xx-xx | Х | xx | xx-xx | Х | XX | xx-xx |
| | Severe | х | xx | xx-xx | X | XX | xx-xx | X | xx | xx-xx | Х | xx | xx-xx | Х | XX | xx-xx |
| Any Systemic<br>Symptom | None | Х | xx | xx-xx | Х | xx | xx-xx | X | xx | xx-xx | х | XX | XX-XX | Х | XX | xx-xx |
| | Mild | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Severe | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Fever | None | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Mild | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Severe | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Feverishness | None | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Mild | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Severe | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Fatigue | None | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Mild | X | XX | xx-xx | X | XX | xx-xx | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Severe | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Malaise | None | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |

Table 83: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity and Treatment Arm – Post Any Study Vaccination – Safety Population (continued)

| | | 3.75 | Group 1<br>mcg A/I<br>+ AS03<br>(N=X) | H7N9 | | Group 2<br>mcg A/H<br>+ AS03<br>(N=X) | 17N9 | 15 1 | Group 3<br>mcg A/H<br>+ AS03<br>(N=X) | 7N9 | | Group 4<br>mcg A/H<br>(N=X) | | | Group :<br>mcg A/H<br>(N=X) | I7N9 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | 95% CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI |
| | Mild | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | Х | XX | xx-xx |
| | Moderate | х | XX | xx-xx | X | XX | xx-xx | Х | XX | xx-xx | X | XX | xx-xx | х | XX | xx-xx |
| | Severe | X | xx | xx-xx | X | XX | xx-xx | Х | XX | xx-xx | Х | xx | xx-xx | х | XX | xx-xx |
| Myalgia | None | х | xx | xx-xx | X | XX | xx-xx | X | xx | xx-xx | X | XX | xx-xx | х | XX | xx-xx |
| | Mild | х | xx | xx-xx | X | XX | xx-xx | X | xx | xx-xx | X | XX | xx-xx | х | XX | xx-xx |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Severe | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Arthralgia | None | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Mild | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Severe | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Headache | None | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Mild | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Severe | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Nausea | None | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Mild | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Moderate | X | XX | XX-XX | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Severe | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Any Local Symptom | None | Х | XX | XX-XX | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Mild | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Moderate | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | Х | XX | xx-xx |

Table 83: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity and Treatment Arm – Post Any Study Vaccination – Safety Population (continued)

| | | 3.75 | Group<br>mcg A/2<br>+ AS03<br>(N=X) | H7N9 | | Group 2<br>mcg A/H<br>+ AS03<br>(N=X) | 17N9 | | Group 3<br>mcg A/H<br>+ AS03<br>(N=X) | 17N9 | | Group 4<br>mcg A/H<br>(N=X) | | 45 1 | Group :<br>ncg A/H<br>(N=X) | 17N9 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | 95% CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI |
| | Severe | Х | xx | xx-xx | X | xx | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Pain | None | х | xx | xx-xx | X | xx | xx-xx | Х | XX | xx-xx | Х | xx | xx-xx | X | XX | xx-xx |
| | Mild | х | xx | xx-xx | X | xx | xx-xx | X | XX | xx-xx | X | xx | xx-xx | X | XX | xx-xx |
| | Moderate | Х | xx | xx-xx | X | xx | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Severe | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Tenderness | None | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Mild | X | xx | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Severe | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Pruritus | None | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Mild | X | XX | xx-xx | X | xx | xx-xx | X | xx | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Severe | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Ecchymosis | None | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Mild | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Severe | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Ecchymosis (measurement) | None | х | XX | xx-xx | х | XX | xx-xx | х | XX | xx-xx | х | XX | xx-xx | X | XX | xx-xx |
| | Mild | X | XX | xx-xx | X | xx | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | X | xx | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| _ | Severe | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |

Table 83: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity and Treatment Arm – Post Any Study Vaccination – Safety Population (continued)

| | | 3.75 | Group :<br>5 mcg A/I<br>+ AS03<br>(N=X) | H7N9<br>3 | | Group 2<br>mcg A/H<br>+ AS03<br>(N=X) | 17N9 | 15 | Group 3<br>mcg A/H<br>+ AS03<br>(N=X) | 7N9 | | Group 4<br>mcg A/H<br>(N=X) | | 45 1 | Group :<br>mcg A/H<br>(N=X) | 17N9 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | 95% CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI |
| Erythema | None | х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | х | XX | xx-xx | X | XX | xx-xx |
| | Mild | х | xx | xx-xx | Х | XX | xx-xx | Х | XX | xx-xx | х | xx | xx-xx | Х | XX | xx-xx |
| | Moderate | х | xx | xx-xx | X | xx | xx-xx | X | XX | xx-xx | х | xx | xx-xx | X | XX | xx-xx |
| | Severe | х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | х | XX | xx-xx | X | XX | xx-xx |
| Erythema (measurement) | None | х | XX | xx-xx | X | xx | xx-xx | х | XX | xx-xx | Х | XX | XX-XX | Х | XX | XX-XX |
| | Mild | х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | х | XX | xx-xx | X | XX | xx-xx |
| | Moderate | х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | х | XX | xx-xx | X | XX | xx-xx |
| | Severe | х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | х | XX | xx-xx | X | XX | xx-xx |
| Induration/Swelling | None | х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | х | XX | xx-xx | X | XX | xx-xx |
| | Mild | х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | х | XX | xx-xx | X | XX | xx-xx |
| | Moderate | Х | xx | xx-xx | X | XX | xx-xx | х | xx | xx-xx | х | XX | xx-xx | х | XX | xx-xx |
| | Severe | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | х | XX | xx-xx | X | XX | xx-xx |
| Induration/Swelling (measurement) | None | Х | XX | XX-XX | X | XX | xx-xx | X | XX | xx-xx | Х | XX | xx-xx | X | XX | xx-xx |
| | Mild | х | xx | xx-xx | X | XX | xx-xx | X | xx | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Moderate | х | xx | xx-xx | X | XX | xx-xx | X | xx | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Severe | Х | xx | xx-xx | X | XX | xx-xx | х | xx | xx-xx | х | XX | xx-xx | х | XX | xx-xx |

N = Number of subjects in the Safety Population who received any study vaccination.

Severity is the maximum severity reported over all solicited symptoms post dosing for each subject.

<sup>95%</sup> CI estimated using Clopper-Pearson exact method

Table 84: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity and Treatment Arm Post Study Vaccination 1 – Safety Population \*

[Footnote Update] N = Number of subjects in the Safety Analysis Population who received the first study vaccination.

Table 85: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity and Treatment Arm Post Study Vaccination 2 – Safety Population \*

[Footnote Update] N = Number of subjects in the Safety Analysis Population who received the second study vaccination.

Table 86: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, Treatment Arm and Age Stratum Post Any Study Vaccination – Safety Population \*

| | | 3.75 | Group<br>5 mcg A/2<br>+ AS03<br>(N=X) | H7N9<br>3 | 7.5 | Group 2<br>mcg A/H<br>+ AS03<br>(N=X) | | 15 | Group 3<br>mcg A/H<br>+ AS03<br>(N=X) | | 15 | Group 4<br>mcg A/H'<br>(N=X) | | 45 | Group 5<br>mcg A/H<br>(N=X) | ;<br>7N9 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | 95% CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI |
| | | | | | | | Age 19 | -64 | | | | | | | | • |
| Any Symptom | None | X | XX | xx-xx | X | XX | xx-xx | X | xx | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Mild | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | XX-XX |
| | Severe | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Any Systemic<br>Symptom | None | X | XX | xx-xx | X | XX | xx-xx | X | xx | xx-xx | X | XX | xx-xx | Х | XX | XX-XX |
| | Mild | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | х | XX | xx-xx |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Severe | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Fever | None | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Mild | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Severe | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Feverishness | None | x | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Mild | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Severe | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Fatigue | None | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | х | XX | xx-xx |
| | Mild | Х | XX | xx-xx | Х | XX | xx-xx | X | XX | xx-xx | Х | XX | xx-xx | X | XX | xx-xx |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |

Table 86: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, Treatment Arm and Age Stratum – Post Any Study Vaccination – Safety Population (continued)

| | | 3.7 | Group<br>5 mcg A/<br>+ AS03<br>(N=X) | H7N9<br>3 | 7.5 | Group 2<br>mcg A/H<br>+ AS03<br>(N=X) | 17N9 | 15 | Group 3<br>mcg A/H<br>+ AS03<br>(N=X) | | 15 | Group 4<br>mcg A/H<br>(N=X) | 7N9 | 45 | Group 5<br>mcg A/H<br>(N=X) | 7N9 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | 95% CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI |
| | Severe | X | XX | xx-xx | X | XX | xx-xx | Х | XX | xx-xx | Х | XX | xx-xx | Х | XX | xx-xx |
| Malaise | None | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | Х | XX | xx-xx | Х | XX | xx-xx |
| | Mild | Х | xx | xx-xx | X | XX | xx-xx | Х | XX | xx-xx | X | XX | xx-xx | х | XX | xx-xx |
| | Moderate | X | xx | xx-xx | X | XX | xx-xx | х | XX | xx-xx | X | XX | xx-xx | Х | XX | xx-xx |
| | Severe | X | xx | xx-xx | X | XX | xx-xx | х | XX | xx-xx | X | XX | xx-xx | Х | XX | xx-xx |
| Myalgia | None | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | Х | XX | xx-xx |
| | Mild | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | Х | XX | xx-xx |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | Х | XX | xx-xx |
| | Severe | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | Х | XX | xx-xx |
| Arthralgia | None | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | Х | XX | xx-xx |
| | Mild | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | Х | XX | xx-xx |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | Х | XX | xx-xx |
| | Severe | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Headache | None | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Mild | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Severe | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Nausea | None | X | xx | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | х | XX | xx-xx |
| | Mild | X | xx | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | х | XX | xx-xx |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | х | XX | xx-xx |
| | Severe | X | XX | xx-xx | Х | XX | xx-xx | X | xx | xx-xx | X | XX | xx-xx | Х | XX | xx-xx |

Table 86: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, Treatment Arm and Age Stratum – Post Any Study Vaccination – Safety Population (continued)

| | | 3.75 | Group<br>5 mcg A/2<br>+ AS03<br>(N=X) | H7N9<br>3 | 7.5 | Group 2<br>mcg A/H<br>+ AS03<br>(N=X) | | 15 | Group 3<br>mcg A/H'<br>+ AS03<br>(N=X) | | 15 | Group 4<br>mcg A/H<br>(N=X) | 7N9 | 45 | Group 5<br>mcg A/H<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | 95% CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI |
| Any Local<br>Symptom | None | Х | XX | xx-xx | X | xx | xx-xx | X | XX | xx-xx | Х | xx | xx-xx | X | xx | XX-XX |
| | Mild | X | XX | xx-xx | X | XX | xx-xx | Х | XX | xx-xx | х | XX | xx-xx | X | XX | xx-xx |
| | Moderate | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | Х | XX | xx-xx | X | XX | xx-xx |
| | Severe | X | XX | xx-xx | X | XX | xx-xx | Х | XX | xx-xx | Х | XX | xx-xx | X | XX | xx-xx |
| Pain | None | X | XX | xx-xx | X | XX | xx-xx | Х | XX | xx-xx | Х | XX | xx-xx | X | XX | xx-xx |
| | Mild | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Moderate | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Severe | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Tenderness | None | Х | XX | xx-xx | X | XX | xx-xx | х | XX | xx-xx | х | XX | xx-xx | Х | xx | xx-xx |
| | Mild | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Severe | X | XX | xx-xx | X | XX | xx-xx | Х | XX | xx-xx | х | XX | xx-xx | X | XX | xx-xx |
| Pruritus | None | X | XX | xx-xx | X | XX | xx-xx | Х | XX | xx-xx | Х | XX | xx-xx | X | XX | xx-xx |
| | Mild | X | XX | xx-xx | X | XX | xx-xx | Х | XX | xx-xx | Х | XX | xx-xx | X | XX | xx-xx |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | Х | XX | xx-xx | Х | XX | xx-xx | X | XX | xx-xx |
| | Severe | Х | XX | xx-xx | X | XX | xx-xx | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Ecchymosis | None | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | Х | XX | xx-xx | X | XX | xx-xx |
| | Mild | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | Х | XX | xx-xx | X | XX | xx-xx |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | Х | XX | xx-xx | X | XX | xx-xx |
| | Severe | X | XX | xx-xx | X | XX | xx-xx | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |

Table 86: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, Treatment Arm and Age Stratum – Post Any Study Vaccination – Safety Population (continued)

| | | 3.75 | Group<br>5 mcg A/<br>+ AS03<br>(N=X) | H7N9<br>3 | 7.5 | Group 2<br>mcg A/H<br>+ AS03<br>(N=X) | 17N9 | 15 | Group 3<br>mcg A/H<br>+ AS03<br>(N=X) | | 15 | Group 4<br>mcg A/H<br>(N=X) | | 45 | Group 5<br>mcg A/H<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | 95% CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI |
| Ecchymosis (measurement) | None | Х | xx | xx-xx | X | XX | XX-XX | X | xx | XX-XX | X | xx | XX-XX | X | xx | XX-XX |
| | Mild | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Moderate | X | xx | xx-xx | X | XX | xx-xx | Х | XX | xx-xx | Х | XX | xx-xx | Х | XX | xx-xx |
| | Severe | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Erythema | None | X | xx | xx-xx | X | XX | xx-xx | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Mild | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Moderate | X | xx | xx-xx | X | XX | xx-xx | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Severe | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Erythema (measurement) | None | Х | xx | xx-xx | Х | xx | xx-xx | X | xx | XX-XX | X | xx | XX-XX | X | xx | xx-xx |
| | Mild | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | XX-XX |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | XX-XX |
| | Severe | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | XX-XX |
| Induration/Swelling | None | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | XX-XX |
| | Mild | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | XX-XX |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Severe | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | XX-XX |
| Induration/Swelling (measurement) | None | X | xx | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | XX-XX |
| | Mild | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | XX-XX |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | XX-XX |

Table 86: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, Treatment Arm and Age Stratum – Post Any Study Vaccination – Safety Population (continued)

| | | 3.75 | Group<br>5 mcg A/<br>+ AS03<br>(N=X) | H7N9<br>3 | 7.5 | Group 2<br>mcg A/H<br>+ AS03<br>(N=X) | | | Group 3<br>mcg A/H'<br>+ AS03<br>(N=X) | | 15 | Group 4<br>mcg A/H<br>(N=X) | | 45 | Group 5<br>mcg A/H<br>(N=X) | ;<br>7N9 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | 95% CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI |
| | Severe | Х | XX | xx-xx | Х | XX | xx-xx | Х | XX | xx-xx | X | XX | xx-xx | Х | XX | xx-xx |
| | | | | | | • | Age 65 | <u>;</u> + | • | • | | • | • | | • | |
| Any Symptom | None | X | xx | xx-xx | x | xx | xx-xx | X | XX | xx-xx | X | xx | xx-xx | X | xx | xx-xx |
| | Mild | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Severe | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Any Systemic<br>Symptom | None | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | xx | XX-XX | X | xx | xx-xx |
| | Mild | X | xx | xx-xx | X | XX | xx-xx | X | XX | xx-xx | х | XX | xx-xx | X | XX | xx-xx |
| | Moderate | X | xx | xx-xx | x | xx | xx-xx | X | XX | XX-XX | х | XX | xx-xx | X | xx | xx-xx |
| | Severe | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Fever | None | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Mild | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Severe | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Feverishness | None | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Mild | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Severe | Х | XX | xx-xx | Х | XX | xx-xx | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Fatigue | None | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Mild | х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | Х | XX | xx-xx | X | XX | XX-XX |

Table 86: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, Treatment Arm and Age Stratum – Post Any Study Vaccination – Safety Population (continued)

| | | 3.75 | Group<br>5 mcg A/2<br>+ AS03<br>(N=X) | H7N9 | 7.5 | Group 2<br>mcg A/H<br>+ AS03<br>(N=X) | | 15 | Group 3<br>mcg A/H<br>+ AS03<br>(N=X) | | 15 | Group 4<br>mcg A/H<br>(N=X) | | 45 | Group 5<br>mcg A/H<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | 95% CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI |
| | Moderate | X | XX | xx-xx | x | XX | xx-xx | Х | XX | xx-xx | Х | XX | xx-xx | Х | XX | xx-xx |
| | Severe | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | х | XX | xx-xx | х | XX | xx-xx |
| Malaise | None | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Mild | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Severe | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Myalgia | None | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Mild | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Severe | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Arthralgia | None | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Mild | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Severe | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Headache | None | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Mild | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Severe | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Nausea | None | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Mild | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |

Table 86: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, Treatment Arm and Age Stratum – Post Any Study Vaccination – Safety Population (continued)

| | | 3.75 | Group<br>5 mcg A/<br>+ AS03<br>(N=X) | H7N9<br>3 | 7.5 | Group 2<br>mcg A/H<br>+ AS03<br>(N=X) | | 15 | Group 3<br>mcg A/H'<br>+ AS03<br>(N=X) | | 15 | Group 4<br>mcg A/H<br>(N=X) | | 45 | Group 5<br>mcg A/H<br>(N=X) | ;<br>7N9 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | 95% CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI |
| | Severe | X | xx | xx-xx | X | XX | xx-xx | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Any Local<br>Symptom | None | X | XX | xx-xx | X | xx | XX-XX | Х | xx | xx-xx | Х | xx | xx-xx | Х | XX | xx-xx |
| | Mild | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Severe | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | XX-XX |
| Pain | None | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Mild | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Severe | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Tenderness | None | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Mild | X | xx | xx-xx | X | XX | xx-xx | х | XX | xx-xx | Х | XX | xx-xx | X | XX | xx-xx |
| | Moderate | X | xx | xx-xx | X | XX | xx-xx | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Severe | X | xx | xx-xx | X | XX | xx-xx | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Pruritus | None | X | xx | xx-xx | X | XX | xx-xx | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Mild | X | xx | xx-xx | X | XX | xx-xx | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | X | XX | XX-XX | X | XX | xx-xx | X | XX | XX-XX |
| | Severe | X | xx | xx-xx | X | XX | xx-xx | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Ecchymosis | None | X | xx | xx-xx | X | XX | xx-xx | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Mild | X | xx | xx-xx | X | XX | xx-xx | Х | XX | xx-xx | X | XX | xx-xx | Х | XX | xx-xx |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |

Table 86: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, Treatment Arm and Age Stratum – Post Any Study Vaccination – Safety Population (continued)

| | | 3.7 | Group<br>5 mcg A/<br>+ AS03<br>(N=X) | H7N9<br>3 | 7.5 | Group 2<br>mcg A/H<br>+ AS03<br>(N=X) | 17N9 | 15 | Group 3<br>mcg A/H<br>+ AS03<br>(N=X) | | 15 | Group 4<br>mcg A/H<br>(N=X) | | 45 | Group 5<br>mcg A/H<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | 95% CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI |
| | Severe | х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Ecchymosis (measurement) | None | х | xx | xx-xx | X | XX | XX-XX | X | xx | XX-XX | X | xx | XX-XX | Х | XX | xx-xx |
| | Mild | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Severe | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Erythema | None | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Mild | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Severe | х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | xx | xx-xx | Х | XX | xx-xx |
| Erythema (measurement) | None | Х | xx | xx-xx | X | XX | XX-XX | X | xx | XX-XX | X | xx | XX-XX | X | XX | xx-xx |
| | Mild | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Severe | х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| Induration/Swelling | None | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Mild | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Severe | х | XX | xx-xx | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | XX-XX |
| Induration/Swelling (measurement) | None | х | xx | xx-xx | X | XX | XX-XX | X | xx | XX-XX | X | xx | xx-xx | X | XX | xx-xx |
| | Mild | Х | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |

Table 86: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, Treatment Arm and Age Stratum – Post Any Study Vaccination – Safety Population (continued)

| | | 3.75 | Group 1<br>5 mcg A/l<br>+ AS03<br>(N=X) | H7N9 | 7.5 | Group 2<br>mcg A/H<br>+ AS03<br>(N=X) | | 15 | Group 3<br>mcg A/H'<br>+ AS03<br>(N=X) | | 15 | Group 4<br>mcg A/H'<br>(N=X) | | <b>45</b> 1 | Group 5<br>mcg A/H'<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | 95% CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI |
| | Moderate | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx | X | XX | xx-xx |
| | Severe | X | XX | xx-xx | X | XX | XX-XX | X | XX | xx-xx | X | XX | XX-XX | X | XX | xx-xx |

N = Number of subjects in the Safety Population who received any study vaccination.

<sup>95%</sup> CI estimated using Clopper-Pearson exact method

Severity is the maximum severity reported over all solicited symptoms post dosing for each subject.

Table 87: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, Treatment Arm and Age Stratum Post Study Vaccination 1 – Safety Population \*

[Footnote Update] N = Number of subjects in the Safety Analysis Population who received the first study vaccination.

Table 88: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, Treatment Arm and Age Stratum Post Study Vaccination 2 – Safety Population \*

[Footnote Update] N = Number of subjects in the Safety Analysis Population who received the second study vaccination.

Table 89: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Day Post Study Vaccination, Treatment Arm and Age Stratum Post Any Study Vaccination – Safety Population

| Crimitan | Severity | Dwa | -Vac. | | ost-<br>ac. | Ъ | 1 | D | y 2 | D. | 2 | D. | ıy 4 | D | ıy 5 | D. | ny 6 | D. | 7 | D- | y 8+ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | -vac. | n | ac. | - | ay 1<br>% | n | y 2<br>% | n | y 3 | n | 1y 4<br> % | n | ly 5<br>% | n | 1y 6<br>% | n | y 7<br>% | n | y 8+<br>% |
| | | 11 | | <u> </u> | <u> </u> | | 1 | <u> </u> | AS03 ( | <u> </u> | | 11 | /0 | _ 11 | /0 | | /0 | | /0 | | /0 |
| All Subjects | | | G | Toup | 1. 5. | 75 IIIC | g M/II | 7117 | 1505 | (11 21) | , | | | | | | | | | | |
| Any Symptom | None | | | | | | | | | | | | | | | | | | | | |
| 7 my Symptom | Mild | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | |
| Any Systemic Symptom | None | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | |
| Fever | None | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | |
| Feverishness | None | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | |
| Fatigue | None | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | |
| Malaise | None | | | | | | | | | | | | | | | | | | | | |

Table 89: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Day Post Study Vaccination, Treatment Arm and Age Stratum – Post Any Study Vaccination – Safety Population (continued)

| Symptom | Severity | Pre | -Vac. | Po<br>V | ost-<br>ac. | Da | ay 1 | Da | ay 2 | Da | ıy 3 | Da | ay 4 | Da | ny 5 | Da | ıy 6 | Da | ny 7 | Da | y 8+ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | Mild | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | |
| Myalgia | None | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | |
| Arthralgia | None | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | |
| Headache | None | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | |
| Nausea | None | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | |
| Any Local Symptom | None | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | |

Table 89: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Day Post Study Vaccination, Treatment Arm and Age Stratum – Post Any Study Vaccination – Safety Population (continued)

| Symptom | Severity | Pre | -Vac. | Po<br>V | ost-<br>ac. | Da | ay 1 | Da | ny 2 | Da | ıy 3 | Da | ıy 4 | Da | ny 5 | Da | ny 6 | Da | ıy 7 | Da | y 8+ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Pain | None | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | |
| Tenderness | None | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | |
| Pruritus | None | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | |
| Ecchymosis | None | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | |
| Ecchymosis (measurement) | None | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | |
| Erythema | None | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | |

Table 89: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Day Post Study Vaccination, Treatment Arm and Age Stratum – Post Any Study Vaccination – Safety Population (continued)

| Symptom | Severity | Pre | -Vac. | | ost-<br>ac. | Da | ay 1 | Da | ny 2 | Da | ıy 3 | Da | ıy 4 | Da | ıy 5 | Da | y 6 | Da | ıy 7 | Da | y 8+ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | Severe | | | | | | | | | | | | | | | | | | | | |
| Erythema (measurement) | None | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | |
| Induration/Swelling | None | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | |
| Induration/Swelling (measurement) | None | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | |

[Repeat for Ages 19-64 and  $\geq$  65]

## [repeat for all treatment arms]

N = Number of subjects in the Safety Analysis Population who received any study vaccination. Severity is the maximum severity reported post dosing for each subject for each day.

Table 90: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Day Post Study Vaccination, Treatment Arm and Age Stratum Post Study Vaccination 1 – Safety Population

Footnote update: N = Number of subjects in the Safety Analysis Population who received the first study vaccination.

Table 91: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Day Post Study Vaccination, Treatment Arm and Age Stratum Post Study Vaccination 2 – Safety Population

Footnote update: N = Number of subjects in the Safety Analysis Population who received the second study vaccination.

Table 92: Number and Percentage of Subjects Experiencing Solicited Systemic Events for Dose 1 Compared with Dose 2 by Treatment Arm and Age Stratum – Safety Population

| | | | | Study Vaccination 2 | |
|---|---|---|---|---|---|
| Treatment<br>Arm | Age Stratum | Study Vaccination 1 | Subjects with No<br>Symptoms | Subjects with Mild or Greater<br>Symptoms | Total Number of Subjects<br>n (Percent)<br>[p-value*] |
| Group 1<br>3.75 mcg | Ages 19-64 | Subjects with No<br>Symptoms | x (%) | x (%) | x (%) |
| A/H7N9 +<br>AS03 | | Subjects with Mild or<br>Greater Symptoms | x (%) | x (%) | x (%) |
| | | Total Number of Subjects | x (%) | x (%) | x (100%)<br>[0.xxx] |
| | Ages ≥ 65 | Subjects with No<br>Symptoms | x (%) | x (%) | x (%) |
| | | Subjects with Mild or<br>Greater Symptoms | x (%) | x (%) | x (%) |
| | | Total Number of Subjects | x (%) | x (%) | x (100%)<br>[0.xxx] |
| | All Subjects | Subjects with No<br>Symptoms | x (%) | x (%) | x (%) |
| | | Subjects with Mild or<br>Greater Symptoms | x (%) | x (%) | x (%) |
| | | Total Number of Subjects | x (%) | x (%) | x (100%)<br>[0.xxx] |
| Group 2<br>7.5 mcg | Ages 19-64 | Subjects with No<br>Symptoms | x (%) | x (%) | x (%) |
| A/H7N9 +<br>AS03 | | Subjects with Mild or<br>Greater Symptoms | x (%) | x (%) | x (%) |
| | | Total Number of Subjects | x (%) | x (%) | x (100%)<br>[0.xxx] |
| | Ages ≥ 65 | Subjects with No Symptoms | x (%) | x (%) | x (%) |
| | | Subjects with Mild or<br>Greater Symptoms | x (%) | x (%) | x (%) |

Table 92: Number and Percentage of Subjects Experiencing Solicited Systemic Events for Dose 1 Compared with Dose 2 by Treatment Arm and Age Stratum – Safety Population (continued)

| | | | | Study Vaccination 2 | |
|---|---|---|---|---|---|
| Treatment<br>Arm | Age Stratum | Study Vaccination 1 | Subjects with No<br>Symptoms | Subjects with Mild or Greater<br>Symptoms | Total Number of Subjects<br>n (Percent)<br>[p-value*] |
| | | Total Number of Subjects | x (%) | x (%) | x (100%)<br>[0.xxx] |
| | All Subjects | Subjects with No<br>Symptoms | x (%) | x (%) | x (%) |
| | | Subjects with Mild or<br>Greater Symptoms | x (%) | x (%) | x (%) |
| | | Total Number of Subjects | x (%) | x (%) | x (100%)<br>[0.xxx] |
| Group 3<br>15 mcg | Ages 19-64 | Subjects with No<br>Symptoms | x (%) | x (%) | x (%) |
| A/H7N9 +<br>AS03 | | Subjects with Mild or<br>Greater Symptoms | x (%) | x (%) | x (%) |
| | | Total Number of Subjects | x (%) | x (%) | x (100%)<br>[0.xxx] |
| | Ages ≥ 65 | Subjects with No<br>Symptoms | x (%) | x (%) | x (%) |
| | | Subjects with Mild or<br>Greater Symptoms | x (%) | x (%) | x (%) |
| | | Total Number of Subjects | x (%) | x (%) | x (100%)<br>[0.xxx] |
| | All Subjects | Subjects with No<br>Symptoms | x (%) | x (%) | x (%) |
| | | Subjects with Mild or<br>Greater Symptoms | x (%) | x (%) | x (%) |
| | | Total Number of Subjects | x (%) | x (%) | x (100%)<br>[0.xxx] |
| | Ages 19-64 | Subjects with No<br>Symptoms | x (%) | x (%) | x (%) |

Table 92: Number and Percentage of Subjects Experiencing Solicited Systemic Events for Dose 1 Compared with Dose 2 by Treatment Arm and Age Stratum – Safety Population (continued)

| | | | | Study Vaccination 2 | |
|---|---|---|---|---|---|
| Treatment<br>Arm | Age Stratum | Study Vaccination 1 | Subjects with No<br>Symptoms | Subjects with Mild or Greater<br>Symptoms | Total Number of Subjects<br>n (Percent)<br>[p-value*] |
| Group 4<br>15 mcg | | Subjects with Mild or<br>Greater Symptoms | x (%) | x (%) | x (%) |
| A/H7N9 | | Total Number of Subjects | x (%) | x (%) | x (100%)<br>[0.xxx] |
| | Ages ≥ 65 | Subjects with No<br>Symptoms | x (%) | x (%) | x (%) |
| | | Subjects with Mild or<br>Greater Symptoms | x (%) | x (%) | x (%) |
| | | Total Number of Subjects | x (%) | x (%) | x (100%)<br>[0.xxx] |
| | All Subjects | Subjects with No<br>Symptoms | x (%) | x (%) | x (%) |
| | | Subjects with Mild or<br>Greater Symptoms | x (%) | x (%) | x (%) |
| | | Total Number of Subjects | x (%) | x (%) | x (100%)<br>[0.xxx] |
| Group 5<br>45 mcg | Ages 19-64 | Subjects with No<br>Symptoms | x (%) | x (%) | x (%) |
| A/H7N9 | | Subjects with Mild or<br>Greater Symptoms | x (%) | x (%) | x (%) |
| | | Total Number of Subjects | x (%) | x (%) | x (100%)<br>[0.xxx] |
| | Ages ≥ 65 | Subjects with No<br>Symptoms | x (%) | x (%) | x (%) |
| | | Subjects with Mild or<br>Greater Symptoms | x (%) | x (%) | x (%) |
| | | Total Number of Subjects | x (%) | x (%) | x (100%)<br>[0.xxx] |

Table 92: Number and Percentage of Subjects Experiencing Solicited Systemic Events for Dose 1 Compared with Dose 2 by Treatment Arm and Age Stratum – Safety Population (continued)

| | | | Study Vaccination 2 | | |
|---|---|---|---|---|---|
| Treatment<br>Arm | Age Stratum | Study Vaccination 1 | Subjects with No<br>Symptoms | Subjects with Mild or Greater<br>Symptoms | Total Number of Subjects<br>n (Percent)<br>[p-value*] |
| | All Subjects | Subjects with No Symptoms | x (%) | x (%) | x (%) |
| | | Subjects with Mild or<br>Greater Symptoms | x (%) | x (%) | x (%) |
| | | Total Number of Subjects | x (%) | x (%) | x (100%)<br>[0.xxx] |

Note: Denominators for percentages are the number of subjects in the safety population who received both the first and second study vaccination. [x] subjects did not get the second dose and are not included in this table.

Table with similar format:

Table 93: Number and Percentage of Subjects Experiencing Solicited Local Events for Dose 1 Compared with Dose 2 by Treatment Arm and Age Stratum – Safety Population

<sup>\*</sup> P-value is calculated from McNemar's test for each group and age stratum pair.

## 14.3.1.2 Unsolicited Adverse Events

Table 94: Number and Percentage of Subjects Experiencing Unsolicited Adverse Events with 95% Confidence Intervals by MedDRA System Organ Class and Preferred Term, and Treatment Arm – Safety Population \*

| | | 3.75<br>A/H<br>+ A | oup 1<br>5 mcg<br>17N9<br>AS03<br>=X) | Group 2<br>7.5 mcg A/H7N9<br>+ AS03<br>(N=X) | | 7.5 mcg A/H7N9<br>+ AS03 | | Group 3<br>15 mcg A/H7N9<br>+ AS03<br>(N=X) | | 15 mcg A/H7N9<br>+ AS03 | | Group 4<br>15 mcg A/H7N9<br>(N=X) | Group 5<br>45 mcg A/H7N<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| MedDRA System<br>Organ Class | MedDRA<br>Preferred Term | n | %<br>(95%<br>CI) | n | %<br>(95%<br>CI) | n | %<br>(95%<br>CI) | n | %<br>(95%<br>CI) | n | %<br>(95%<br>CI) | | |
| Any SOC | Any PT | X | xx<br>(xx-xx) | Х | xx<br>(xx-xx) | х | xx<br>(xx-xx) | х | xx<br>(xx-xx) | х | xx<br>(xx-xx) | | |
| [SOC 1] | Any PT | | | | | | | | | | | | |
| | [PT 1] | | | | | | | | | | | | |
| | [PT 2] | | | | | | | | | | | | |
| [SOC 2] | Any PT | | | | | | | | | | | | |
| | [PT 1] | | | | | | | | | | | | |
| | [PT 2] | | | . 1 | · | . 1.1 | . 1 | | | 1: .: | 1 . 1 | | |

Note: N = number of subjects in the Safety Analysis Population who received any study vaccination. This table presents number and percentage of subjects. A subject is only counted once per PT.

Table 95: Number and Percentage of Subjects Experiencing Unsolicited Adverse Events with 95% Confidence Intervals by MedDRA System Organ Class and Preferred Term, Treatment Arm and Age Stratum – Safety Population \*

| MedDRA<br>System<br>Organ<br>Class | MedDRA<br>Preferred<br>Term | | Group 1<br>3.75 mcg A/H7N9<br>+ AS03<br>(N=X) | | | Group 2<br>7.5 mcg A/H7N9<br>+ AS03<br>(N=X) | | | Group 3<br>15 mcg A/H7N9<br>+ AS03<br>(N=X) | | | N9 | | 15 mcg | roup 4<br>g A/H7N9<br>N=X) | | | Gro<br>45 mcg .<br>(N= | A/H7N | N9 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 1 | 9-64 | 2 | ≥ 65 | 1: | 9-64 | 2 | ≥ 65 | 1 | 9-64 | 2 | ≥ 65 | 1 | 9-64 | 2 | ≥ 65 | 1 | 9-64 | 2 | ≥ 65 |
| | | n | %<br>(95%<br>CI) | n | %<br>(95%<br>CI) | n | %<br>(95%<br>CI) | n | %<br>(95%<br>CI) | n | %<br>(95%<br>CI) | n | %<br>(95%<br>CI) | n | %<br>(95%<br>CI) | n | %<br>(95%<br>CI) | n | %<br>(95%<br>CI) | n | %<br>(95%<br>CI) |
| Any SOC | Any PT | Х | xx<br>(xx-<br>xx) | Х | xx<br>(xx-<br>xx) | Х | xx<br>(xx-<br>xx) | Х | xx<br>(xx-<br>xx) | Х | xx<br>(xx-<br>xx) | Х | xx<br>(xx-<br>xx) | х | xx<br>(xx-<br>xx) | Х | xx<br>(xx-<br>xx) | Х | xx<br>(xx-<br>xx) | Х | xx<br>(xx-<br>xx) |
| [SOC 1] | Any PT | | | | | | | | | | | | | | | | | | | | |
| | [PT 1] | | | | | | | | | | | | | | | | | | | | |
| | [PT 2] | | | | | | | | | | | | | | | | | | | | |
| [SOC 2] | Any PT | | | | | | | | | | | | | | | | | | | | |
| | [PT 1] | | | | | | | | | | | | | | | | | | | | |
| | [PT 2] | | | | | | | | | | | | | | | | | | | | |

Note: N = number of subjects in the Safety Analysis Population who received any study vaccination. This table presents number and percentage of subjects. A subject is only counted once per PT.

Table 96: Number and Percentage of Subjects Experiencing Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Maximum Severity, Relationship, Treatment Arm and Age Stratum – Safety Population\*

| MedDRA System Organ Class | MedDRA Preferred Term | Any In | cidence | | | Sever | ity [1] | | | Rela | ationship to | Treatme | nt [2] |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | Mild | | Moderate | | vere | Not Related | | Related | |
| | | n | % | n | % | n | % | n | % | n | % | n | % |
| | Gr | oup 1 3.7 | 5 mcg A/l | H7N9 + | AS03 ( | (N = X) | | | | | | | |
| All Subjects | | | | | | | | | | | | | |
| Any SOC | Any PT | х | XX | х | XX | х | XX | X | xx | X | xx | х | XX |
| [SOC 1] | Any PT | | | | | | | | | | | | |
| | [PT 1] | | | | | | | | | | | | |
| | [PT 2] | | | | | | | | | | | | |
| [SOC 2] | Any PT | | | | | | | | | | | | |
| | [PT 1] | | | | | | | | | | | | |
| | [PT 2] | | | | | | | | | | | | |
| [repeat for Ages 19-64 and $\geq$ 65] | • | • | | | | | • | | | | • | • | • |
| | | [Repea | t for all t | reatme | nt arms | s] | | | | | | | |

<sup>[1]</sup> For severity, a subject is counted once per preferred term and is summarized according to their highest severity.

<sup>[2]</sup> For relationship, a subject is only counted once per preferred term and is summarized according to their closest relationship.

Table 97: Number and Percentage of Subjects Experiencing Non-Serious Related Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Maximum Severity, Treatment Arm and Age Stratum – Safety Population

| MedDRA System Organ Class | MedDRA Preferred Term | Any Ir | icidence | | | Sever | ity [1] | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | M | lild | Mod | erate | Sev | vere |
| | | n | % | n | % | n | % | n | % |
| | Group 1 3.75 mcg A/H | 7N9 + AS03 ( | N=X) | • | | | | | |
| All Subjects | | | | | | | | | |
| Any SOC | Any PT | х | xx | X | XX | х | XX | х | XX |
| [SOC 1] | Any PT | х | xx | X | XX | х | XX | х | XX |
| | [PT 1] | | | | | | | | |
| | [PT 2] | | | | | | | | |
| [SOC 2] | Any PT | | | | | | | | |
| | [PT 1] | | | | | | | | |
| | [PT 2] | | | | | | | | |
| [Repeat for Ages 19-64 and ≥ 65] | | • | | • | • | • | • | • | • |
| | [Repeat for all tre | atment arms | | | | | | | |
| Note: N = Number of subjects in the Safety A | nalysis Population. This table presents numb | er and percent | age of subject | cts. | | | | | |

[1] For severity, a subject is counted once per preferred term and is summarized according to their highest severity.

Table 98: Number and Percentage of Subjects Experiencing Unsolicited Adverse Events Within 21 Days Post Study Vaccination by MedDRA System Organ Class and Preferred Term, Day Post Vaccination, Treatment Arm and Age Stratum – Safety Population

| | | Day 1-8<br>Post Vac 1 | | Day 9-22<br>Post Vac 1 | | Day 1-22<br>Post Vac 1 | | Day 1-8<br>Post Vac 2 | | Day 9-22<br>Post Vac 2 | | Day 1-22<br>Post Vac 2 | | Day 1-22<br>Post Any<br>Vaccination | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| MedDRA System Organ Class | MedDRA Preferred<br>Term | n | % | n | n % n % n % n % | | % | n | % | | | | | | |
| | | Group | p 1 3.75 | mcg A/l | H7N9 + | AS03, ( | N=X) | | | | | | | | |
| All Subjects | | | | | | | | | | | | | | | |
| Any SOC | Any PT | X | XX | х | XX | X | XX | x | XX | x | XX | X | XX | х | XX |
| [SOC 1] | Any PT | | | | | | | | | | | | | | |
| | [PT 1] | | | | | | | | | | | | | | |
| | [PT 2] | | | | | | | | | | | | | | |
| [SOC 2] | Any PT | | | | | | | | | | | | | | |
| | [PT 1] | | | | | | | | | | | | | | |
| | [PT 2] | | | | | | | | | | | | | | |
| [Repeat for Ages 19-64 and $\geq$ 65] | 1 | | | • | | | • | • | | • | | • | | • | |
| | | ı | Repeat | for all t | reatmen | t arms] | | | | | | | | | |

Note: N = Number of subjects in the Safety Analysis Population. This table presents number and percentage of subjects. For each time period, a subject is only counted once per PT.

Table 99: Number and Percentage of Subjects Experiencing Non-Serious, Related Unsolicited Adverse Events Within 21 Days Post Vaccination by MedDRA System Organ Class and Preferred Term, Study Vaccination, Treatment Arm and Age Stratum – Safety Population

| | | | y 1-8<br>Vac 1 | Day<br>Post | | | Day 1-22 Post Vac 1 Post Vac 2 Post Vac 2 | | Day 1-22<br>Post Vac 2 | | Day 1-22<br>Post Any<br>Vaccinatio | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| MedDRA System Organ Class | MedDRA Preferred<br>Term | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | | Group | p 1 3.75 | mcg A/l | H7N9 + | AS03 ( | N=X) | | | | | | | | |
| All Subjects | | | | | | | | | | | | | | | |
| Any SOC | Any PT | х | xx | X | XX | X | xx | х | xx | х | xx | х | XX | x | xx |
| [SOC 1] | Any PT | | | | | | | | | | | | | | |
| | [PT 1] | | | | | | | | | | | | | | |
| | [PT 2] | | | | | | | | | | | | | | |
| [SOC 2] | Any PT | | | | | | | | | | | | | | |
| | [PT 1] | | | | | | | | | | | | | | |
| | [PT 2] | | | | | | | | | | | | | | |
| [Repeat for Ages 19-64 and $\geq$ 65] | • | • | • | | | | • | | • | | | | • | • | |
| | | ſ | Repeat | for all ti | eatmen | t arms] | | | | | | | | | |

Table 100: Number of Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Day Post Vaccination, Treatment Arm and Age Stratum – Safety Population

| | | Day 1-8<br>Post Vac 1 | Day 9-22<br>Post Vac 1 | Day 1-22<br>Post Vac 1 | Day 1-8<br>Post Vac 2 | Day 9-22<br>Post Vac 2 | Day 1-22<br>Post Vac 2 | Day 1-22<br>Post Any<br>Vaccination |
|---|---|---|---|---|---|---|---|---|
| MedDRA System Organ Class | MedDRA Preferred Term | # of Events | # of<br>Events | # of Events | # of Events | # of Events | # of Events | # of Events |
| | ( | Group 1 3.75 n | ncg A/H7N9 + | AS03 (N=X) | | | | |
| All Subjects | | | | | | | | |
| Any SOC | Any PT | х | X | X | X | X | X | X |
| [SOC 1] | Any PT | | | | | | | |
| | [PT 1] | | | | | | | |
| | [PT 2] | | | | | | | |
| [SOC 2] | Any PT | | | | | | | |
| | [PT 1] | | | | | | | |
| | [PT 2] | | | | | | | |
| [Repeat for Ages 19-64 and $\geq$ 65] | | | | | | | | |
| | | [Repeat fo | r all treatmer | nt arms] | | | | |
| Note: $N = Number of subjects in th$ | e Safety Analysis Population. T | his table presen | ts number of e | vents; a subject | may be counted | multiple times. | | |
## 14.3.2 Listings of Serious and Significant Adverse Events

## Table 101: Listing of Serious Adverse Events – Safety Population \*

[Implementation Note: This listing is included in the table shells document, as it is included in the body of the CSR. If the event is ongoing (no stop date), indicate "ongoing" in the "Duration" column. If more than one reason is selected for the reason reported as an SAE, list all reasons in the column, separated by a comma. In the "If Not Related, Alternate Etiology" column, merge the 2 data fields for collecting alternate etiology, separate by a colon. In the CSR, Subject ID should be USUBJID (not PATID) for purposes of de-identification.]

| Adverse<br>Event | Associated<br>with Vac # | # of Days<br>Post<br>Associated<br>Dose<br>(Duration) | # of Days Post Vac the Event Became Serious | Reason<br>Reported<br>as an SAE | Severity | Relationship<br>to Study<br>Treatment | In Not<br>Related,<br>Alternative<br>Etiology | Action<br>Taken with<br>Study<br>Treatment | Subject<br>Discontinued<br>Due to AE | Outcome | MedDRA<br>System<br>Organ<br>Class | MedDRA<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject II | ): , Treatmo | ent Arm: , A | E Numbe | er: | | | | | | | | |
| Comments | : | | | | | | | | | | | |
| Subject II | ): , Treatmo | ent Arm: , A | E Numbe | er: | | | | | | | | |
| Comments | : | | <u>'</u> | | | | | • | 1 | | | |

## Table 102: Listing of Adverse Events of Special Interest – Safety Population \*

[Implementation Note: This listing is included in the tables section, as it is included in the body of the CSR. If the event is ongoing (no stop date), indicate "ongoing" in the "Duration" column. In the "If Not Related, Alternate Etiology" column, merge the 2 data fields for collecting alternate etiology, separate by a colon.]

| Adverse<br>Event | Associated with Vac # | # of Days Post Associated Vac (Duration) | SAE?<br>Severity | Relationship<br>to Study<br>Treatment | In Not<br>Related,<br>Alternative<br>Etiology | Action<br>Taken<br>with<br>Study<br>Treatment | Subject<br>Discontinued<br>Due to AE | Outcome | MAAE | MedDRA<br>System<br>Organ<br>Class | MedDRA<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject II | D: , Treatm | ent Arm: , | AE Number | <b>:</b> | | | | | | | |
| | | | SAE: No<br>Mild | | | | | | | | |
| Comments | S: | | | | | | | | | | |
| Subject II | D: , Treatm | ent Arm: , | AE Number | ·: | | | | | | | |
| Comments | s: | | | | | | | | | | |

Tables with similar format:

Table 103: Listing of New Onset Chronic Medical Conditions – Safety Population \*

Table 104: Listing of Non-Serious, Unsolicited, Moderate or Severe Adverse Events - Safety Population \*

# 14.3.3 Narratives of Deaths, Other Serious and Significant Adverse Events

(not included in SAP, but this is a placeholder for the CSR)

## 14.3.4 Displays of Laboratory Results

Table 105: Laboratory Results by Parameter, Maximum Severity, Study Day, Treatment Group and Age Stratum, All Laboratory Parameters – Safety Population \*

| Treatment<br>Group | Age<br>Stratum | Study Day | N | N* | N | one | | ild/<br>ide 1 | | erate/<br>ide 2 | | ere/<br>de 3 | Mis | ssing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | n | % | n | % | n | % | n | % | n | % |
| Group 1<br>3.75 mcg<br>A/H7N9 +<br>AS03 | Ages 19-64 | Baseline | х | х | X | xx | х | xx | X | xx | х | xx | х | XX |
| | | Day 8 | | | | | | | | | | | | |
| | | Day 22 | | | | | | | | | | | | |
| | | Day 29 | | | | | | | | | | | | |
| | | Max Severity Post<br>Baseline | | | | | | | | | | | | |
| | Ages ≥ 65 | Baseline | | | | | | | | | | | | |
| | | Day 8 | | | | | | | | | | | | |
| | | Day 22 | | | | | | | | | | | | |
| | | Day 29 | | | | | | | | | | | | |
| | | Max Severity Post<br>Baseline | | | | | | | | | | | | |
| | All<br>Subjects | Baseline | | | | | | | | | | | | |
| | | Day 8 | | | | | | | | | | | | |
| | | Day 22 | | | | | | | | | | | | |
| | | Day 29 | | | | | | | | | | | | |
| | | Max Severity Post<br>Baseline | | | | | | | | | | | | |
| [Repeat for all<br>Treatment<br>Arms] | | | | | | | | | | | | | | |

Table 105: Laboratory Results by Parameter, Maximum Severity, Study Day, Treatment Group and Age Stratum, All Laboratory Parameters – Safety Population \* (continued)

| Treatment<br>Group | Age<br>Stratum | Study Day | N | N* | No | one | Mi<br>Gra | ild/<br>ide 1 | Mode<br>Gra | erate/<br>de 2 | Sev<br>Gra | | Mis | sing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | n | % | n | % | n | % | n | % | n | % |

Note: The "Max Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments. N\* is the denominator for calculating percentages.

N=Number of subjects in the Safety population; N\*=Number of subjects who completed the indicated visit.

#### Tables with similar format:

- Table 106: Laboratory Results by Parameter, Maximum Severity, Study Day, Treatment Group and Age Stratum, Hemoglobin Safety Population \*
- Table 107: Laboratory Results by Parameter, Maximum Severity, Study Day, Treatment Group and Age Stratum, Alanine Safety Population aminotransferase (ALT)\*
- Table 108: Laboratory Results by Parameter, Maximum Severity, Study Day, Treatment Group and Age Stratum, Total Bilirubin Safety Population \*
- Table 109: Laboratory Results by Parameter, Maximum Severity, Study Day, Treatment Group and Age Stratum, Creatinine Safety Population \*

Table 110: Laboratory Results by Parameter, Maximum Severity, Study Day, Treatment Arm and Age Stratum, White Blood Cells – Safety Population \*

| Treatment<br>Group | Age<br>Stratum | Study Day | N | N* | None | | Gra | ild/<br>ide 1<br>ow) | Gra | ild/<br>ide 1<br>igh) | Gra | erate/<br>de 2<br>ow) | Gra | erate/<br>ide 2<br>igh) | Gra | rere/<br>ide 3<br>ow) | Gra | rere/<br>ide 3<br>igh) | Mis | sing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Group 1<br>3.75 mcg<br>A/H7N9 +<br>AS03 | Ages 19-<br>64 | Baseline | Х | Х | х | xx | х | xx | х | xx | х | xx | х | xx | х | xx | х | xx | х | XX |
| | | Day 8 | | | | | | | | | | | | | | | | | | |
| | | Day 22 | | | | | | | | | | | | | | | | | | |
| | | Day 29 | | | | | | | | | | | | | | | | | | |
| | | Max<br>Severity<br>Post<br>Baseline | | | | | | | | | | | | | | | | | | |
| | Ages ≥ 65 | Baseline | | | | | | | | | | | | | | | | | | |
| | | Day 8 | | | | | | | | | | | | | | | | | | |
| | | Day 22 | | | | | | | | | | | | | | | | | | |
| | | Day 29 | | | | | | | | | | | | | | | | | | |
| | | Max<br>Severity<br>Post<br>Baseline | | | | | | | | | | | | | | | | | | |
| | All<br>Subjects | Baseline | | | | | | | | | | | | | | | | | | |
| | | Day 8 | | | | | | | | | | | | | | | | | | |
| | | Day 22 | | | | | | | | | | | | | | | | | | |
| | | Day 29 | | | | | | | | | | | | | | | | | | |

Table 110: Laboratory Results by Parameter, Maximum Severity, Study Day, Treatment Arm and Age Stratum – White Blood Cells – Safety Population (continued)

| Treatment<br>Group | Age<br>Stratum | Study Day | N | N* | None | | Gra | ild/<br>de 1<br>ow) | Mi<br>Gra<br>(Hi | | Gra | erate/<br>de 2<br>ow) | Gra | erate/<br>de 2<br>gh) | Sev<br>Gra<br>(Lo | | Gra | ere/<br>de 3<br>igh) | Mis | sing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | | Max<br>Severity<br>Post<br>Baseline | | | | | | | | | | | | | | | | | | |
| [Repeat for all<br>Treatment<br>Arms] | | | | | | | | | | | | | | | | | | | | |

Note: The "Max Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments. N\* is the denominator for calculating percentages.

N=Number of subjects in the Safety population; N\*=Number of subjects who completed the indicated visit.

Table with similar format:

Table 111: Laboratory Results by Parameter, Maximum Severity, Study Day, Treatment Arm and Age Stratum, Platelets – Safety Population \*

Table 112: Laboratory Summary Statistics by Parameter, Study Day, Treatment Arm and Age Stratum, White Blood Cells – Safety **Population \*** 

| Treatment Group | Age Stratum | Study Day | N | Mean | Standard<br>Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|---|
| Group 1<br>3.75 mcg A/H7N9 + AS03 | Ages 19-64 | Baseline | Х | xx.x | xx.x | XX | xx, xx |
| | | Day 8 | | | | | |
| | | Day 22 | | | | | |
| | | Day 29 | | | | | |
| | Ages ≥ 65 | Baseline | | | | | |
| | | Day 8 | | | | | |
| | | Day 22 | | | | | |
| | | Day 29 | | | | | |
| | All Subjects | Baseline | | | | | |
| | | Day 8 | | | | | |
| | | Day 22 | | | | | |
| | | Day 29 | | | | | |
| [Repeat for all Treatment Arms] | | | | | | | |

#### Tables with similar format:

- Table 113: Laboratory Summary Statistics by Parameter, Study Day, Treatment Arm and Age Stratum, Hemoglobin Safety **Population \***
- Table 114: Laboratory Summary Statistics by Parameter, Study Day, Treatment Arm and Age Stratum, Platelets Safety Population \*
- Table 115: Laboratory Summary Statistics by Parameter, Study Day, Treatment Arm and Age Stratum, Alanine Aminotransferase **Safety Population \* (ALT)**
- Table 116: Laboratory Summary Statistics by Parameter, Study Day, Treatment Arm and Age Stratum, Total Bilirubin Safety **Population \***

- Table 117: Laboratory Summary Statistics by Parameter, Study Day, Treatment Arm and Age Stratum, Creatinine Safety Population \*
- Table 118: Laboratory Summary Statistics of Change from Baseline by Parameter, Study Day, Treatment Arm and Age Stratum, White Blood Cells Safety Population \*
- Table 119: Laboratory Summary Statistics of Change from Baseline by Parameter, Study Day, Treatment Arm and Age Stratum, Hemoglobin Safety Population \*
- Table 120: Laboratory Summary Statistics of Change from Baseline by Parameter, Study Day, Treatment Arm and Age Stratum, Platelets Safety Population \*
- Table 121: Laboratory Summary Statistics of Change from Baseline by Parameter, Study Day, Treatment Arm and Age Stratum, Alanine aminotransferase (ALT) Safety Population \*
- Table 122: Laboratory Summary Statistics of Change from Baseline by Parameter, Study Day, Treatment Arm and Age Stratum, Total Bilirubin Safety Population \*
- Table 123: Laboratory Summary Statistics of Change from Baseline by Parameter, Study Day, Treatment Arm and Age Stratum, Creatinine Safety Population \*

# 14.3.4.5 Clinical Laboratory Reference Ranges

(Placeholder for the CSR)

# 14.3.5 Abnormal Laboratory Value Listings (by Subject)

**Table 124: Listing of Abnormal Laboratory Results - Chemistry** 

| Subject<br>ID | Treatment<br>Arm | Age<br>Stratum | Sex | Age<br>(years) | Planned<br>Time<br>Point | Actual<br>Study<br>Day | Laboratory<br>Parameter<br>(Units) | Result<br>(Severity) | Relationship<br>to Treatment | If Not<br>Related,<br>Alternate<br>Etiology | Action<br>Taken<br>with Study<br>Treatment | Subject Discontinued Due to Result? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|

| Subject<br>ID | Treatment<br>Arm | Age<br>Stratum | Sex | Age<br>(years) | Planned<br>Time<br>Point | Actual<br>Study<br>Day | Laboratory<br>Parameter<br>(Units) | Result<br>(Severity) | Relationship<br>to Treatment | If Not<br>Related,<br>Alternate<br>Etiology | Action<br>Taken<br>with Study<br>Treatment | Subject Discontinued Due to Result? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|

## 14.3.6 Displays of Vital Signs

Table 126: Vital Signs by Assessment, Maximum Severity, Study Day, Treatment Arm and Age Stratum, Any Assessment – Safety Population \*

| Treatment | Age | Study Day | N | N* | No | ne | M | ild | Mod | erate | Sev | ere | Mis | sing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Group | Stratum | | | | n | % | n | % | n | % | n | % | n | % |
| Group 1<br>3.75 mcg A/H7N9<br>+ AS03 | Ages 19-64 | Baseline | х | х | X | XX | X | XX | X | XX | Х | XX | X | XX |
| | | Day 22 | | | | | | | | | | | | |
| | | Max Severity Post<br>Baseline | | | | | | | | | | | | |
| | Ages ≥ 65 | Baseline | | | | | | | | | | | | |
| | | Day 22 | | | | | | | | | | | | |
| | | Max Severity Post<br>Baseline | | | | | | | | | | | | |
| | All Subjects | Baseline | | | | | | | | | | | | |
| | | Day 22 | | | | | | | | | | | | |
| | | Max Severity Post<br>Baseline | | | | | | | | | | | | |
| [Repeat for all<br>Treatment Arms] | | | | | | | | | | | | | | |

Note: The "Max Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments. N\* is the denominator for calculating percentages.

N=Number of subjects in the Safety population; N\*=Number of subjects who completed the indicated visit.

Table with similar format:

Table 127: Vital Signs by Assessment, Maximum Severity, Study Day, Treatment Arm and Age Stratum, Oral Temperature – Safety Population

Table 128: Vital Signs by Assessment, Maximum Severity, Study Day, Treatment Arm and Age Stratum, Systolic Blood Pressure – Safety Population

| Treatment<br>Group | Age<br>Stratum | Study Day | N | N* | No | one | | ild<br>ow) | | ild<br>gh) | | erate<br>ow) | | erate<br>gh) | | vere<br>ow) | | ere<br>igh) | Mis | ssing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Group 1<br>3.75 mcg<br>A/H7N9 +<br>AS03 | Ages 19-64 | Baseline | х | Х | х | xx | х | xx | Х | XX | х | xx | Х | XX | х | xx | х | xx | х | XX |
| | | Day 22 | | | | | | | | | | | | | | | | | | |
| | | Max Severity<br>Post Baseline | | | | | | | | | | | | | | | | | | |
| | Ages ≥ 65 | Baseline | | | | | | | | | | | | | | | | | | |
| | | Day 22 | | | | | | | | | | | | | | | | | | |
| | | Max Severity<br>Post Baseline | | | | | | | | | | | | | | | | | | |
| | All Subjects | Baseline | | | | | | | | | | | | | | | | | | |
| | | Day 22 | | | | | | | | | | | | | | | | | | |
| | | Max Severity<br>Post Baseline | | | | | | | | | | | | | | | | | | |
| [Repeat for<br>all<br>Treatment<br>Arms] | M. D. (D. | | | | | | | | | | | 1: | | | | | | | | |

Note: The "Max Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments. N\* is the denominator for calculating percentages.

N=Number of subjects in the Safety population; N\*=Number of subjects who completed the indicated visit.

### Tables with similar format:

- Table 129: Vital Signs by Assessment, Maximum Severity, Study Day, Treatment Arm and Age Stratum, Diastolic Blood Pressure Safety Population
- Table 130: Vital Signs by Assessment, Maximum Severity, Study Day, Treatment Arm and Age Stratum, Pulse Safety Population

## 14.4 Summary of Concomitant Medications

Table 131: Number and Percentage of Subjects with Prior and Concurrent Medications by WHO Drug Classification and Treatment Arm – Safety Population

| WHO Drug Code<br>Level 1, Anatomic Group | WHO Drug Code<br>Level 2, Therapeutic<br>Subgroup | 3.75 mcg<br>+ A | oup 1<br>g A/H7N9<br>aS03<br>=X) | 7.5 mcg<br>+ A | oup 2<br>A/H7N9<br>.S03<br>=X) | 15 mcg<br>+ A | oup 3<br>A/H7N9<br>S03<br>=X) | 15 mcg | up 4<br>A/H7N9<br>=X) | 45 mcg | oup 5<br>A/H7N9<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | n | % | n | % | n | % | n | % |
| Any Level 1 Codes | Any Level 2 Codes | х | xx | x | xx | х | xx | х | xx | х | xx |
| [ATC Level 1 - 1] | Any [ATC 1 – 1] | | | | | | | | | | |
| | [ATC 2 - 1] | | | | | | | | | | |
| | [ATC 2 - 2] | | | | | | | | | | |
| | [ATC 2 - 3] | | | | | | | | | | |
| [ATC Level 1 – 2] | [ATC 2 - 1] | | | | | | | | | | |
| | [ATC 2 - 2] | | | | | | | | | | |
| N. N. J. C. Lincial C. | [ATC 2 - 3] | 6 1: | | | | | | | | | |

N= Number of subjects in the Safety population. n=Number of subjects reporting taking at least one medication in the specific WHO Drug Class.

Table 132: Number and Percentage of Subjects with Prior and Concurrent Medications by WHO Drug Classification, Treatment Arm and Age Stratum – Safety Population

| WHO Drug Code<br>Level 1, Anatomic<br>Group | WHO Drug Code<br>Level 2,<br>Therapeutic<br>Subgroup | Group 1 3.75 mcg A/H7N9 + AS03 (N=X) 19-64 ≥ 65 | | Group 2<br>7.5 mcg A/H7N9<br>+ AS03<br>(N=X) | | | Group 3<br>15 mcg A/H7N9<br>+ AS03<br>(N=X) | | | Group 4<br>15 mcg A/H7N9<br>(N=X) | | | Group 5<br>45 mcg A/H7N9<br>(N=X) | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | ≥ 65 | | 19-64 | | ≥ 65 | 19-64 | | ≥ | 65 | 19-64 | | ≥ 65 | | 19-64 | | ≥ 65 | | |
| | | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Any Level 1 Codes | Any Level 2 Codes | Х | XX | Х | xx | Х | XX | X | XX | X | xx | Х | XX | X | xx | X | XX | Х | XX | X | xx |
| [ATC Level 1 - 1] | Any [ATC 1 – 1] | | | | | | | | | | | | | | | | | | | | |
| | [ATC 2 - 1] | | | | | | | | | | | | | | | | | | | | |
| | [ATC 2 - 2] | | | | | | | | | | | | | | | | | | | | |
| | [ATC 2 - 3] | | | | | | | | | | | | | | | | | | | | |
| [ATC Level 1 – 2] | [ATC 2 - 1] | | | | | | | | | | | | | | | | | | | | |
| | [ATC 2 - 2] | | | | | | | | | | | | | | | | | | | | |
| | [ATC 2 - 3] | | | | | | | | | | | | | | | | | | | | |

N= Number of subjects in the Safety population. n=Number of subjects reporting taking at least one medication in the specific WHO Drug Class.

# APPENDIX 2. FIGURE MOCK-UPS

# **LIST OF FIGURES**

| Figure 1: | CONSORT Flow Diagram*157 |
|---|---|
| Figure 2: | Reverse Cumulative Distribution of Hemagglutination Inhibition Antibody |
| C | against 2017 A/H7N9 by Study Day, Treatment Arm and Age Stratum, Modified Intent |
| | to Treat Population* |
| Figure 3: | Reverse Cumulative Distribution of Hemagglutination Inhibition Antibody against |
| | 2017 A/H7N9 by Study Day, Treatment Arm and Age Stratum, Per Protocol |
| | Population* |
| Figure 4: | Reverse Cumulative Distribution of Neutralizing Antibody Against 2017 A/H7N9 by |
| | Study Day, Treatment Arm and Age Stratum, Modified Intent to Treat Population* 158 |
| Figure 5: | Reverse Cumulative Distribution of Neutralizing Antibody against 2017 A/H7N9 by |
| | Study Day, Treatment Arm and Age Stratum, Per Protocol Population*158 |
| Figure 6: | Geometric Mean Titers of Hemagglutination Inhibition Antibody Against 2017 |
| | A/H7N9 by Study Day, Treatment Arm and Age Stratum, Modified Intent to Treat |
| | Population* |
| Figure 7: | Geometric Mean Titers of Hemagglutination Inhibition Antibody against A/H5N8 by |
| | Study Day, Treatment Arm and Age Stratum, Per Protocol Population*159 |
| Figure 8: | Geometric Mean Titers of Neutralizing Antibody against A/H5N8 Study Day, |
| | Treatment Arm and Age Stratum, Modified Intent to Treat Population*159 |
| Figure 9: | Geometric Mean Titers of Neutralizing Antibody against A/H5N8 by Study Day, |
| | Treatment Arm and Age Stratum, Per Protocol Population* |
| Figure 10: | Correlation of Hemagglutination Inhibition Antibody and Neutralizing Antibody |
| | Against 2017 A/H7N9 by Study Day, Treatment Arm and Age Stratum, Modified |
| | Intent-to-Treat Population* |
| Figure 11: | Correlation of Hemagglutination Inhibition Antibody and Neutralizing Antibody |
| | Against 2017 A/H7N9 by Study Day, Treatment Arm and Age Stratum, Per Protocol |
| | Population* |
| Figure 12: | Reverse Cumulative Distribution of Hemagglutination Inhibition Antibody against |
| | [Antigenically Drifted Strain] by Study Day, Treatment Arm and Age Stratum, Per |
| | Protocol Population*161 |
| Figure 13: | Reverse Cumulative Distribution of Neutralizing Antibody against [Antigenically |
| | Drifted Strain] by Study Day, Treatment Arm and Age Stratum, Per Protocol |
| | Population |
| Figure 14: | Geometric Mean Titers of Hemagglutination Inhibition Antibody against |
| | [Antigenically Drifted Strain] by Study Day, Treatment Arm and Age Stratum, Per |
| | Protocol Population 162 |
| Figure 15: | Geometric Mean Titers of Hemagglutination Inhibition Antibody against |
| | [Antigenically Drifted Strain] by Study Day, Treatment Arm and Age Stratum, Per |
| | Protocol Population 162 |
| Figure 16: | Correlation of Hemagglutination Inhibition Antibody and Neutralizing Antibody |
| | Against [Antigenically Drifted Strain] by Study Day, Treatment Arm and Age Stratum, |
| D: 15 | Per Protocol Population |
| Figure 17: | Correlation of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 and |
| | [Antigenically Drifted Strain] by Study Day, Treatment Arm and Age Stratum, Per |
| E: 10 | Protocol Population 163 |
| Figure 18: | Correlation of Neutralizing Antibody Against 2017 A/H7N9 and [Antigenically Drifted |
| | Strain] by Study Day, Treatment Arm and Age Stratum, Per Protocol Population 163 |

| Figure 19: | Maximum Severity of Solicited Systemic Symptoms per Subject by Day Post Study |
|---|---|
| | Vaccination |
| Figure 20: | Maximum Severity of Solicited Local Symptoms per Subject by Day Post Study |
| | Vaccination |
| Figure 21: | Frequency of Unsolicited Adverse Events by MedDRA System Organ Class and |
| | Severity |
| Figure 22: | Incidence of Unsolicited Adverse Events by MedDRA System Organ Class and |
| | Severity |
| Figure 23: | Frequency of Adverse Events by MedDRA System Organ Class and Relationship to |
| | Treatment |
| Figure 24: | Incidence of Adverse Events by MedDRA System Organ Class and Relationship to |
| | Treatment |
| Figure 25: | Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory |
| | Parameter and Treatment Arm – White Blood Cells |
| Figure 26: | Laboratory Summary Statistics of Change from Baseline by Parameter, Maximum |
| | Severity, Study Day, and Treatment Arm – Hemoglobin |
| Figure 27: | Laboratory Summary Statistics of Change from Baseline Results by Parameter, |
| | Maximum Severity, Study Day, and Treatment Arm – Platelets |
| Figure 28: | Laboratory Summary Statistics of Change from Baseline by Parameter, Maximum |
| | Severity, Study Day, and Treatment Arm – Alanine Aminotransferase (ALT) 169 |
| Figure 29: | Laboratory Summary Statistics of Change from Baseline Results by Parameter, |
| | Maximum Severity, Study Day, and Treatment Arm – Total Bilirubin |
| Figure 30: | Laboratory Summary Statistics of Change from Baseline Results by Parameter, |
| | Maximum Severity, Study Day, and Treatment Arm – Creatinine |

## 10.1 Disposition of Subjects Figures

Figure 1: CONSORT Flow Diagram\*



#### 14.2.2 Immunogenicity Figures

Figure 2: Reverse Cumulative Distribution of Hemagglutination Inhibition Antibody against 2017 A/H7N9 by Study Day, Treatment Arm and Age Stratum, Modified Intent to Treat Population\*

[Implementation Note: A generic sample figure is shown below. The RCD curves should be presented in a single figure with separate panels for each study day (, Day 8, Day 22, Day 29, Day 43, Day 202). Figures generated for expedited interim analysis and preliminary report will include data from all available visits at the time of report generation. Visit labels should be included in the panel headers. Within each panel individual curves should be used for each treatment arm and strata within treatment arm (ten curves). Each treatment arm should have a separate color and marker with dashed/solid lines used to distinguish strata  $(19-65, \ge 65)$ .]



Figures with similar format:

Figure 3: Reverse Cumulative Distribution of Hemagglutination Inhibition Antibody against 2017 A/H7N9 by Study Day, Treatment Arm and Age Stratum, Per Protocol Population\*

Figure 4: Reverse Cumulative Distribution of Neutralizing Antibody Against 2017 A/H7N9 by Study Day, Treatment Arm and Age Stratum, Modified Intent to Treat Population\*

Figure 5: Reverse Cumulative Distribution of Neutralizing Antibody against 2017 A/H7N9 by Study Day, Treatment Arm and Age Stratum, Per Protocol Population\*

Figure 6: Geometric Mean Titers of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 by Study Day, Treatment Arm and Age Stratum, Modified Intent to Treat Population\*

[Implementation Note: A generic sample figure is shown below. Planned Study Day is plotted along the x-axis, with visit labels as tick labels. Titer is plotted on the y-axis on the log-10 scale. GMT should be plotted at each visit with upper and lower error bars for the 95% CI for each treatment group with different marker shapes/colors for each treatment arm. Each treatment arm should have a separate color and marker shape, with open/closed markers and dashed/solid lines used to distinguish strata (19-65, ≥65)]

Note: this figure will be generated for the preliminary report including data through Day 43, then regenerated for the final CSR to include all data through Day 202.



Figures with similar format:

- Figure 7: Geometric Mean Titers of Hemagglutination Inhibition Antibody against A/H5N8 by Study Day, Treatment Arm and Age Stratum, Per Protocol Population\*
- Figure 8: Geometric Mean Titers of Neutralizing Antibody against A/H5N8 Study Day, Treatment Arm and Age Stratum, Modified Intent to Treat Population\*
- Figure 9: Geometric Mean Titers of Neutralizing Antibody against A/H5N8 by Study Day, Treatment Arm and Age Stratum, Per Protocol Population\*

Figure 10: Correlation of Hemagglutination Inhibition Antibody and Neutralizing Antibody Against 2017 A/H7N9 by Study Day, Treatment Arm and Age Stratum, Modified Intent-to-Treat Population\*

[Implementation Note: A generic sample figure is shown below. The scatter plots should be presented in a single figure with separate panels for each visit (Baseline, D8, D22, D29, D43, D202. Visit labels should be included in the panel header. Within each panel distinct marker types and colors should be used to indicate the treatment arms, with treatment group labels included in a legend. ). Each treatment arm should have a unique color and marker shape, with open/closed markers used to distinguish strata within treatment arm  $(19-65, \ge 65)$  The spearman correlation should be calculated over all subjects and annotated within each panel as "Spearman Correlation (r=0.xx, p=0.xx)"]



Figure with Similar format:

Figure 11: Correlation of Hemagglutination Inhibition Antibody and Neutralizing Antibody Against 2017 A/H7N9 by Study Day, Treatment Arm and Age Stratum, Per Protocol Population\*

Figure 12: Reverse Cumulative Distribution of Hemagglutination Inhibition Antibody against [Antigenically Drifted Strain] by Study Day, Treatment Arm and Age Stratum, Per Protocol Population\*

[Implementation Note: A generic sample figure is shown below. The RCD curves should be presented in a single figure with separate panels for each study day (Baseline[Day1], Day 8, Day 22, Day 29, Day 43, Day 202. Visit labels should be included in the panel headers. Within each panel individual curves should be used for each treatment arm and strata within treatment arm (ten curves). Each treatment arm should have a separate color with dashed/solid lines used to distinguish strata (19-65, ≥65)]

[Implementation Note: repeat for all heterologous strains]



Figure with Similar Format:

Figure 13: Reverse Cumulative Distribution of Neutralizing Antibody against [Antigenically Drifted Strain] by Study Day, Treatment Arm and Age Stratum, Per Protocol Population

Figure 14: Geometric Mean Titers of Hemagglutination Inhibition Antibody against [Antigenically Drifted Strain] by Study Day, Treatment Arm and Age Stratum, Per Protocol Population

[Implementation Note: A generic sample figure is shown below. Planned Study Day is plotted along the x-axis, with visit labels as tick labels. Titer is plotted on the y-axis on the log-10 scale. GMT should be plotted at each visit with upper and lower error bars for the 95% CI for each treatment group with different marker shapes/colors for each treatment arm. Each treatment arm should have a separate color and marker shape, with open/closed markers and dashed/solid lines used to distinguish strata (19-65, ≥65)]

[Implementation Note: repeat for all heterologous strains]



Figure with similar format:

Figure 15: Geometric Mean Titers of Hemagglutination Inhibition Antibody against
[Antigenically Drifted Strain] by Study Day, Treatment Arm and Age Stratum, Per
Protocol Population

Figure 16: Correlation of Hemagglutination Inhibition Antibody and Neutralizing Antibody Against [Antigenically Drifted Strain] by Study Day, Treatment Arm and Age Stratum, Per Protocol Population

[Implementation Note: A generic sample figure is shown below. The scatter plots should be presented in a single figure with separate panels for each visit (Baseline, D8, D22, D29, D43, D202. Visit labels should be included in the panel header. Within each panel distinct marker types and colors should be used to indicate the treatment arms, with treatment group labels included in a legend. Each treatment arm should have a unique color and marker shape, with open/closed markers used to distinguish strata within treatment arm  $(19-65, \ge 65)$  The spearman correlation should be calculated over all subjects and annotated within each panel as "Spearman Correlation (r=0.xx, p=0.xx)"]

[Implementation Note: repeat for all heterologous strains]



Figures with similar format (may repeat as needed for additional strains):

- Figure 17: Correlation of Hemagglutination Inhibition Antibody Against 2017 A/H7N9 and [Antigenically Drifted Strain] by Study Day, Treatment Arm and Age Stratum, Per Protocol Population
- Figure 18: Correlation of Neutralizing Antibody Against 2017 A/H7N9 and [Antigenically Drifted Strain] by Study Day, Treatment Arm and Age Stratum, Per Protocol Population

#### 14.3.1 Safety Figures

#### 14.3.1.1 Solicited Adverse Events

Figure 19: Maximum Severity of Solicited Systemic Symptoms per Subject by Day Post Study Vaccination

[Implementation Note: A Generic figure is shown below. A <u>vertical</u> bar chart should be presented *in* 3 *image files (overall and by strata)* with separate panels for each treatment arm, age strata and study vaccination (5 rows (treatment arms) x 2 columns (vaccination #)). Axes should be labeled as follows: x-axis label: Study Day, y-axis label: Percentage of Subjects (%). The treatment arms should be indicated in the panel headers including "(N=X)", where N = the number of subjects in the in the Safety Population who received the relevant dose. Subjects are counted at most once at the maximum severity across all systemic events reported for the specified time point]



Figure with similar format:

Figure 20: Maximum Severity of Solicited Local Symptoms per Subject by Day Post Study Vaccination

#### 14.3.1.2 Unsolicited Adverse Events

# Figure 21: Frequency of Unsolicited Adverse Events by MedDRA System Organ Class and Severity

[Implementation Note: A Generic figure is shown below. This figure includes all unsolicited events across all vaccinations. A *horizontal* bar chart should be presented *in 3 image files (overall and by strata)* with separate panels for each treatment arm (5 columns (treatment arms)). Axes should be labeled as follows: y-axis label: System Organ Class, y-axis label: Number of Events. The treatment arms should be indicated in the panel headers including "(N=X)", where N = the number of subjects in the in the Safety Population. The y-axis should present all SOCs reported by at least 1 subject and an "All Events" category. Y-axis should be sorted with "All Events first, then in decreasing order of total incidence]



Figure 22: Incidence of Unsolicited Adverse Events by MedDRA System Organ Class and Severity

[Implementation Note: A Generic figure is shown below. This figure includes all unsolicited events across all vaccinations. A *horizontal* bar chart should be presented *in 3 image files* with separate panels for each treatment arm (5 columns). Axes should be labeled as follows: y-axis label: System Organ Class, x-axis label: Percentage of Subjects (%). The treatment arms should be indicated in the panel headers including "(N=X)", where N = the number of subjects in the in the Safety Population. Subjects are counted at most once at the maximum severity across for any events in the applicable SOC. The y-axis should present all SOCs reported by at least 1 subject and an "All Events" category. Y-axis should be sorted with "All Events" first then in decreasing order of total incidence]



Figure 23: Frequency of Adverse Events by MedDRA System Organ Class and Relationship to Treatment

[Implementation Note: A generic sample figure is shown below. This figure includes all unsolicited events across all vaccinations. A *horizontal* bar chart should be presented *in 3 image files* with separate panels for each treatment arm, age strata and study vaccination (5 columns (treatment arms). Axes should be labeled as follows: y-axis label: System Organ Class, y-axis label: Number of Events. The treatment arms should be indicated in the panel headers including "(N=X)", where N = the number of subjects in the in the Safety Population. The y-axis should present all SOCs reported by at least 1 subject and an "All Events" category. Y-axis should be sorted with "All Events first—then in decreasing order of total frequency]



Figure 24: Incidence of Adverse Events by MedDRA System Organ Class and Relationship to Treatment

[Implementation Note: A Generic figure is shown below. This figure includes all unsolicited events across all vaccinations. A <u>horizontal</u> bar chart should be presented *in a 3 image files (overall and by strata)* with separate panels for each treatment arm (5 columns (treatment arms). Axes should be labeled as follows: y-axis label: System Organ Class, x-axis label: Percentage of Subjects (%). The treatment arms should be indicated in the panel headers including "(N=X)", where N = the number of subjects in the in the Safety Population. Subjects are counted at most once at the maximum relationship (related >not-related) across for any events in the applicable SOC. The y-axis should present all SOCs reported by at least 1 subject and an "All Events" category. Y-axis should be sorted with "All Events first, then in decreasing order of total incidence across groups]



#### 14.3.5 Displays of Laboratory Results

Figure 25: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter and Treatment Arm – White Blood Cells

[Implementation note: A generic figure is shown below. Plot should be generated with all treatment groups in a single image file with panels for each treatment arm and strata (5 rows (treatment arms) x 2 columns (strata)) with a box plot shown for each post-baseline study day that labs are drawn (D8, D22, D29). Y-axis should be labeled "[Parameter] Change from baseline ([units]). Repeat for all clinical laboratory parameters: WBC, Hgb, PLT, ALT, T. Bili, Cr]



Figures with similar format:

- Figure 26: Laboratory Summary Statistics of Change from Baseline by Parameter, Maximum Severity, Study Day, and Treatment Arm Hemoglobin
- Figure 27: Laboratory Summary Statistics of Change from Baseline Results by Parameter, Maximum Severity, Study Day, and Treatment Arm Platelets
- Figure 28: Laboratory Summary Statistics of Change from Baseline by Parameter, Maximum Severity, Study Day, and Treatment Arm Alanine Aminotransferase (ALT)

- Figure 29: Laboratory Summary Statistics of Change from Baseline Results by Parameter, Maximum Severity, Study Day, and Treatment Arm Total Bilirubin
- Figure 30: Laboratory Summary Statistics of Change from Baseline Results by Parameter, Maximum Severity, Study Day, and Treatment Arm Creatinine

# APPENDIX 3. LISTINGS MOCK-UPS

# LIST OF LISTINGS

| Listing 1: | 16.1.6 - Listing of Subjects Receiving Investigational Product | 172 |
|---|---|---|
| Listing 2: | 16.2.1 - Early Terminations or Discontinued Subjects | 173 |
| Listing 3: | 16.2.2.1 - Subject-Specific Protocol Deviations | |
| Listing 4: | 16.2.2.2 - Non-Subject-Specific Protocol Deviations | 175 |
| Listing 5: | 16.2.3 - Subjects Excluded from Analysis Populations | |
| Listing 6: | 16.2.4.1 - Demographics Data | 177 |
| Listing 7: | 16.2.4.2 – Pre-Existing and Concurrent Medical Conditions | 178 |
| Listing 8: | 16.2.6 - Individual Immunogenicity Response Data | 180 |
| Listing 9: | 16.2.7.1 - Solicited Events – Systemic Symptoms | |
| Listing 10: | 16.2.7.2 - Solicited Events – Local Symptoms | 182 |
| Listing 11: | 16.2.7.3 - Unsolicited Adverse Events | 183 |
| Listing 12: | 16.2.8.1 - Clinical Laboratory Results – Hematology | 184 |
| Listing 13: | 16.2.8.2 - Clinical Laboratory Results – Hematology | 185 |
| Listing 14: | 16.2.9.1 - Vital Signs | |
| Listing 15: | 16.2.9.2 - Physical Exam Findings | |
| Listing 16: | 16.2.10 - Concomitant Medications | 188 |
| Listing 17: | 16.2.11.1 - Pregnancy Reports – Maternal Information | 189 |
| Listing 18: | 16.2.11.2 - Pregnancy Reports – Gravida and Para | 190 |
| Listing 19: | 16.2.11.3 - Pregnancy Reports – Live Birth Outcomes | |
| Listing 20: | 16.2.11.4 - Pregnancy Reports – Still Birth Outcomes | 190 |
| Listing 21: | 16.2.11.5 - Pregnancy Reports – Spontaneous, Elective, or Therapeutic Abortion | |
| | Outcomes | 191 |

# 16.1.6 Listing of Subjects Receiving Investigational Product

## **Listing 1: 16.1.6 - Listing of Subjects Receiving Investigational Product**

| Subject ID | Randomized<br>Treatment Arm | Age Stratum | Product Received Study<br>Vaccination 1 | Product Received Study<br>Vaccination 2 |
|---|---|---|---|---|

## 16.2 Database Listings by Subject

## **16.2.1 Discontinued Subjects**

## **Listing 2: 16.2.1 - Early Terminations or Discontinued Subjects**

[Implementation Note: Category will be either "Early Termination" or "Treatment Discontinuation." In the "Reason" column, concatenate any "specify" fields, including AE number and DV number.]

| Subject ID | Treatment Arm | Age Stratum | Category | Reason for Early Termination or Treatment Discontinuation | Study Day |
|---|---|---|---|---|---|
#### **16.2.2 Protocol Deviations**

## **Listing 3: 16.2.2.1 - Subject-Specific Protocol Deviations**

[Implementation Note: In the "Deviation" column, concatenate any and all "specify" fields (including visit number, etc.). If "Reason for Deviation" is "Other," concatenate "specify" field, separate by a colon, e.g., "Other: Subject refusal."]

| Subject<br>ID | Treatmen<br>t<br>Group | Age<br>Stratum | DV<br>Number | Deviatio<br>n | Deviati<br>on<br>Catego<br>ry | Study<br>Day | Reason<br>for<br>Deviation | Deviation<br>Resulted<br>in AE? | Deviation<br>Resulted in<br>Subject<br>Termination? | Deviation<br>Affected<br>Product<br>Stability? | Deviation<br>Resolution | Commen ts |
|---|---|---|---|---|---|---|---|---|---|---|---|---|

## **Listing 4: 16.2.2.2 - Non-Subject-Specific Protocol Deviations**

[Implementation Note: In the "Deviation" column, concatenate any and all "specify" fields (including visit number, etc.). If "Reason for Deviation" is "Other," concatenate "specify" field, separate by a colon, e.g., "Other: Subject refusal."]

| Site | Deviation | Start<br>Date | End Date | Reason for<br>Deviation | Deviation<br>Resulted in<br>Subject<br>Termination<br>? | Deviation<br>Affected<br>Product<br>Stability? | Deviation<br>Category | Deviation<br>Resolution | Comments |
|---|---|---|---|---|---|---|---|---|---|

## 16.2.3 Subjects Excluded from the Analysis

#### **Listing 5: 16.2.3 - Subjects Excluded from Analysis Populations**

[Implementation Note: This data in this listing should be congruent with the "Analysis Populations by Treatment Group" table. The reasons included here should match the SAP text that describes who will be excluded from analyses.]

| Treatment Group | Age Stratum | Subject ID | Analyses in which<br>Subject is Included | Analyses from which<br>Subject is Excluded | Results Available? | Reason Subject<br>Excluded |
|---|---|---|---|---|---|---|
| | | | [e.g., Safety, ITT, PP] | [e.g., Safety, ITT, PP, Day x] | | |
| | | | | | | _ |

Note: "Yes" in the "Results available" column indicates that available data were removed from the analysis. "No" indicates that no data were available for inclusion in the analysis.

## 16.2.4 Demographic Data

## **Listing 6: 16.2.4.1 - Demographics Data**

[Implementation Note: If a subject is multi-racial, in "Race" column, note "Multiple: (list races, separated by a comma)."]

| Subject ID | Treatment Group | Age Stratum | Sex | Age at Enrollment<br>(years) | Ethnicity | Race | BMI | Seasonal<br>Influenza<br>Received<br>(2016-2017) | Seasonal<br>Influenza<br>Received<br>(2017-2018) |
|---|---|---|---|---|---|---|---|---|---|

## **Listing 7: 16.2.4.2 – Pre-Existing and Concurrent Medical Conditions**

[Implementation Note: "Condition Start Day" and "Condition End Day" are relative to enrollment (which is Day 1, day before enrollment is Day 1). If ongoing, display "Ongoing" in the "Condition End Day" column

| Subject<br>ID | Treatment<br>Group | Age<br>Stratum | MH<br>Number | Medical History<br>Term | Condition Start<br>Day | Condition End<br>Day | MedDRA System Organ<br>Class | MedDRA Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|

# 16.2.5 Compliance and/or Drug Concentration Data (if available)

Not applicable for this study.

# 16.2.6 Individual Immunogenicity Response Data

**Listing 8: 16.2.6 - Individual Immunogenicity Response Data** 

| Subject<br>ID | Treatment<br>Group | Age Stratum | Planned Time Point | Actual Study<br>Day | Assay | Strain | Titer Replicate 1 | Titer Replicate 2 |
|---|---|---|---|---|---|---|---|---|

## 16.2.7 Adverse Events

**Listing 9: 16.2.7.1 - Solicited Events – Systemic Symptoms** 

| Subject ID | Treatment Arm | Age Stratum | Vac Number | Post Vac Day | Assessmenta | Symptom | Severity | Attributed to<br>Alternate<br>Etiology? <sup>b</sup> | Alternate<br>Etiology |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | MA | | | | |
| | | | | | Clinic | | | | |

<sup>&</sup>lt;sup>a</sup> MA = Data reported by subject on the Memory Aid and reviewed by clinic staff and reported in Solicited Events eCRF.

Clinic = Data collected by clinic staff during physical exam or symptom assessment (treatment administration record, in-clinic assessment, etc.)

<sup>&</sup>lt;sup>b</sup> Grade 3 events only.

**Listing 10: 16.2.7.2 - Solicited Events – Local Symptoms** 

| Subject ID | Treatment Arm | Age Stratum | Vac Number | Post Vac Day | Assessment <sup>a</sup> | Symptom | Severity |
|---|---|---|---|---|---|---|---|
| | | | | | MA | | |
| | | | | | Clinic | | |

<sup>&</sup>lt;sup>a</sup> MA = Data reported by subject on the Memory Aid and reviewed by clinic staff and reported in Solicited Events eCRF.

Clinic = Data collected by clinic staff during physical exam or symptom assessment (treatment administration record, in-clinic assessment, etc.)

**Listing 11: 16.2.7.3 - Unsolicited Adverse Events** 

| Adverse<br>Event | Associated with Vac # | # of Days Post Associated Vac (Duration) | Severity | SAE?<br>MAAE?<br>PIMMC? | Relationship<br>to Study<br>Treatment | In Not<br>Related,<br>Alternative<br>Etiology | Action<br>Taken<br>with<br>Study<br>Treatment | Subject<br>Discontinued<br>Due to AE | Outcome | MedDRA<br>System<br>Organ<br>Class | MedDRA<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID | : , Treatment | Arm: , AE Nu | ımber: | | | | | | | | |
| | | | | SAE: No<br>MAAE: Yes<br>PIMMC: No | | | | | | | |
| Comments: | | | | | | | | | | | |
| Subject ID | :, Treatment | Arm: , AE Nu | ımber: | | | | | | | | |
| Comments: | • | | | | 1 | <u>'</u> | | 1 | | | 1 |
| Note: For a | Note: For additional details about SAEs, see Section 14.3.3 | | | | | | | | | | |

#### 16.2.8 Individual Laboratory Measurements

#### **Listing 12: 16.2.8.1 - Clinical Laboratory Results – Hematology**

[Implementation Note: These listings (for hematology and chemistry) include all laboratory results, scheduled and unscheduled. These listings are not color-coded, but the severity should be included in parentheses after the result for abnormal results, e.g., 16.2 (Mild). The "extra" fields that are completed for abnormal results are not included in this listing; they are included in the listing of abnormal laboratory results that is included in the table shells.]

| Subject ID | Treatment Arm | Age<br>Stratum | Sex | Age<br>(years) | Planned<br>Time<br>Point | Actual<br>Study<br>Day | Alanine<br>aminotransferase<br>(IU/L) | Total Bilirubin<br>(mg/dL) | Creatinine<br>(mg/dL) |
|---|---|---|---|---|---|---|---|---|---|

**Listing 13: 16.2.8.2 - Clinical Laboratory Results – Hematology** 

| Subject ID | Treatment Arm | Age<br>Stratum | Sex | Age<br>(years) | Planned<br>Time<br>Point | Actual<br>Study<br>Day | White Blood Cell<br>(10³/μL) | Hemoglobin<br>(g/dL) | Platelets<br>(10³/μL) |
|---|---|---|---|---|---|---|---|---|---|

## 16.2.9 Vital Signs and Physical Exam Findings

## **Listing 14: 16.2.9.1 - Vital Signs**

[Implementation Note: This listing includes all vital sign assessments, scheduled and unscheduled. These listings are not color-coded, but the severity should be included in parentheses after the result for abnormal assessments, e.g., 100.7 (Mild).]

| Subject ID | Treatment Arm | Age Stratum | Planned<br>Time Point | Actual<br>Study Day | Temperature<br>(°C) | Systolic Blood<br>Pressure<br>(mmHg) | Diastolic Blood<br>Pressure<br>(mmHg) | Pulse<br>(beats/min) |
|---|---|---|---|---|---|---|---|---|

### Listing 15: 16.2.9.2 - Physical Exam Findings

[Implementation Note: This listing includes all physical exam findings, scheduled and unscheduled. If a subject does not have any findings upon examination, they will not be included in this listing. If reported as an AE, display "Yes" with the AE Number in parentheses, e.g., "Yes (7)".]

| Subject ID | Treatment Arm | Age<br>Stratum | Planned<br>Time<br>Point | Actual<br>Study Day | Body System | Abnormal Finding | Reported as an AE?<br>(AE Number) |
|---|---|---|---|---|---|---|---|

#### **16.2.10** Concomitant Medications

#### **Listing 16: 16.2.10 - Concomitant Medications**

[Implementation Note: "Medication Start Day" and "Medication End Day" are relative to enrollment (which is Day 1, day before enrollment is Day -1). For medication start dates that are > 30 days prior to enrollment, rather than use exact study days, categorize as follows:

- > 5 years prior to enrollment
- 1-5 years prior to enrollment
- 1-12 months prior to enrollment

If ongoing, display "Ongoing" in the "Medication End Day" column. If taken for an AE or MH, display "Yes" with the AE or MH Number in parentheses, e.g., "Yes (7)".]

| Subject<br>ID | Treatment<br>Group | Age<br>Stratum | CM<br>Number | Medication | Medication Start<br>Day | Medication End<br>Day | Indication | Taken for an<br>AE?<br>(AE Number) | Taken for a<br>condition on Medical<br>History?<br>(MH Number) |
|---|---|---|---|---|---|---|---|---|---|

#### 16.2.11 Pregnancy Reports

[Implementation Note: Only include the "Pregnancy Number" column if a subject has more than 1 pregnancy. Date of Conception will be calculated based on estimated delivery date. BMI will be calculated based on pre-pregnancy height and weight. Mother's weight gain will be calculated based on pre-pregnancy weight and end of pregnancy weight. If a major congenital anomaly with previous pregnancy, display "Yes" and the text from the "specify" field, separated by a colon. If any substance use is reported, include a listing of substance use. If autopsy revealed an alternate etiology, display "Yes" and the text from the "specify" field, separated by a colon.]

Listing 17: 16.2.11.1 - Pregnancy Reports – Maternal Information

| Subject ID | Treatment<br>Arm | Pregnancy<br>Number | Study Day<br>Corresponding<br>to Estimated<br>Date of<br>Conception | Source of<br>Maternal<br>Information | Pregnancy<br>Status | Mother's<br>Pre-<br>Pregnancy<br>BMI | Mother's<br>Weight<br>Gain<br>During<br>Pregnancy | Tobacco, Alcohol, or Drug Use During Pregnancy? | Medications<br>During<br>Pregnancy? | Maternal<br>Complications<br>During<br>Pregnancy? | Maternal<br>Complications<br>During Labor,<br>Delivery, or<br>Post-Partum? |
|---|---|---|---|---|---|---|---|---|---|---|---|

Note: Maternal Complications are included in the Adverse Event listing. Medications taken during pregnancy are included in the Concomitant Medications Listing.

Listing 18: 16.2.11.2 - Pregnancy Reports – Gravida and Para

| | | | | Live Births | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>ID | Pregnancy<br>Number | Gravida | Extremely PB <sup>1</sup> | Very<br>Early<br>PB <sup>1</sup> | Early<br>PB <sup>1</sup> | Late<br>PB <sup>1</sup> | Early<br>TB <sup>2</sup> | Full<br>TB <sup>2</sup> | Late<br>TB <sup>2</sup> | Post<br>TB <sup>2</sup> | Still<br>Births | Spontaneous<br>Abortion/<br>Miscarriage | Elective<br>Abortions | Therapeutic<br>Abortions | Major<br>Congenital<br>Anomaly with<br>Previous<br>Pregnancy? |

<sup>&</sup>lt;sup>1</sup> Preterm Birth

Note: Gravida includes the current pregnancy, para events do not.

**Listing 19: 16.2.11.3 - Pregnancy Reports – Live Birth Outcomes** 

| Subject<br>ID | Pregnancy<br>Number | Fetus<br>Number | Pregnancy<br>Outcome<br>(for this<br>Fetus) | Fetal Distress During Labor and Delivery? | Delivery<br>Method | Gestational<br>Age at Live<br>Birth | Size for<br>Gestational<br>Age | Apgar<br>Score,<br>1<br>minute | Apgar<br>Score, 5<br>minutes | Cord<br>pH | Congenital Anomalies? | Illnesses/<br>Hospitalizations<br>within 1 Month<br>of Birth? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|

Note: Congenital Anomalies are included in the Adverse Event listing.

**Listing 20: 16.2.11.4 - Pregnancy Reports – Still Birth Outcomes** 

| Subject<br>ID | Date of<br>Initial<br>Report | Fetus<br>Number | Pregnancy<br>Outcome<br>(for this<br>Fetus) | Fetal Distress During Labor and Delivery? | Delivery<br>Method | Gestational<br>Age at Still<br>Birth | Size for<br>Gestational<br>Age | Cord pH | Congenital Anomalies? | Autopsy<br>Performed? | If Autopsy,<br>Etiology for Still<br>Birth Identified? |
|---|---|---|---|---|---|---|---|---|---|---|---|

<sup>&</sup>lt;sup>2</sup> Term Birth

## Listing 21: 16.2.11.5 - Pregnancy Reports – Spontaneous, Elective, or Therapeutic Abortion Outcomes

| Subject<br>ID | Date of Initial<br>Report | Fetus Number | Pregnancy<br>Outcome (for this<br>Fetus) | Gestational Age at<br>Termination | Abnormality in Product of Conception? | Reason for Therapeutic<br>Abortion |
|---|---|---|---|---|---|---|